

#### STATISTICAL ANALYSIS PLAN

Study Title: A Phase 2, Open-label, Translational Biology Study of

Momelotinib in Transfusion-Dependent Subjects with Primary Myelofibrosis (PMF) or Post-polycythemia Vera or Post-essential

Thrombocythemia Myelofibrosis (Post-PV/ET MF)

Name of Test Drug: Momelotinib (MMB)

Study Number: GS-US-352-1672

**Protocol Version (Date):** 18 May 2015

**Analysis Type:** Final Analysis

**Analysis Plan Version:** Version 1.0

**Analysis Plan Date:** 16 October 2017

**Analysis Plan Author:** Yafeng Zhang

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TA | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF T | TABLES | 4 |
| LIS | T OF A | ABBREVIATIONS | 5 |
| 1. | INTR | INTRODUCTION | |
| •• | | Study Objectives | |
| | 1.1.<br>1.2. | | |
| | 1.2. | Study Design | |
| | | 1.2.1. Design Configuration and Subject Population | |
| | | 1.2.3. Inclusion Criteria | |
| | | 1.2.4. Exclusion Criteria | |
| | | 1.2.5. Efficacy Endpoints | |
| | | 1.2.6. Safety | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | E OF PLANNED ANALYSIS | 13 |
| | 2.1. | Data Monitoring Committee | 13 |
| | 2.2. | Interim Analysis | 13 |
| | 2.3. | Final Analysis | 13 |
| | 2.4. | Follow-up Analysis | 13 |
| 3. | GENI | IERAL CONSIDERATIONS FOR DATA ANALYSES | 14 |
| 3. | 3.1. | Analysis Sets | 14 |
| | | 3.1.1. Safety Analysis Set | 14 |
| | | 3.1.2. Biomarker Analysis Set | |
| | | 3.1.3. Pharmacokinetic Analysis Set | |
| | 3.2. | Strata and Covariates | |
| | 3.3. | Examination of Subject Subsets | |
| | 3.4. | Multiple Comparisons | |
| | 3.5. | Missing Data and Outliers | |
| | | 3.5.1. Missing Data | |
| | 2.6 | 3.5.2. Outliers | |
| | 3.6. | Data Handling Conventions and Transformations | |
| | | 3.6.2. Data Handling for PK Data | |
| | | 3.6.3. Data Handling for Efficacy Endpoints | |
| | 3.7. | Visit Windows | |
| | 3.7. | 3.7.1. Definition of Study Day | |
| | | 3.7.2. Analysis Windows | |
| | | 3.7.3. Selection of Data in the Event of Multiple Records i | |
| | | Window | |
| 4. | SUBJ | JECT DISPOSITION | 23 |
| | 4.1. Subject Enrollment and Disposition | | |
| | 4.2. | Extent of Exposure | |
| | | 4.2.1. Duration of Exposure to MMB | |
| | | 4.2.2. Adherence to MMB | 24 |
| | 4.3. | Protocol Deviations | 25 |
| 5. | BASI | ELINE CHARACTERISTICS | 27 |
| | 5.1. | Demographics | 27 |

| | 5.2. | Other Baseline Characteristics | |
|---|---|---|---|
| | 5.3. | Medical History | |
| | | 5.3.1. General Medical History | |
| | | 5.3.2. Myelofibrosis Disease History | |
| | 5.4. | Myelofibrosis Disease-Specific Prior Therapy | |
| 6. | EFFI | CACY ANALYSES | 29 |
| | 6.1. | Primary Efficacy Endpoint | 29 |
| | | 6.1.1. Definition of the Primary Efficacy Endpoint | 29 |
| | | 6.1.2. Statistical Hypothesis for the Primary Efficacy Endpoint | 30 |
| | | 6.1.3. Analysis of the Primary Efficacy Endpoint | 30 |
| | | 6.1.4. Exploratory Analysis | |
| | 6.2. | Secondary Efficacy Endpoints | |
| | | 6.2.1. Definition of Secondary Efficacy Endpoints | |
| | | 6.2.2. Analysis Methods for Secondary Efficacy Endpoints | |
| | 6.3. | Exploratory Efficacy Endpoint | |
| | | 6.3.1. Definition of Exploratory Efficacy Endpoints | |
| | | 6.3.2. Analysis Methods for Exploratory Efficacy Endpoints | |
| | 6.4. | Changes From Protocol-Specified Efficacy Analyses | 39 |
| 7. | SAFE | ETY ANALYSES | 40 |
| | 7.1. | Adverse Events and Deaths | 40 |
| | | 7.1.1. Adverse Event Dictionary | 40 |
| | | 7.1.2. Adverse Event Severity | |
| | | 7.1.3. Relationship of Adverse Events to MMB | |
| | | 7.1.4. Serious Adverse Events | |
| | | 7.1.5. Treatment-Emergent Adverse Events | |
| | | 7.1.6. Summaries of Adverse Events and Deaths | |
| | | 7.1.7. Additional Analysis of Adverse Events | |
| | 7.2. | Laboratory Evaluations | |
| | | 7.2.1. Graded Laboratory Values | |
| | <i>7</i> .0 | 7.2.2. Shifts Relative to the Baseline Value | |
| | 7.3. | | |
| | 7.4. | Prior and Concomitant Medications | |
| | 7.5 | 7.4.1. Prior Medications and Concomitant Medications | |
| | 7.5.<br>7.6. | Electrocardiogram Results | |
| | 7.0. | Other Safety Measures | |
| 8. | РΗΔΙ | RMACOKINETIC ANALYSES | |
| | | ERENCES | |
| 9. | | | |
| 10. | | TWARE | |
| 11. | SAP I | REVISION | 51 |
| 12. | APPE | ENDICES | 52 |
| | | ndix 1. Table of Contents for Statistical Tables, Figures, and Listings | |
| | | ndix 2. Study Procedures Table | |
| | | ndix 3. Peripheral Neuropathy SMQ AEs | |
| | | ndix 4. Cataract MST AEs | |
| | | ndix 5. Leukemic Transformation MST AEs | |
| | | ndix 6. Validation document of hepcidin testing from Radboud University | |
| | Appe | ndix 7. Validation document of pSTAT testing from Covance | |

# LIST OF TABLES

| Table 3-1. | Analysis Windows for Efficacy Endpoints MRI Spleen Volume Response Assessment and MRI Liver Iron Content | 19 |
|---|---|---|
| Table 3-2. | Analysis Windows for Efficacy Analyses of TSS Response Rate at Week 24 | |
| Table 3-3. | Analysis Windows for Hepcidin | |
| Table 3-4. | Analysis Windows for Anemia Related Biomarkers <sup>a</sup> | |
| Table 3-5. | Analysis Windows for Erythropoietin | 20 |
| Table 3-6. | Analysis Windows for C-reactive Protein | |
| Table 3-7. | Analysis Windows for Pharmacodynamics Biomarker pSTAT3 | |
| Table 7-1. | Grading of Hemoglobin Severity | |

### LIST OF ABBREVIATIONS

AE adverse event

ADME absorption, distribution, metabolism and elimination

ALT alanine aminotransferase
ANC absolute neutrophil count
AST aspartate aminotransferase

ATC Anatomical-Therapeutic-Chemical (drug coding system)

BCRP breast cancer resistant protein
BLQ below the limit of quantitation

BMI body mass index
BUN blood urea nitrogen
CBC complete blood count

CFR Code of Federal Regulations

 ${
m CI}$  confidence interval  ${
m CL}_{cr}$  creatinine clearance

CML chronic myelogenous leukemia

CR complete remission
CK creatine kinase
CRF case report form

CRO contract (or clinical) research organization

CRP C-reaction protein
CSR clinical study report

CT computed tomography/computed axial tomography scan
CTCAE Common Terminology Criteria for Adverse Events

CYP450 cytochrome P450

Da dalton

DIPSS Dynamic International Prognostic Scoring System

DMC data monitoring committee

DSPH Drug Safety and Public Health

ECG electrocardiogram

eCRF electronic case report form(s)

EDC electronic data capture

eDiary electronic diary
EOT end of treatment
EPO erythropoietin

ESDD Early Study Drug Discontinuation

ET essential thrombocythemia

FAS Full Analysis Set

FDA (United States) Food and Drug Administration

FSH follicle stimulating hormone

GCP Good Clinical Practice(guidelines)

Gilead Gilead Sciences

GLP Good Laboratory Practice(guidelines)

hCG human chorionic gonadotropin

Hgb hemoglobin

HLGT high-level group term HLT high-level term

HIV human immunodeficiency virus

IB investigator's brochure

ICH International Conference on Harmonisation (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

ID subject identification IP investigational product

IPSS International Prognostic Scoring System

ITT intent to treat

IWG International Working Group
LIC liver iron concentration
LLOQ lower limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

MF myelofibrosis
MMB momelotinib

MPN myeloproliferative neoplasm

MPN-SAF TSS Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score

MRI magnetic resonance imaging
MST MedDRA Search Term
ORR overall response rate

PGIC Patient Global Impression of Change

PK pharmacokinetic
PMF primary myelofibrosis

PP per protocol

PRO patient-reported outcome

PT preferred term
PV polycythemia vera

Q1, Q3 first quartile, third quartile

RBC red blood cell

SAP statistical analysis plan

SE standard error

SI (units) international system of units

SOC system organ class

SRR24 splenic response rate at Week 24

StD standard deviation

TD transfusion-dependent/ dependence
TEAE treatment-emergent adverse event

TFLs tables, figures, and listings

TI transfusion-independent/independence

TSAT transferrin saturation
TSS total symptom score

U units

ULN upper limit of normal

WHO World Health Organization

## 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for Study GS-US-352-1672. This SAP is based on the study protocol dated 18 May 2015 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

# 1.1. Study Objectives

The primary objective of this study is as follows:

• To determine the transfusion independence response rate for transfusion dependent myelofibrosis (MF) subjects treated with momelotinib (MMB)

The secondary objectives of this study are as follows:

- To evaluate baseline levels and changes in markers of iron metabolism in transfusion dependent MF subjects treated with MMB
- To assess inhibition of JAK1/2 in transfusion dependent MF subjects treated with MMB
- To evaluate MMB pharmacokinetics (PK) in transfusion dependent MF subjects
- To evaluate changes in circulating cytokine and inflammatory markers in transfusion dependent MF subjects treated with MMB

#### 1.2. Study Design

#### 1.2.1. Design Configuration and Subject Population

This is a Phase 2, single-arm, open-label study of MMB to determine the transfusion independent response rate for transfusion-dependent subjects with primary myelofibrosis (PMF) or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (Post-PV/MF). Study candidates will be adult males or females who are transfusion dependent with PMF or Post-PV/MF.

Eligible subjects will receive MMB tablet once daily for 24 weeks ( $\pm$  7 days) on study. The starting dose of MMB for all subjects will be 200 mg tablet. The dose of MMB may be withheld or adjusted according to the criteria in the protocol.

Study visits will be completed at 2 weeks and 4 weeks following the initiation of MMB treatment, and every 4 weeks thereafter until Week 24. Following the screening, subjects will receive an electronic diary (eDiary) for daily completion of the modified Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS). Subjects will

complete the modified MPN-SAF TSS daily starting from screening and through 24 weeks of study participation. Laboratory analyses (serum chemistry, liver tests, hematology, urinalysis, pregnancy testing for females of childbearing potential), vital signs, adverse events (AEs), concomitant medications and disease assessments will be completed at regular study visits as defined in Appendix 3.

After completion of the 24-week ( $\pm$  7 days) treatment phase visit procedures, subjects who respond to treatment, at the investigator's discretion, will have the option of continuing on maintenance therapy with MMB on Study GS-US-352-1154 at the MMB dose level they tolerated and/or derived clinical benefit from during the 24-week treatment period.

## 1.2.2. Number of Subjects Planned

Approximately 40

#### 1.2.3. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

- 1) Age  $\geq$  18 years old
- 2) Diagnosis of PMF or Post PV/ET-MF
- 3) Requires myelofibrosis therapy, in the opinion of the investigator
- 4) High risk or intermediate-2 risk defined by the Dynamic International Prognostic Scoring System (DIPSS) or intermediate-1 risk defined by DIPSS and associated with symptomatic splenomegaly and/or hepatomegaly
- 5) Transfusion dependent at baseline, defined as ≥ 4U red blood cell (RBC) transfusion in the 8 weeks prior to first dose of MMB
- 6) Acceptable organ function as evidenced by the following:
  - a) Platelet Count  $\geq 50 \times 10^9/L$
  - b) AST/SGOT and ALT/SGPT  $\leq$  3 x upper limit of normal (ULN) or AST/SGOT or ALT/SGPT  $\leq$  5 x ULN if liver is involved by disease process as judged by the investigator
  - c) Serum creatinine  $\leq 2.0 \text{ mg/dL}$  or calculated creatinine clearance of  $\geq 60 \text{mL/min}$
  - d) Direct bilirubin  $\leq 2.0 \text{ x ULN}$
- 7) Peripheral blood blast count < 20%
- 8) Life expectancy of > 24 weeks

- 9) A negative serum pregnancy test for female subjects (unless surgically sterile or greater than two years postmenopausal)
- 10) Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Appendix 3 in the protocol
- 11) Lactating females must agree to discontinue nursing before MMB administration
- 12) Able to understand and willing to sign the informed consent form

#### 1.2.4. Exclusion Criteria

Subject who meet any of the following exclusion criteria are not to be enrolled in this study:

- 1) Prior splenectomy
- 2) Splenic irradiation within 3 months prior to the first dose of MMB
- 3) Prior treatment with MMB
- 4) Known positive status of human immunodeficiency virus (HIV)
- 5) Chronic active or acute viral hepatitis A, B, or C infection (testing required for hepatitis B and C), or hepatitis B or C carrier
- 6) Use of strong CYP3A4 inducer within 2 weeks prior to the first dose of MMB
- 7) Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician
- 8) History of a prior diagnosis of any malignancy other than PMF or Post PV/ET-MF except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for >1 year prior to enrollment, or any other cancer that has been in complete remission without treatment for ≥ 5 years prior to enrollment.
- 9) Treatment with a JAK inhibitor within 21 days of the planned first dose of MMB
- 10) Documented myocardial infarction or unstable/uncontrolled cardiac disease (eg, unstable angina, congestive heart failure [New York Heart Association > Class III]) within 6 months of randomization
- 11) Presence of peripheral neuropathy  $\geq$  CTCAE Grade 2

- 12) Unwilling or unable to undergo Magnetic Resonance Imaging (MRI) per requirements (Please see the Section 6.2.11.2 in the protocol)
- 13) Unwilling to consent to genomics sampling
- 14) Pregnant or breast-feeding
- 15) Known hypersensitivity to the study investigational medicinal products, the metabolites, or formulation excipients

# 1.2.5. Efficacy Endpoints

#### **Primary Endpoint**

The primary endpoint is transfusion independence response rate by Week 24, defined as becoming transfusion independent for  $\geq$  12 weeks at any time on study. A subject is considered as transfusion independent on study if no RBC transfusion occurs in any 12 weeks during the 24-week treatment period.

#### **Secondary Endpoints**

The secondary endpoints are:

- Transfusion response rate by Week 24, defined as becoming not transfusion dependent for
   ≥ 8 weeks at any time on study
- Baseline and change in markers of anemia (eg, hepcidin, ferritin)
- Change in pharmacodynamic biomarker pSTAT3
- Splenic response rate at Week 24, defined as ≥ 35% reduction in spleen volume from baseline as measured by MRI/CT
- Response rate in total symptom score (TSS) at Week 24, defined as achieving a ≥ 50% reduction from baseline in TSS as measured by the modified MPNSAF TSS diary
- Pharmacokinetics parameters (Cmax, Clast, Ctau, and AUClast, if available) for MMB
- Change in circulating cytokine and inflammatory markers (eg, IL-6, IL-8, IFN-gamma, TNF-alpha)

## **Exploratory Endpoints**

The exploratory endpoints are:

 Baseline and change in markers of orthogonal or parallel signaling pathways (eg, RAS/MAPK, PI3K/AKT)

- Baseline and change in gene expression profiles in whole blood and somatic mutations in whole blood, if applicable.
- Baseline and change in immune subsets in whole blood
- Change in exploratory pharmacodynamics markers of signaling mediated by JAK1 and/or JAK2 (eg, pSTAT1, pSTAT5, and pSTAT6)

#### **Pharmacokinetics**

Blood samples will be collected at the time points specified in the protocol.

# **1.2.6.** Safety

The overall safety profile of MMB will be characterized by the type, frequency, severity, timing of onset, duration, and relationship to MMB of any adverse events (AEs) or abnormalities of laboratory tests; serious adverse events (SAEs); or AEs leading to discontinuation of MMB.

## 1.3. Sample Size and Power

This study will enroll approximately 40 subjects. Due to the exploratory nature, the study is not designed to detect a specific effect size. A sample size of 40 subjects is considered adequate for this exploratory study.

## 2. TYPE OF PLANNED ANALYSIS

# 2.1. Data Monitoring Committee

This study does not have a data monitoring committee (DMC).

### 2.2. Interim Analysis

No formal interim efficacy analysis is planned.

## 2.3. Final Analysis

After all subjects have completed the study, outstanding data queries have been resolved, and the database has been cleaned and finalized, the final analysis of the data will be performed.

## 2.4. Follow-up Analysis

After the final analysis, additional supplemental analyses of efficacy and safety may be performed to satisfy regulatory requirements and to perform long-term efficacy, safety, and overall survival follow-up.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects [n], mean, standard deviation [StD] or standard error [SE], median, first quartile [Q1], third quartile [Q3], minimum, and maximum will be presented.

All statistical tests will be 2-sided and performed at the 10% significance level unless otherwise specified.

Data collected in the study will be presented in by-subject listings for all enrolled subjects, regardless of whether or not they received MMB. All by-subject listings will be presented by subject identification (ID) number in ascending order, unless otherwise specified.

### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. For each analysis set, the number and percentage of subjects eligible for inclusion, as well as the number and percentage of subjects who were excluded and the reasons for their exclusion, will be provided. A listing of reasons for exclusion from analysis sets will be provided by subject.

# 3.1.1. Safety Analysis Set

The Safety Analysis Set includes all subjects who receive  $\geq 1$  dose of MMB. Since this study is a non-randomized study, the Safety Analysis Set will be used for subject's characteristics, efficacy and safety endpoints, and study treatment administration. This is the primary analysis set for safety analyses.

### 3.1.2. Biomarker Analysis Set

The Biomarker Analysis Set consists of all subjects in the Safety Analysis Set who have the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest. The Biomarker Analysis Set will be used for biomarkers and the correlation analyses between biomarkers and efficacy clinical endpoints.

### 3.1.3. Pharmacokinetic Analysis Set

The Pharmacokinetic (PK) Analysis Set includes all subjects who have been administered at least 1 dose of investigational drug and have at least 1 non-missing postdose concentration value for the corresponding analysis in serum or plasma.

#### 3.2. Strata and Covariates

This study does not use a stratified randomization schedule in enrolling subjects.

# 3.3. Examination of Subject Subsets

The primary efficacy endpoints will be examined using the following subsets:

- Age (< 65 years and  $\ge 65$  years)
- Gender (male and female)
- Race (white and all other races)
- DIPSS assessment (Intermediate-1/2 and high risk)
- Type of MF (PMF, Post-PV MF, and Post ET MF)
- JAK2V617F mutation status at baseline (positive and negative)
- Hemoglobin level at baseline ( $\frac{8g}{dL}$  and  $\frac{8g}{dL}$ )
- TSS at baseline (<median and ≥median)
- Spleen volume at baseline (<median and ≥median)
- Hepcidin at baseline morning time point (<median and ≥median)
- Liver iron content at baseline (<median and ≥median)
- Transferrin saturation at baseline (<50% and  $\ge 50\%$ )

Pharmacokinetics endpoints, AEs and lab abnormalities may be examined in the following subgroups:

- Age (< 65 years and  $\ge$  65 years)
- Gender (male and female)
- Race (white and all other races)

### 3.4. Multiple Comparisons

All endpoint tests will be done at the significance level of 0.1 unless otherwise specified. No multiplicity adjustment will be made for testing, because the endpoints are considered exploratory in nature.

# 3.5. Missing Data and Outliers

## 3.5.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified.

For missing last dosing date of MMB, imputation rules are described in Section 4.2.1. The handling of missing or incomplete dates for disease diagnosis is described in Section 5.3.2.1, for AE onset is described in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.1.

#### 3.5.2. Outliers

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

## 3.6. Data Handling Conventions and Transformations

By-subject listings will be presented for all subjects in the primary analysis set that these listings are supporting and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within subject.

Age (in years) on the date of the first dose of MMB will be used for analyses and presentation in listings.

If a subject was not dosed with MMB at all, the date the informed consent was signed will be used instead of the first dose date of MMB. For some countries, only birth year is collected on the CRF. In those cases, "01 January" will be used for the unknown birth day and month for the purpose of age calculation, unless age is captured on the CRF.

#### 3.6.1. Data Handling for Non-PK Laboratory Data

Non-PK data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows:

- A value that is one unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the limit of quantitation). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception to this rule is any value reported as < 1. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.
- A value that is one unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the limit of quantitation). Values with decimal points will follow the same logic as above.

• The limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the limit of quantitation).

If methods based on the assumption that the data are normally distributed are not adequate, analyses may be performed on transformed or nonparametric analysis methods may be used, as appropriate.

## 3.6.2. Data Handling for PK Data

Natural logarithm transformation will be used for plasma/blood concentrations. Plasma concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the lower limit of quantitation (LLOQ) at post-baseline time points, where LLOQ is corrected for the dilution factor (i.e., reported LLOQ/dilution factor) for determination of summary and order statistics.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

# 3.6.3. Data Handling for Efficacy Endpoints

If there is a significant degree of non-normality for a continuous endpoint, analysis may be performed on log-transformed data or using nonparametric methods, as appropriate.

For MRI spleen response, TSS response, and transfusion-independence (TI) response subjects will be considered as non-responder and as transfusion-dependent (TD) for TD response status in the primary analysis, if subjects early discontinued in the MMB treatment phase prior to the visit or with missing assessments at the corresponding visit.

### 3.7. Visit Windows

## 3.7.1. Definition of Study Day

Study Day 1 will be defined as the day of first dose of MMB administration in the study.

Study day will be calculated from the date of first dose of MMB administration and derived as follows:

- For post dose study days: Assessment Date First Dosing Date + 1
- For days prior to the first dose: Assessment Date First Dosing Date

The last participation date is defined as:

- If subject did not roll over to the GS-US-352-1154 study: the last date from the datasets including BM\_MF2 (bone marrow biopsy), COVLAB (Covance lab), ECG\_EG(Electrocardiogram), EPRO\_ERT (patient-reported outcomes), QS\_PGIC(patient-reported outcomes), EX (MMB administration), IWG (IWG-MRT/ELN response assessment), LVSPQL\_MF (Length of palpable spleen size), VISDT (visit date), VSPERF (vital signs), MRI\_PAREXEL (MRI/CT Spleen Volume).
- If subject was rolled over to the GS-US-352-1154 study: as the last date from previous datasets but prior to or on the Day 1 of GS-US-352-1154
- If subject discontinued MMB treatment due to death, the date of death will be the last participation date in the study.

Note AE, CM (con meds), PR\_TFSN (transfusion), LAB (local lab), LABHGB, LABHEM, PK\_EX\_SERIAL and PK\_SERIAL will not be included in the derivation.

## 3.7.2. Analysis Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

In general, the baseline value will be the last nonmissing value on or prior to the first dose date of MMB. If multiple measurements occur on the same day, the last nonmissing value prior to the time of first dose of MMB will be considered as the baseline value. If these multiple measurements occur at the same time or the time is not available, the average of these measurements (for continuous data) or the worst among these measurements (for categorical data) will be considered the baseline value.

# 3.7.2.1. Analysis Windows for Efficacy Analyses

For efficacy analyses in MMB treatment, observations will be assigned to analysis windows for efficacy analyses of the endpoints MRI splenic response, TSS response rate, hepcidin, anemia related biomarkers, erythropoietin, MRI liver iron content, C-reactive protein, and pharmacodynamics biomarkers, as provided in Table 3-1 through Table 3-7.

The 8-weeks period for RBC transfusion dependence status at baseline is defined as the period from Day -55 to Day 1.

Nominal Day referenced in the below Table 3-1 through Table 3-7 are the Study Day calculated from the date of first dose of MMB.

Table 3-1. Analysis Windows for Efficacy Endpoints MRI Spleen Volume Response Assessment and MRI Liver Iron Content

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline for MRI Spleen<br>Volume/Liver Iron Content | 1 | -30 | 1 |
| Week 24 <sup>a</sup> | 169 | 141 | 197 |

a Due to the challenge of scheduling the imaging scan, assessment after a subject rolls over to the GS-US-352-1154 study and satisfying the analysis window will:

- be used for the corresponding nominal visit, if no assessment prior to or on the date of the first dose of MMB in the GS-US-352-1154 study is available in the analysis window;
- not be used for the corresponding nominal visit, when there are assessments from the GS-US-352-1672 study, prior to or on the date of the first dose of MMB in the GS-US-352-1154 study, and satisfying the corresponding analysis window; instead assessments from GS-US-352-1672 will be used.

Table 3-2. Analysis Windows for Efficacy Analyses of TSS Response Rate at Week 24

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---|---|---|---|
| Baseline for TSS | 1 | -7 | -1 |
| Week 24 <sup>a</sup> | 169 | 28 days period with last day as Day 162. | 28 days period with last day as Day 176. |

a Last 28 consecutive days with ≥ 20 available daily TSS, with the last day of the 28 days period searched backward from the earliest date of "Upper limit" or the last participation date, through "Lower Limit", on days with non-missing Daily TSS.

Table 3-3. Analysis Windows for Hepcidin

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Baseline | -1 | -30 | -1 |
| Enrollment | 1 | 1 | 1 |
| Week 2 | 15 | 8 | 21 |
| Week 4 | 29 | 22 | 42 |
| Week 8 | 57 | 43 | 70 |
| Week 12 | 85 | 71 | 98 |
| Week 16 | 113 | 99 | 126 |
| Week 20 | 141 | 127 | 154 |
| Week 24 | 169 | 155 | 182 |

Table 3-4. Analysis Windows for Anemia Related Biomarkers<sup>a</sup>

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Baseline | 1 | -30 | 1 |
| Week 2 | 15 | 8 | 21 |
| Week 4 | 29 | 22 | 42 |
| Week 8 | 57 | 43 | 70 |
| Week 12 | 85 | 71 | 98 |
| Week 16 | 113 | 99 | 126 |
| Week 20 | 141 | 127 | 154 |
| Week 24 | 169 | 155 | 182 |

a Anemia related biomarkers include iron related biomarkers (iron, iron binding capacity, ferritin, non-transferrin bound iron, transferrin saturation, soluble transferrin receptor) and hematology biomarkers (hemoglobin, hematocrit, platelets, WBC, differential, reticulocyte count, % blasts, erythropoietin). For erythropoietin, observations will be assigned to different analysis windows from the rest of anemia related biomarkers.

Table 3-5. Analysis Windows for Erythropoietin

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Baseline | 1 | -30 | 1 |
| Week 8 | 57 | 29 | 85 |
| Week 20 | 141 | 113 | 169 |

Table 3-6. Analysis Windows for C-reactive Protein

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Baseline | 1 | -30 | 1 |
| Week 2 | 15 | 8 | 43 |
| Week 12 | 85 | 57 | 113 |
| Week 24 | 169 | 141 | 197 |

Table 3-7. Analysis Windows for Pharmacodynamics Biomarker pSTAT3

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Enrollment | 1 | 1 | 1 |
| Week 4 | 29 | 8 | 57 |
| Week 24 | 169 | 141 | 197 |

## 3.7.3. Selection of Data in the Event of Multiple Records in an Analysis Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple non-missing numeric observations exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last available record on or prior to the date of the first dose of MMB will be selected. If there are multiple records with the same time or no time recorded on the same day, average (arithmetic or geometric mean, as appropriate) will be used for the baseline value.
- For post-baseline visits:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken, unless otherwise specified.

If multiple valid non-missing categorical observations exist in a window, records will be selected as follows:

- For baseline, the last available record on or prior to the date of the first dose of MMB will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal for safety electrocardiogram [ECG] findings).
- For post-baseline visits, if there are multiple records with the same time or no time recorded on the same day, the most conservative value within the window will be selected (eg, abnormal will be selected over normal for safety ECG findings).

## 4. SUBJECT DISPOSITION

## 4.1. Subject Enrollment and Disposition

A summary of subject enrollment and disposition will be provided. This summary will present the number of subjects screened, the number of subjects rescreened, the number of subjects enrolled, and the number and percentage of subjects in each of the categories listed below. For the "Treated", the denominator for the percentage calculation will be the total number of subjects enrolled for each column. For all other categories, the denominator for the percentage calculation will be the total number of subjects in the Safety Analysis Set for each column.

- Screened
- Treated (Safety Analysis Set)
- Completed MMB
- Did not complete MMB with reason for premature discontinuation of MMB
- Completed the study
- Did not complete the study with reason for discontinuation of study
- Entered the roll over study of GS-US-352-1154
- Biomarker analysis.
- Pharmacokinetics analysis

In addition, the total number of subjects who were enrolled in the study and the number and percentage of subjects in each of the disposition categories listed above will be displayed in a flow chart.

The following by-subject listings will be provided by subject ID number in ascending order to support the above summary tables:

- Reasons for discontinuation of MMB or study
- Reasons for screen failure (will be provided by screening ID number in ascending order)
- Lot number and kit ID

#### 4.2. Extent of Exposure

Extent of exposure to MMB will be examined by assessing the total duration of exposure to MMB and the level of adherence to the MMB specified in the protocol.

# 4.2.1. **Duration of Exposure to MMB**

Total duration of exposure to MMB will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in MMB administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks).

When the stopping date of the study drug is missing or partial, the following rule will be used to impute the stopping date:

- If subjects are continuing on study drug, use the earliest of the date of death or data cutoff date or date of rolling over to GS-US-352-1154 study for analysis to impute the last dosing date for the calculation of the duration of exposure to study drug.
- If the stopping date is partial, then stopping date will be imputed with the earliest of the last date of the month (if month and year are available) or the last month of the year (if only year is available), the date of one day prior to the first dose in the rollover study, or the early study drug discontinuation date or date of death.

The total duration of exposure to MMB will be summarized using descriptive statistics (number of subjects [n], mean, StD, median, Q1, Q3, minimum, and maximum) and using the number (ie, cumulative counts) and percentage of subjects exposed through the following time periods:

```
Baseline (Day 1), Week 4 (Day 29), Week 8 (Day 57), Week 12 (Day 85), Week 16 (Day 113), Week 20 (Day 141), and Week 24 (Day 169).
```

Summaries will be provided for the Safety Analysis Set.

The number of subjects who have dose reduction or interruptions, and the reasons, will be summarized.

No inferential statistics will be provided.

#### 4.2.2. Adherence to MMB

The total number of tablets administered will be summarized using descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum).

The presumed total number of tablets administered to a subject will be determined by the data collected on the drug accountability CRF using the following formula:

```
Total Number of Tablets Administer ed = (\sum \text{No. of Tablets Dispensed}) - (\sum \text{No. of Tablets Not Administer ed})
```

where the number of tablets not administered is the sum of (a) the number of doses returned and (b) the number of (reported) missed tablets that were not returned.

If returned tablets were missing for the last dispensed bottle at the data cutoff date for subjects who were continuing on study drug, it will be assumed that these subjects had received the correct number of or tablets at the time of the data cutoff date.

The average daily dose (mg) will be calculated using the following formula:

Average Daily Dose (mg) = 
$$\frac{\sum (Daily Dose in mg)}{Total Number of Days on Study Drug}$$

Total Number of Days on Study Drug = Last Dosing Date – First Dosing + 1

The level of adherence with the MMB regimen while subjects were on treatment (i.e., on-treatment adherence) will be determined by the total amount of MMB administered relative to the total amount of MMB expected to be administered during subject's actual on-treatment period based on the MMB regimen.

The level of on-treatment adherence will be expressed in percentage using the following formula:

On - Treatment Adherence(%) = 
$$\left(\frac{\text{Total Amount of MMB Administered}}{\text{MMB Expected to Be Administered on Treatment}}\right) \times 100$$

Study drug expected to be administered on treatment (mg) is the dose (mg) prescribed, taking into account for dose reduction and interruption (ie, if dose reduced or interrupted for certain period, the dose expected to be administered should be the reduced dose level or 0mg if interrupted for that particular period) until the date of study drug withdrawn prematurely or completion.

Descriptive statistics for the level of on-treatment adherence (n, mean, StD, median, Q1, Q3, minimum, and maximum) with the number and percentage of subjects belonging to adherence categories (eg, <75%,  $\geq75$  to <90%,  $\geq90\%$ ) will be provided by treatment group for the Safety Analysis Set.

No inferential statistics will be provided.

A separate by-subject listing of MMB administration and MMB accountability will be provided by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of subjects who did not meet at least 1 entry criterion and the number of subjects who violated specific entry criteria based on all enrolled subjects. A by-subject listing will be provided for those subjects who violated at least 1 inclusion or exclusion criterion. The listing will present the entry criterion (or criteria if more than 1 violation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by deviation reason (eg, nonadherence to MMB, violation of inclusion/exclusion criteria) will be summarized for the all enrolled subjects. A by-subject listing will be provided for those subjects with any protocol deviation.

## 5. BASELINE CHARACTERISTICS

## 5.1. Demographics

Subject demographic variables (ie, age, sex, race, and ethnicity) will be summarized using descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum) for age, and using the numbers and percentages of subjects for gender, age (<65 yrs vs ≥65 yrs), race, and ethnicity. Age is calculated in years at the date of initial MMB administration. If a subject did not receive MMB after enrollment, the subject's age will be calculated from the date that the subject signed the informed consent form. The summary of demographic data will be provided for the Safety Analysis Set. Partial date of birth will be imputed per Section 5.3.2.1.

A by-subject demographic listing, which includes the date the informed consent was signed, will be provided by subject ID number in ascending order.

#### **5.2.** Other Baseline Characteristics

Other baseline characteristics include body weight (in kg), height (in cm), body mass index (BMI; in kg/m²), and disease and baseline characteristics will include type of MF (PMF, Post-PV MF, or post-ET MF), spleen volume(cm³), TSS, RBC units transfused within 8 weeks prior to enrollment, bone marrow fibrosis grade, cytogenetics findings, DIPSS risk level, hemoglobin level (continuous and categorical by <8 or  $\ge$ 8 g/dL), WBC (x10^3/uL), ANC (x10^3/uL), Platelet count (x10^3/uL), JAK2V617F mutation status (positive or negative) at baseline. These baseline characteristics will be summarized using descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum) for continuous variables and using the numbers and percentages of subjects for categorical variables. The summary of baseline characteristics will be provided for the Safety Analysis Set.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

## 5.3. Medical History

#### **5.3.1.** General Medical History

General medical history (ie, conditions not specific to the disease being studied) data will be collected at screening and listed only. A by-subject listing of general medical history will be provided by subject ID number in ascending order.

## 5.3.2. Myelofibrosis Disease History

Myelofibrosis disease history will be collected at screening for disease-specific conditions.

Time since disease diagnosis (years) will be calculated by (date of first dosing date of MMB - date of MF diagnosis + 1) / 365.25. Time since disease diagnosis will be summarized using summary statistics for a continuous variable. No inferential statistics will be generated.

Myelofibrosis disease type (PMF, post-PV MF, and post-ET MF) will be summarized by using number and percentage of subjects.

A by-subject listing of disease-specific conditions will be provided by subject ID number in ascending order.

# 5.3.2.1. Incomplete Dates

All partial dates of diagnosis and last regimen will be identified, and the partial dates will be imputed as follows:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.
- Partial date will not be imputed if the year is missing.

## 5.4. Myelofibrosis Disease-Specific Prior Therapy

Myelofibrosis disease-specific prior medication, defined as any medication for the purpose of treating MF disease with a start date that is prior to the enrollment, will be summarized by preferred term (PT) (collected through concomitant medication eCRF page) using the number and percentage of subjects on the medication. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by descending overall frequency of PT term. For drugs with the same frequency, sorting will be done alphabetically. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to or the same as the enrollment will be included in the prior medication summary. Medication with day, month and year all missing for start date will also be taken as MF disease-specific prior medication. All MF disease-specific prior medication will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

## 6. EFFICACY ANALYSES

# 6.1. Primary Efficacy Endpoint

## 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint of this study is transfusion independence (TI) response rate by Week 24 defined as becoming transfusion independent for  $\geq 12$  weeks at any time on study.

Twelve-week transfusion independent response by Week 24: ≥84 days transfusion independence response for subjects who are transfusion dependent at baseline, where transfusion dependent is defined as receiving at least 4 units of RBC transfusion in the 8 weeks prior to screening (or first dose of MMB). The subject will be considered as 12-week transfusion independent in post-baseline if at least 1 of the following 4 criteria is satisfied:

- 1) There is a time duration of at least 84 days between the first dose of MMB and the first RBC transfusion in post-baseline, where the duration will be calculated as follows:
  - Duration between the first dose of MMB to the first RBC transfusion in post-baseline (days) = Date of first RBC transfusion in post-baseline Date of first dose of MMB + 1
- 2) There is a time duration of at least 84 days between 2 consecutive RBC transfusions in post-baseline, where the duration will be calculated as follows:
  - Duration between the 2 consecutive RBC transfusions in post-baseline (days) = Date of the second RBC transfusion in the consecutive RBC transfusions in post-baseline Date of the first RBC transfusion in the successive RBC transfusions in post-baseline + 1
- 3) There is a time duration of at least 84 days between the last RBC transfusion in post-baseline and the last visit date, where the duration will be calculated as follows:
  - Duration between the last RBC transfusion in post-baseline and the last available visit in post-baseline (days) = Date of the last available visit in post-baseline Date of the last RBC transfusion in post-baseline + 1
- 4) No transfusion during the entire study in post-baseline and the length of the study is at least 84 days, where the duration will be determined as follows:
  - Duration between the date of first dose of MMB and the last available visit in post-baseline (days) = Date of the last available visit in post-baseline Date of the first dose of MMB + 1

Twelve-week transfusion independent response by Week 12: a subject is considered as 12-week transfusion independent by Week 12, if he did not have any transfusion in the first 84 days on study.

Any enrolled subject in the Safety Analysis Set who did not meet any of the criteria listed above will be considered a 12-week transfusion independent non-responder.

## Calculation of 12-week transfusion independent response rate by Week 24 and Week 12:

$$\hat{p}_{12-TF} = \\ 100 \times \frac{\textit{Number of patients with twelve-week transfusion independent response}}{\textit{Total number of enrolled patients in Safety Analysis Set}}$$

The denominator for calculation of the percentage of 12-week transfusion independent rate by Week 24 and Week 12 included all enrolled subjects in Safety Analysis Set.

## 6.1.2. Statistical Hypothesis for the Primary Efficacy Endpoint

There is no formal hypothesis testing in this study due to the exploratory nature of the primary end points.

## 6.1.3. Analysis of the Primary Efficacy Endpoint

The purpose of the primary analysis is to investigate the 12-week transfusion independence response rate by Week 24 with the treatment of MMB. In order to evaluate the proportion,  $\hat{p}_{12-TF}$ , a conventional 2-sided  $100(1-\alpha)\%$  exact confidence limits based on Clopper-Pearson method {Clopper 1934} for binominal distribution will be calculated, where  $\alpha$  is the confidence level. Unless otherwise indicated, it is equal to 0.10 in this study. Number and percent will be provided for subjects with or without Hgb < 8g/dL during 12-week transfusion-free window.

### **6.1.4.** Exploratory Analysis

An exploratory analysis will be performed to investigate the potential prognostic factors influencing transfusion independent response rate using the logistic regression model approach. The variables with prognostic potential will be included in the model to identify plausible significant factors on transfusion independent response rate:

- Age (< 65 years and  $\ge$  65 years)
- Gender (male and female)
- Race (white and all other races)
- DIPSS assessment (Intermediate-1/2 and high risk)
- Type of MF (PMF, Post-PV MF and Post ET MF)
- JAK2V617F mutation status at baseline (positive and negative)
- Hemoglobin level at baseline ( $\frac{8g}{dL}$  and  $\frac{8g}{dL}$ )

- TSS at baseline (<median and ≥median)
- Spleen volume at baseline (<median and ≥median)
- Hepcidin at baseline morning time point (<median and ≥median)
- Liver iron content at baseline (<median and ≥median)
- Transferrin saturation at baseline (<50% and  $\ge 50\%$ )

Each prognostic factor will be preliminarily evaluated in the logistic regression model. Only the variables with significance level less than 0.2 will be considered to build the multivariate model. A stepwise selection process with significance level of 0.2 for entering variables and significance level of 0.10 for keeping variables will be applied to those candidate variables to identify the final subset of relevant covariates in the logistic regression model.

# 6.1.4.1. Duration of TI Response (DOR-TI)

Duration of TI response is defined as the interval from the first onset date of TI response to the earliest onset date of loss of TI response or censoring date among subjects who achieved TI response, ie, duration of TI response (weeks) = (date of loss of TI response or censoring – date of first TI response + 1) / 7. The loss of TI response is defined as the date of the first transfusion post the TI response. Subjects who remain TI will be censored at the last participation date.

Duration of TI response will be summarized using Kaplan-Meier method for TI response by Week 24 only. Number of subjects with events and subjects censored, median, Q1, Q3, min and max estimates will be presented.

# 6.1.4.2. Time to TI Response (TtTI)

Time to TI response (TtTI) among subjects who achieved TI response is defined as the interval from the date of the first dose of MMB administration to the first onset date of TI response, ie, time to TI (weeks) = (the date of first TI response onset – date of the first dose of MMB + 1) / 7. No censoring is needed.

Time to TI response will be summarized only for TI response by Week 24 through descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum).

# 6.2. Secondary Efficacy Endpoints

## 6.2.1. Definition of Secondary Efficacy Endpoints

The following endpoints of this study are designated as secondary endpoints:

## 6.2.1.1. Transfusion Response Rate for $\geq$ 8 Weeks

Transfusion response for  $\geq 8$  weeks: defined as no RBC transfusions for at least 8 weeks at any time on study. A subject will be considered to achieve transfusion response for  $\geq 8$  weeks post-baseline if at least one of the following 2 criteria is satisfied:

(1) If there is no any transfusion event post-baseline and the length of study is  $\geq$  56 days.

Duration between dates in post-baseline = the last participant date - first dose date of MMB + 1.

(2) If there is any time interval between any 2 consecutive transfusion events post-baseline, or the time interval between the first dose of MMB date and the first transfusion date post-baseline, or the last transfusion date and the time interval between the last available visit date≥56 days

Duration between dates in post-baseline = later date - former date + 1.

# 6.2.1.2. Splenic Response Rate at Week 24

Splenic response rate at Week 24: defined proportion of subjects who achieve a  $\geq$  35% reduction in spleen volume at Week 24 (SRR24) from baseline as measured by MRI. The spleen volume will be obtained through the assessment of MRI scan by a central imaging laboratory described in the Section 6.2.11.2 in the protocol.

The baseline spleen volume is defined as the last spleen volume measured by MRI from the baseline period prior to or on the date of first dose of MMB administration (Day -30 to Day 1, Day 1 is defined as the day of first dose of MMB administration in the study).

The Week 24 spleen volume is defined as the spleen volume measurement by MRI at Week 24 (Day 141 to 197). When multiple records are existent between Day 141 and Day 197, the rules specified in Section 3.7.3 are applied. Due to the challenge of scheduling the imaging scan, assessment after the first MMB dose in the rollover study and between Day 141 to 197 for the subjects who were rolled over to Study GS-US-352-1154 will:

- Be used for Week 24 spleen volume, if no assessment prior to or on the date of the first rollover study MMB dosing and between Day 141 and Day 197 is available;
- Not be used for Week 24 spleen volume, if there are assessments in Study GS-US-352-1672, prior to or on the date of first rollover study MMB dosing and between Day 141 and Day 197; instead assessments in Study GS-US-352-1672 will be selected per rules specified in Section 3.7.3.

The %Change in spleen volume from baseline to Week 24 is calculated by:

$$\% change = 100 \times \frac{\textit{Week 24 Spleen Volume} - \textit{Baseline Spleen Volume}}{\textit{Baseline Spleen Volume}}$$

## 6.2.1.3. Response Rate of Total Symptom Score (TSS) at Week 24

The modified MPN-SAF TSS is an 8-item questionnaire developed to assess symptom burden and quality of life in patients with myeloproliferative neoplasms (MPNs). The TSS is assessed over time to evaluate changes in MPN-related symptoms. The modified MPN-SAF TSS is completed daily on an electronic diary (eDiary) device. NOTE: scores for the question of inactivity in the diary will not be included in TSS assessments.

The proportion of subjects who have achieved  $\geq 50\%$  reduction from baseline to Week 24 in TSS based on the modified MPN-SAF TSS will be determined as follows.

The diary is completed at the end of each day with a 24-hour recall period, and the daily TSS is defined as the sum of 7 individual symptom scores (each with a 0 to 10 point scale) collected on the same day. The daily TSS will be missing if there are any missing individual scores. If multiple records are available on the same day, the last record will be used as an assessment for that day.

The baseline TSS is defined as the average of the daily TSS from the 7-day baseline period (Day -7 through Day -1). The baseline TSS will be missing if there are more than 3 days of missing daily TSS during the 7-day baseline period.

The Week 24 TSS is defined as the average of the daily TSS from a consecutive 28-day period at Week 24. The consecutive 28-day period at Week 24 is defined as the latest eligible period of 28 consecutive days that has  $\geq$  20 available daily TSS; the last day of that 28-day period must be prior to or on the last participation date, have nonmissing daily TSS, and fall between Days 162 and 176, inclusive. If no such consecutive 28-day period with  $\geq$  20 available daily TSS is available or the last participation day was prior to Day 162, the Week 24 TSS will be considered missing.

The percentage change in TSS from baseline to Week 24 is calculated as follows:

### 6.2.1.4. Change in Hepcidin

Hepcidin is measured twice at each study visit, one predose in the morning and one 6 hours postdose. Hepcidin is measure at the Baseline Visit (both morning and 6 hour samples are predose), at the Enrollment Visit and Weeks 2, 4, 8, 12, 16, and 24. Change and % change from baseline will calculated for predose and postdose values, respectively. Hepcidin value is obtained through the assessment by hepcidin analysis (Radbound).

The baseline visit for hepcidin is defined as the last visit in the baseline period prior to the date of first dose of MMB administration (Day -30 to Day -1, Day 1 is defined as the day of first dose of MMB administration in the study). Hepcidin value at predose time point in the morning at the baseline visit will be used as the baseline value for predose hepcidin measurement. Hepcidin value at 6 hours postdose at the baseline visit will be used as the baseline value for 6 hours postdose hepcidin measurement.

The post-baseline visits for hepcidin are defined using the analysis window specified in Section 3.7.2. Predose value and 6 hours postdose value at each post-baseline visit will be used to calculate the change and % change from baseline for hepcidin measured at predose time point and 6 hours postdose.

Daily hepcidin change will also be calculated at each study visit using the formula below:

Daily hepcidin change = 6 hours postdose hepcidin value - predose hepcidin value

Daily hepcidin change at the baseline visit will be used as the baseline value for daily hepcidin change. Daily hepcidin change at post-baseline visits is defined by the analysis window specified in Section 3.7.2. Change and % change from baseline of daily hepcidin change will be calculated.

## 6.2.1.5. Baseline and Change in Anemia Related Biomarkers

Change and % change from baseline will be calculated for anemia related biomarkers, including iron related biomarkers (iron, iron binding capacity, ferritin, non-transferrin bound iron, transferrin saturation, and soluble transferrin receptor) and hematology biomarkers (hemoglobin, hematocrit, platelets, WBC, RBC, reticulocyte count, reticulocyte/erythrocyte %, % blasts, and erythropoietin). The values of these biomarkers are obtained from the central laboratory assessment as described in Protocol Section 6.2.7

The baseline biomarker value is defined as the last value from the baseline period prior to or on the date of first dose of MMB administration (Day -30 to Day 1, Day 1 is defined as the day of first dose of MMB administration in the study).

The post-baseline biomarker value is defined as the value measured within the analysis windows of post-baseline visits specified in Section 3.7.2. When multiple records are in the analysis window of a post-baseline visit, the rules specified in Section 3.7.3 are applied.

#### 6.2.1.5.1. Anemia Related Biomarker for TI Responders

For TI responders, change and % change from pre-TI response will be calculated for anemia related biomarker values during the period of TI response. Anemia related biomarker for this analysis include predose hepcidin, hepcidin 6 hour postdose, hepcidin daily change, iron, iron binding capacity, ferritin, non-transferrin bound iron, transferrin saturation, soluble transferrin receptor, hemoglobin, hematocrit, platelets, WBC, RBC, reticulocyte count, reticulocyte/erythrocyte %, % blasts, and erythropoietin.

The pre-TI response anemia biomarker value is defined as the last value prior to the start of the TI response window defined in Section 6.1.1. Anemia related biomarker values used for pre-TI response and during the period of TI response should be chosen from the baseline and post-baseline anemia related biomarker values defined above, and change and % change from pre-TI response will be calculated at 2 weeks, 4 weeks, 8 weeks, 12 weeks etc., after the pre-TI response anemia related biomarker value.

## 6.2.1.6. Change in Liver Iron Content

Change and % change from baseline will be calculated for liver iron content. The liver iron content is obtained from the central imaging laboratory MRI assessment described in Protocol Section 6.2.8.2.

The baseline liver iron content is defined as the last value from the baseline period prior to or on the date of first dose of MMB administration (Day -30 to Day 1, Day 1 is defined as the day of first dose of MMB administration in the study).

The Week 24 liver iron content is defined as the value measured within the analysis window of the Week 24 visit specified in Section 3.7.2. When multiple records are in the analysis window of a post-baseline visit, the rules specified in Section 3.7.3 are applied.

#### 6.2.1.7. Change in C-reactive Protein

Change and % change from baseline will be calculated for C-reactive protein. The value of C-reactive protein is obtained from the central laboratory assessment described in Protocol Section 6.2.7.

The baseline C-reactive protein value is defined as the last value from the baseline period prior to or on the date of first dose of MMB administration (Day -30 to Day 1, Day 1 is defined as the day of first dose of MMB administration in the study).

The post-baseline C-reactive protein value is defined as the value measured within the analysis window of post-baseline visits specified in Section 3.7.2. When multiple records are in the analysis window of a post-baseline visit, the rules specified in Section 3.7.3 are applied.

#### 6.2.1.8. Change in Pharmacodynamics Biomarker pSTAT3

Change and % change from baseline will be calculated for the pharmacodynamics biomarker pSTAT3, including %pSTAT Stimulated CD3+/4+ T cell and ratio between %pSTAT Stimulated CD3+/4+ T cell and %tSTAT Stimulated CD3+/4+ T cell. Ratio between %pSTAT Stimulated CD3+/4+ T cell and %tSTAT Stimulated CD3+/4+ T cell is calculated as 100%× (%pSTAT Stimulated CD3+/4+ T cell ÷ %tSTAT Stimulated CD3+/4+ T cell). pSTAT3 is measured at time points of predose, 2, 4 and 6 hour postdose at Enrollment, Week 4 and 24. The value of pSTAT3 is obtained from the central laboratory assessment described in Protocol Section 6.2.

The baseline pSTAT3 value is defined as the last predose value from the baseline period prior to or on the date of first dose of MMB administration (Day -30 to Day 1, Day 1 is defined as the day of first dose of MMB administration in the study).

The Week 4 and 24 pSTAT3 values are defined as values measured within the analysis windows of the Week 4 and 24 visits specified in Section 3.7.2. When multiple records are in the analysis window of a post-baseline visit, the rules specified in Section 3.7.3 are applied.

## 6.2.2. Analysis Methods for Secondary Efficacy Endpoints

Similar with the analysis method for the primary efficacy endpoint, the primary analyses of all of the secondary efficacy endpoints will be conducted using the Safety Analysis Set.

#### 6.2.2.1. Transfusion Response Rate $\geq 8$ weeks

Calculation of the transfusion response rate by Week 24:

$$\hat{p}_{8-TF} = 100 \times \frac{Number\ of\ Responders}{Total\ number\ of\ enrolled\ subjects\ in\ the\ Safety\ Analysis\ Set}$$

The denominator for calculation of the transfusion response rate by Week 24 includes all enrolled subjects in Safety Analysis Set.

The proportion,  $\hat{p}_{8-TF}$ , with a conventional 2-sided  $100(1-\alpha)\%$  exact confidence limits based on Clopper-Pearson method for binominal distribution will be calculated.

# 6.2.2.2. Splenic Response Rate at Week 24

Calculation of the splenic response rate at Week 24:

$$\hat{p}_{spleen} =$$

The denominator for calculation of the splenic response rate at Week 24 includes all enrolled subjects in Safety Analysis Set.

If spleen volume of a subject was not assessed by MRI scan between Study Day -30 and Day 1 (including Day 30 and Day 1), the subject will be coded as a non-responder of splenic response. Subjects who discontinue from the treatment before Week 24 and miss the Week 24 spleen volume measurement will also be considered as a non-responder.

The proportion,  $\hat{p}_{spleen}$ , with a conventional 2-sided  $100(1-\alpha)\%$  exact confidence limits based on Clopper-Pearson method for binominal distribution will be calculated.
## 6.2.2.3. Response Rate in TSS

Calculation of the TSS response rate at Week 24:

$$\hat{p}_{TSS} = 100 \times$$

## Number of subjects with ≥ 50% TSS reduction at week 24

Total number of enrolled subjects with non-missing baseline TSS in the Safety Analysis Set

Response rate in TSS at Week 24 will be analyzed for subjects who have a baseline TSS > 0 or subjects who have a baseline TSS = 0 but nonzero or missing TSS at Week 24. Subjects with missing Week 24 TSS will be considered as non-responders.

The proportion,  $\hat{p}_{TSS}$ , with a conventional 2-sided  $100(1-\alpha)\%$  exact confidence limits based on Clopper-Pearson method for binominal distribution will be calculated.

#### 6.2.2.4. Change in Hepcidin

Descriptive summary statistics will be provided for actual value, change, and % change from baseline for hepcidin measured at predose and 6 hours postdose of each study visit by TI response. Exploratory plots, such as median-IQR plot of hepcidin value by visit and TI response, may be provided.

A linear mixed effects model may be fitted to change from baseline for hepcidin with visit, time point, and TI response as the fixed effects and subject as the random effects. Least square mean estimate and 2-sided  $100(1-\alpha)\%$  confidence intervals (CI) will be calculated for change from baseline of hepcidin at the predose and 6 hour postdose time point at each post-baseline study visit. If necessary, log transformation may be applied to hepcidin value.

Descriptive summary statistics will be provided for daily hepcidin change, change, and % change from baseline for daily hepcidin change by study visit and TI response. Exploratory plots, such as median-IQR plot of % change from baseline of daily hepcidin change by visit and TI response, may be provided.

A linear mixed effect model may be fitted to change from baseline for daily hepcidin change with visit and TI response as the fixed effects and subject as the random effects. Least square means and 2-sided  $100(1-\alpha)\%$  confidence intervals (CI) will be calculated for change from baseline of daily hepcidin change at each post-baseline study visit. If necessary, log transformation may be applied to daily hepcidin change.

#### 6.2.2.5. Baseline and Change in Anemia Related Biomarkers

Descriptive summary statistics will be provided for actual value, change, and % change from baseline of anemia related biomarkers by visit and TI response. Exploratory plots, such as median-IQR plot of % change from baseline of anemia related biomarkers by visit and TI response, may be provided.

## 6.2.2.6. Change in Liver Iron Content

Descriptive summary statistics will be provided for actual value, change, and % change from baseline of liver iron content by visit and TI response.

## 6.2.2.7. Change in C-reactive Protein

Descriptive summary statistics will be provided for actual value, change, and % change from baseline of C-reactive protein by visit and TI response. Exploratory plots, such as median-IQR plot of % change from baseline of C-reactive protein by visit and TI response, may be provided.

## 6.2.2.8. Change in Pharmacodynamics Biomarker pSTAT3

Descriptive summary statistics will be provided for actual value, change, and % change from baseline of pSTAT3 at each time point and visit. Exploratory plots, such as median -IQR plot of % change from baseline of pSTAT3 by visit may be provided.

## 6.3. Exploratory Efficacy Endpoint

### 6.3.1. Definition of Exploratory Efficacy Endpoints

#### 6.3.1.1. Duration of TI Response (DOR-TI)

Duration of TI response is defined as the interval from the first onset date of TI response to the earliest onset date of loss of TI response or censoring date among subjects who achieved TI response, ie, duration of TI response (weeks) = (date of loss of TI response or censoring – date of first TI response + 1) / 7. The loss of TI response is defined as the date of the first transfusion post the TI response. Subjects who remain TI will be censored at the last participation date.

Duration of TI response will be summarized using Kaplan-Meier method. Number of subjects with events and subjects censored, median, Q1, Q3, and min and max estimates will be presented.

## 6.3.1.2. Time to TI Response (TtTI)

Time to TI response (TtTI) among subjects who achieved TI response is defined as the interval from the date of the first dose of MMB administration to the first onset date of TI response, ie, time to TI (weeks) = (the date of first TI response onset – date of the first dose of MMB + 1) / 7. No censoring is needed

Time to TI response will be summarized through descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum).

#### 6.3.1.3. Leukemia-Free Survival

Leukemia-free survival (LFS) is defined as the interval first dose date to the date of first documented leukemic transformation or death from any cause, ie, LFS (weeks) = (date of censoring or date of earliest of leukemic transformation or death – first dose date + 1) / 7. Leukemic transformation was documented in long-term follow up and AE eCRF page. Leukemic transformation related AE PTs are listed in Appendix 6.

#### 6.3.1.4. Bone Marrow Fibrosis Score

Bone marrow fibrosis improvement is reduction in bone marrow fibrosis score by one or more than one grade.

### 6.3.2. Analysis Methods for Exploratory Efficacy Endpoints

Time to event endpoints will be summarized using Kaplan-Meier method, with exception that TtTI will be summarized through descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum). Number and percentage of subjects with events and censored subjects, medians and ranges of survival time will be presented. A plot of the Kaplan-Meier curves will be provided. Censoring for each time to event endpoints was specified in Section 3.6.3.

For bone marrow fibrosis score, number and percentage of subjects in each grade will be provided. Number and percentage of subjects whose bone marrow fibrosis improved to grade 0 from baseline bone marrow fibrosis greater than grade 0 will also be provided. Improving rate defined as proportion of subjects with bone marrow fibrosis improvement among subjects with non-missing baseline bone marrow fibrosis score will be calculated, a conventional 2-sided  $100(1-\alpha)\%$  exact confidence limits based on Clopper-Pearson method for binominal distribution will be calculated, where  $\alpha$  is the confidence level.

Corresponding listings will be provided.

### 6.4. Changes From Protocol-Specified Efficacy Analyses

Pharmacokinetics parameters (C<sub>max</sub>, C<sub>last</sub>, C<sub>tau</sub> and AUC<sub>last</sub>, if available) for MMB mentioned in Protocol Section 8.1.3 have been removed as an analysis endpoint in the SAP due to the sparse PK samples collection.

Change in circulating cytokine and inflammatory markers (eg, IL-6, IL-8, IFN-gamma, TNF-alpha) have been removed as an analysis endpoint in the SAP.

The following exploratory endpoints have been removed as analysis endpoints in the SAP

- Baseline and change in markers of orthogonal or parallel signaling pathways (eg, RAS/MAPK, PI3K/AKT)
- Baseline and change in gene expression profiles in whole blood and somatic mutations in whole blood, if applicable.
- Baseline and change in immune subsets in whole blood
- Change in exploratory pharmacodynamics markers of signaling mediated by JAK1 and/or JAK2 (eg, pSTAT1, pSTAT5, and pSTAT6)

## 7. SAFETY ANALYSES

### 7.1. Adverse Events and Deaths

### 7.1.1. Adverse Event Dictionary

Clinical and laboratory adverse events (AEs) will be coded using the current version of MedDRA. System organ class (SOC), preferred term (PT) will be provided in the AE dataset.

## 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), or 5 (fatal) according to the Common Terminology Criteria for Adverse Events [CTCAE] Version 4.03. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

## 7.1.3. Relationship of Adverse Events to MMB

Related AEs are those for which the investigator selected "Related" on the AE case report form (CRF) to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationships to MMB will be considered related to MMB for summary purposes. However, by-subject data listings will show the relationship as missing from that captured on the CRF.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definition of an SAE specified in the study protocol. Serious adverse events captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health Department before database finalization.

#### 7.1.5. Treatment-Emergent Adverse Events

## 7.1.5.1. Definition of Treatment Emergent

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the MMB start date and no later than 30 days after permanent discontinuation of MMB.
- Any AEs leading to premature discontinuation of MMB.

## 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and AE stop date is not prior to the first dosing date of MMB, the month and year (or year alone if month is missing too) of onset determine whether an AE is treatment emergent. The AE is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset is the same as or after the month and year (or year) of the first dosing date of MMB, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of MMB.

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of MMB, will be considered to be treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

A brief high-level summary of TEAEs will be provided by the number and percentage of subjects who had the following: any AE; any AE of Grade 3 or above; any treatment-related AE; any treatment-related AE of Grade 3 or above; any SAE; any treatment-related SAE; any AE that led to premature discontinuation of MMB; and any AE that led to premature discontinuation of study; and any AE of interest. All deaths (including those that are treatment emergent and those that are not treatment emergent) observed will also be summarized and included in this table.

Adverse event summaries will provide the number and percentage of subjects with TEAEs by SOC, PT and Severity, using the Safety Analysis Set as follows:

- All AEs (by SOC, PT and Severity)
- All AEs of Grade 3 or above
- All treatment-related AEs
- All treatment-related AEs of Grade 3 or above
- All SAEs
- All treatment-related SAEs
- All AEs leading to premature discontinuation of MMB
- All AEs leading to a temporary interruption of MMB
- All AEs leading to a dose reduction of MMB

- All AEs leading to death (i.e., outcome of death)
- All AEs of interest
  - Peripheral Neuropathy SMQ (narrow terms only)
  - Cataract

First Dose Effect AE (defined as AE with PT of Dizziness, Flushing, Hot Flush, Headache, Hypotension, or Nausea, which occurred on the day of the first dosing date and resolved by the next day)In addition, all AEs recorded between screening and first dose of study drug will also be summarized for the Safety Analysis Set.

Multiple events will be counted only once per subject in each summary. The AEs will be summarized and listed first by SOC in descending order of incidence and then by PT, also in descending order of incidence, within each SOC of the investigational MMB group. For summaries by severity, the most severe grade will be used for those AEs that occurred in a given subject more than once during the study.

In addition to the presentation by SOC and PT, summaries will also be presented by PT only, ordered by decreasing total frequency for TEAEs that occurred in at least 5% of subjects within any treatment group, treatment-related TEAEs leading to discontinuation of IPs; TEAEs leading to dose modification or interruption of IP; treatment-emergent SAEs; and TEAEs of Grade >= 3 or above.

Summary of all TEAEs will also be presented by SOC, and PT for the following subgroups: gender (Male or Female), age group (<65 or >=65 years) and race (White or Non-White).

In addition to the summaries described above, data listings will be provided for the following:

- All AEs (with a variable indicating whether the event is treatment emergent)
- All AEs of Grade 3 or above
- SAEs
- Deaths
- All SAEs leading to death
- AEs leading to premature discontinuation of study drug
- AEs leading to premature discontinuation of study
- AEs leading to Dose interruption or modification of study drug

- AE related to study drug
- AEs of interest
  - Peripheral Neuropathy SMQ (narrow terms only)
  - Cataract
  - First Dose Effect

## 7.1.7. Additional Analysis of Adverse Events

## 7.1.7.1. Exposure-Adjusted Treatment-Emergent Adverse Events Rate

The exposure-adjusted TEAE rate is defined as the number of subjects with a specific event divided by the total exposure-time among the subjects in the treatment group and at risk of an initial occurrence of the event. Specifically,

$$Exposure - Adjusted TEAE Rate = \frac{n}{\sum t_i}$$

where n is the number of subjects with events;  $t_i$  is the interval (years) from first dosing date of study drug to the onset of first event for subjects with events, or will be censored at the time of the last participation date, or death date, or data cut-off date, whichever is earliest for subjects without events.

The exposure-adjusted TEAE rate will be summarized for all TEAEs, SAEs,  $\geq$  Grade 3 AEs.

## 7.1.7.2. Time to Onset of AE of Interest (Peripheral Neuropathy TEAEs)

Time to onset of AE of interest is defined as the interval from the first dose of study drug to the onset date of the first event of the AE of interest, ie, calculated as (the onset date of the first event of the AE of interest or censoring date – date of the first dose of study drug + 1). In the absence of the occurrence of the AE of interest, the censoring date is the last participation date, or death date, or data cut-off date, whichever is earliest for subjects without events.

Summary and Kaplan-Meier plot will be provided for peripheral neuropathy TEAEs (narrow term only).

### 7.1.7.3. Time to Resolution of AE of Interest (Peripheral Neuropathy TEAEs)

Time to resolution of AE of interest is defined as the interval from the onset date of the first event of the AE of interest to the time that the last event of the AE of interest is resolved, ie, calculated as (the resolution date of the last event of the AE of interest or censoring date – the onset date of the first event of the AE of interest + 1). In the absence of the resolution of the AE of interest, the censoring date is the last participation date, or death date, or data cut-off date, whichever is earliest.

Summary and Kaplan-Meier plot will be provided for peripheral neuropathy TEAEs (narrow term only).

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set. The analysis will be based on values reported in conventional units. When values are below the limit of quantitation, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics. Hemolyzed test results will not be included in the analysis, but they will be listed in by-subject laboratory listings.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, urinalysis and thiamine separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the CTCAE severity grade will be flagged in the data listings, as appropriate.

No inferential statistics will be generated.

## 7.2.1. Graded Laboratory Values

CTCAE Version 4.03 will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis except for anemia (hemoglobin, Hgb) which will be graded using the CTCAE Version 3.0 as defined in Table 7-1. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. Some laboratory tests have criteria for both increased and decreased levels; analyses for each direction (i.e., increased, decreased) will be presented separately.

Table 7-1. Grading of Hemoglobin Severity

| Grade (CTCAE 3.0) | | | | |
|---|---|---|---|---|
| 1 2 3 4 5 | | | | |
| <lln 10.0="" dl<="" g="" td="" –=""><td>&lt;10.0 – 8.0 g/dL</td><td>&lt;8.0 – 6.5 g/dL</td><td>&lt;6.5 g/dL</td><td>Death</td></lln> | <10.0 – 8.0 g/dL | <8.0 – 6.5 g/dL | <6.5 g/dL | Death |
| <LLN $-6.2 mmol/L$ | <6.2 – 4.9 mmol/L | <4.9 – 4.0 mmol/L | <4.0 mmol/L | |
| <LLN $- 100 g/L$ | <100 – 80 g/L | <80 – 65 g/L | <65 g/L | |

## 7.2.1.1. Treatment-Emergent (TE) Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any post-baseline time point, up to and including the date of last dose of MMB plus 30 days for subjects who permanently discontinued MMB. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

## 7.2.1.2. Treatment-Emergent Marked Laboratory Abnormalities

Treatment-emergent marked laboratory abnormalities are defined as values that increase from baseline by at least 3 toxicity grades at any post-baseline time point, up to and including the date of the last dose of MMB plus 30 days for subjects who permanently discontinued MMB. If the relevant baseline laboratory value is missing, any Grade 3 or 4 values observed within the timeframe specified above will be considered treatment-emergent marked abnormalities.

## 7.2.1.3. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test; subjects will be categorized according to the most severe post-baseline abnormality grade for a given lab test:

- All laboratory abnormalities
- Grade 3 or 4 laboratory abnormalities
- Marked laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing post-baseline values.

A by-subject listing of treatment-emergent Grade 3 or 4 laboratory abnormalities or marked laboratory abnormalities, if abnormalities were not graded will be provided by subject ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades or abnormal flags displayed.

#### 7.2.2. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in CTCAE severity grade from baseline to the worst grade post-baseline grade. For lab tests for which a severity scale does not exist, shift tables will be presented showing change in results from baseline value (low, normal and high) to the worst post-baseline value (low, normal, high and "high & low", where "high & low" is for lab tests with both high and low values at post-baseline visits).

### 7.3. Body Weight

Descriptive statistics (n, mean, StD, median, Q1, Q3, minimum, and maximum) will be provided for body weight as follows:

- Baseline value
- Values at each post-baseline time point
- Change from baseline at each post-baseline time point

- Post-baseline maximum value
- Change from baseline to post-baseline maximum value
- Post-baseline minimum value
- Change from baseline to post-baseline minimum value

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose of MMB. Change from baseline to a post-baseline visit will be defined as the post-baseline value minus the baseline value. Body weight measured at unscheduled visits will be included for the baseline and post-baseline maximum and minimum value selection.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.7.3. No inferential statistics will be generated.

Body weight will be summarized by grade, where grade is defined as follows:

The maximum grade of post-baseline weight gain and weight loss will be calculated and summarized based on the below table per CTCAE 4.03:

| Post-baseline Maximum Grade of<br>Weight Gain or Weight Loss | Grade | Criteria for Grade |
|---|---|---|
| Weight Gain | 0 | maximum % change from baseline < 5% |
| | 1 | 5% ≤ maximum % change from baseline < 10% |
| | 2 | 10% ≤ maximum % change from baseline < 20% |
| | 3 | maximum % change from baseline $\geq 20\%$ |
| Weight Loss | 0 | -5% < minimum % change from baseline |
| | 1 | -10% < minimum % change from baseline ≤ -5% |
| | 2 | -20% < minimum % change from baseline ≤ -10% |
| | 3 | minimum % change from baseline ≤ -20% |

#### 7.4. Prior and Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary. The medications will be categorized as prior, concomitant, or both using the following definitions:

- Prior medications: any medications taken and stopped prior to or on the initial MMB dosing date based on the Prior and Concomitant Medication eCRF page
- Concomitant medications: any medications taken after the initial MMB dosing date and up to the last dosing date of MMB

#### 7.4.1. Prior Medications and Concomitant Medications

Prior medications and concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2, Level 4 and preferred name using the number and percentage of subjects for each treatment group and overall. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by descending overall frequency of ATC drug classes and then by preferred names within an ATC drug class of the MMB treatment. For drugs with the same frequency, sorting will be done alphabetically.

Summaries will be based on the Safety Analysis Set. No inferential statistics will be generated.

For purposes of analysis, any medication with a stop date that is prior to or on the initial MMB dosing date will be included in the prior medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the initial MMB dosing date will be included in the prior medication summary.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

## 7.5. Electrocardiogram Results

Electrocardiogram (ECG) data will not be presented in the CSR since ECGs were not assessed in this study other than as part of the screening process for potential new subjects.

## 7.6. Other Safety Measures

## 7.6.1. Overall Survival (OS)

OS, for subjects who died while on study, is defined as the interval from the date of the first dose of study drug to the date of the death from any cause, ie, the date of death—the first dose date +1.

Data from surviving subjects (ie. subjects who do not die while on study) will be censored at the last date that subject was known to be alive, ie, the last study participation date.

Overall survival will be summarized using the Kaplan-Meier method. A plot of the Kaplan-Meier curves will be provided. Number and percentage of subjects with events and censored subjects, medians and ranges of survival time will be presented.

A listing of overall survival will also be provided.

## 8. PHARMACOKINETIC ANALYSES

The concentration data of MMB and major metabolite GS-644603, will be listed and summarized by nominal sampling time using descriptive statistics by study visit if applicable. Summary statistics (n, mean, StD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented.

Individual concentration data listings and summaries will include all subjects with concentration data. The sample size for each time point will be based on the number of subjects with nonmissing concentration data at that time point. The number of subjects with concentration BLQ will be presented for each time point.

The following tables will be provided for each analyte:

• Individual subject concentration data and summary statistics

The following figures may be provided for each analyte by visit:

- Mean (± StD) concentration data versus time (on linear and semilogarithmic scales)
- Median (Q1, Q3) concentration data versus time (on linear and semilogarithmic scales)
- Individual, mean, and median postdose concentration values that are ≤ LLOQ will not be displayed in the figures and remaining points connected.

The following listings will be provided:

 PK sampling details by subject including deviations in scheduled and actual draw times and procedures

## 9. REFERENCES

Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Dec. Biometrika 1934;26 (4):pp. 404-13.

## 10. SOFTWARE

SAS® Software Version 9.2. SAS Institute Inc., Cary, NC, USA.

nQuery Advisor(R) Version X.0. Statistical Solutions, Cork, Ireland.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

## 12. APPENDICES

| Appendix 1. | Table of Contents for Statistical Tables, Figures, and Listings |
|---|---|
| Appendix 2. | Study Procedures Table |
| Appendix 3. | Peripheral Neuropathy SMQ AEs |
| Appendix 4. | Cataract MST AEs |
| Appendix 5. | Leukemic Transformation MST AEs |
| Appendix 6. | Validation document of hepcidin testing from Radboud University |
| Appendix 7. | Validation document of pSTAT testing from Covance |

## **Appendix 1.** Table of Contents for Statistical Tables, Figures, and Listings

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 15.8.1.1 | Enrollment by Country, Region and Investigator | Safety Analysis Set | |
| 15.8.1.2 | Subject Disposition | Safety Analysis Set | |
| 15.8.2.1 | Eligibility Criteria Deviations | Safety Analysis Set | |
| 15.8.2.2 | Important Protocol Deviations | Safety Analysis Set | |
| 15.8.3.1 | Demographics | Safety Analysis Set | |
| 15.8.3.2 | Baseline Characteristics | Safety Analysis Set | |
| 15.8.3.3 | Prior Myelofibrosis Therapy | Safety Analysis Set | |
| 15.8.3.4 | Myelofibrosis Disease History | Safety Analysis Set | |
| 15.8.4 | Adherence to Study Drug Regimen | Safety Analysis Set | |
| 15.8.5 | Analysis Sets | Safety Analysis Set | |
| 15.10.1 | Summary of Plasma Concentration of MMB and GS-644603 | Pharmacokinetic<br>Analysis Set | |
| 15.11.1 | Extent of Exposure to Study Drug | Safety Analysis Set | |
| 15.11.2.1.1 | TEAEs: Overall Summary | Safety Analysis Set | |
| 15.11.2.1.2 | Exposure-Adjusted TEAEs: Overall Summary | Safety Analysis Set | |
| 15.11.2.1.3.1 | TEAEs by PT Occurred in >=5% of Subjects | Safety Analysis Set | |
| 15.11.2.1.3.2 | Exposure-Adjusted TEAEs by PT | Safety Analysis Set | |
| 15.11.2.1.4.1 | TEAEs by SOC, PT, and Severity by Gender | Safety Analysis Set | |
| 15.11.2.1.4.2 | TEAEs by SOC, PT, and Severity by Age Group | Safety Analysis Set | |
| 15.11.2.1.4.3 | TEAEs by SOC, PT, and Severity by Race | Safety Analysis Set | |
| 15.11.2.2.1 | TEAEs by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.2.2.2.1 | TEAEs with Severity of Grade 3 or 4 by PT | Safety Analysis Set | |
| 15.11.2.2.2.2 | TEAEs with Severity of Grade 3 or 4 by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.2.2.2.3 | Exposure-Adjusted TEAEs with Severity of Grade 3 or Above by PT | Safety Analysis Set | |
| 15.11.2.3 | Treatment-Related TEAEs with Severity of Grade 3 or Above by PT | Safety Analysis Set | |
| 15.11.2.4.1 | TEAE Leading to Dose Reduction or Temporary<br>Interruption of Study Drug (MMB) by SOC, PT,<br>and Severity | Safety Analysis Set | |
| 15.11.2.4.2.1 | TEAE of Peripheral Neuropathy SMQ (Narrow<br>Terms only) by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.2.4.2.2 | TEAE of Cataract MST by SOC, PT, and Severity | Safety Analysis Set | |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 15.11.2.4.3.1 | Time to Onset of First Peripheral Neuropathy SMQ (Narrow Term Only) | Safety Analysis Set | |
| 15.11.2.4.3.2 | Time to Resolution of Peripheral Neuropathy SMQ (Narrow Term Only) | Safety Analysis Set | |
| 15.11.2.4.4 | TEAEs for First Dose Effect by PT | Safety Analysis Set | |
| 15.11.3 | TEAEs Leading to Death by SOC,PT and Severity | Safety Analysis Set | |
| 15.11.4.1.1 | Serious TEAEs by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.4.1.2 | Serious TEAEs by PT | Safety Analysis Set | |
| 15.11.4.1.3 | Exposure-Adjusted Serious TEAEs by PT | Safety Analysis Set | |
| 15.11.4.2 | Treatment-Related Serious TEAEs by PT | Safety Analysis Set | |
| 15.11.4.3 | Serious TEAEs for First Dose Effect by PT | Safety Analysis Set | |
| 15.11.5.1.1 | TEAE Leading to Premature Discontinuation of<br>Study Drug (MMB) by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.5.1.2 | TEAE of Peripheral Neuropathy SMQ (Narrow<br>Term Only) Leading to Study Drug (MMB)<br>Discontinuation by SOC, PT, and Severity | Safety Analysis Set | |
| 15.11.6.1 | Hematology: Shift from Baseline for Gradable<br>Tests | Safety Analysis Set | |
| 15.11.6.2 | Chemistry: Shift from Baseline for Gradable Tests | Safety Analysis Set | |
| 15.11.6.3 | Urinalysis: Shift from Baseline for Gradable Tests | Safety Analysis Set | |
| 15.11.6.4.1 | Treatment-Emergent Laboratory Abnormalities | Safety Analysis Set | |
| 15.11.6.4.2 | Treatment-Emergent Grade 3 or 4 Laboratory<br>Abnormalities | Safety Analysis Set | |
| 15.11.6.4.3 | Treatment-Emergent Marked Laboratory<br>Abnormalities | Safety Analysis Set | |
| 15.11.6.4.4 | Exposure-Adjusted Treatment-Emergent<br>Laboratory Abnormalities | Safety Analysis Set | |
| 15.11.6.4.5 | Exposure-Adjusted Treatment-Emergent Marked<br>Laboratory Abnormalities | Safety Analysis Set | |
| 15.11.7.1 | Body Weight (kg) Change and % Change from Baseline | Safety Analysis Set | |
| 15.11.7.2 | Summary of Change of Body Weight (kg) from Baseline by Grade | Safety Analysis Set | |
| 15.11.8.1 | Prior Medications by Drug Class and Preferred<br>Drug Name | Safety Analysis Set | |
| 15.11.8.2 | Concomitant Medications by Drug Class and<br>Preferred Drug Name | Safety Analysis Set | |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 15.12.1.1 | Analysis of Transfusion Independent Response<br>Rate by Week 24 and Week 12 | Safety Analysis Set | |
| 15.12.1.2 | Exploratory Analysis of Transfusion Independent<br>Response Rate by Week 24 and Week 12 with<br>Prognostic Factors | Safety Analysis Set | |
| 15.12.2 | Analysis of Transfusion Response Rate by Week 24 | Safety Analysis Set | |
| 15.12.3 | Analysis of Splenic Response Rate at Week 24 | Safety Analysis Set | |
| 15.12.4 | Analysis of Response Rate in TSS at Week 24 | Safety Analysis Set | |
| 15.12.5.1 | Analysis of Hepcidin Change from Baseline by TI<br>Response | Biomarker<br>Analysis Set | |
| 15.12.5.2 | Analysis of Change from Baseline of Hepcidin<br>Daily Change by TI Response | Biomarker<br>Analysis Set | |
| 15.12.6.1 | Anemia Markers: Change and % Change from Baseline by TI Response | Biomarker<br>Analysis Set | |
| 15.12.6.2 | Anemia Markers: Change after TI Response from before TI Response in TI Responders | Biomarker<br>Analysis Set | TI Responders |
| 15.12.6.3 | Correlation of Anemia Markers in TI Responders | Biomarker<br>Analysis Set | TI Responders |
| 15.12.6.4 | Anemia Markers: Change and % Change from<br>Baseline by TI Response through Week 4 | Biomarker<br>Analysis Set | Subjects with No<br>Transfusion<br>through Week 4 |
| 15.12.7 | Liver Iron Content Change and % Change from<br>Baseline by TI Response | Biomarker<br>Analysis Set | |
| 15.12.8 | C-reactive Protein Change and % Change from<br>Baseline by TI Response | Biomarker<br>Analysis Set | |
| 15.12.9 | Pharmacodynamics Biomarker pSTAT3 Change and % Change from Baseline | Biomarker<br>Analysis Set | |
| 15.12.10.1 | Analysis of Duration of Transfusion Independent<br>Response | Safety Analysis Set | |
| 15.12.10.2 | Analysis of Time to Transfusion Independent (TI) | Safety Analysis Set | |
| 15.12.10.3 | Analysis of Overall Survival | Safety Analysis Set | |
| 15.12.10.4 | Analysis of Leukemia-Free Survival | Safety Analysis Set | |
| 15.12.10.5 | Analysis of Bone Marrow Fibrosis Score | Safety Analysis Set | |
| 15.12.10.6 | Efficacy Profile (Spleen, TSS, Transfusion Independent Response Status) by Week 24 | Safety Analysis Set | |
| 15.8 | Disposition of Study Subjects | Safety Analysis Set | |
| 15.12.3 | Waterfall Plots for % Change from Baseline in<br>Spleen Volume at Week 24 | Safety Analysis Set | |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 15.12.4 | Waterfall Plots for Change and % Change in Average of TSS by Treatment at Week 24 | Safety Analysis Set | |
| 15.12.5.1 | Median (Q1, Q3) plot of Hepcidin by Visit | Biomarker<br>Analysis Set | |
| 15.12.5.2 | Median (Q1, Q3) plot of % Change of Hepcidin by Visit | Biomarker<br>Analysis Set | |
| 15.12.5.3 | Median (Q1, Q3) plot of Hepcidin by Visit and TI<br>Response | Biomarker<br>Analysis Set | |
| 15.12.5.4 | Median (Q1, Q3) plot of % Change of Hepcidin by Visit and TI Response | Biomarker<br>Analysis Set | |
| 15.12.5.5 | Median (Q1, Q3) plot of Daily Hepcidin Change by Visit | Biomarker<br>Analysis Set | |
| 15.12.5.6 | Median (Q1, Q3) plot of % Change of Daily<br>Hepcidin Change by Visit | Biomarker<br>Analysis Set | |
| 15.12.5.7 | Median (Q1, Q3) plot of Daily Hepcidin Change by Visit and TI Response | Biomarker<br>Analysis Set | |
| 15.12.5.8 | Median (Q1, Q3) plot of % Change of Daily<br>Hepcidin Change by Visit and TI Response | Biomarker<br>Analysis Set | |
| 15.12.6.1 | Median (Q1, Q3) plot of Anemia Biomarkers by Visit | Biomarker<br>Analysis Set | |
| 15.12.6.2 | Median (Q1, Q3) plot of % Change from Baseline of Anemia Biomarkers by Visit | Biomarker<br>Analysis Set | |
| 15.12.6.3 | Median (Q1, Q3) plot of Anemia Biomarkers by<br>Visit and TI Response | Biomarker<br>Analysis Set | |
| 15.12.6.4 | Median (Q1, Q3) plot of % Change from Baseline of Anemia Biomarkers by Visit and TI Response | Biomarker<br>Analysis Set | |
| 15.12.6.5 | Median (Q1, Q3) plot of Anemia Biomarkers by<br>Time for TI Responders | Biomarker<br>Analysis Set | TI Responders |
| 15.12.6.6 | Median (Q1, Q3) plot of % Change from Pre-TI<br>Response of Anemia Biomarkers by Time for TI<br>Responders | Biomarker<br>Analysis Set | TI Responders |
| 15.12.6.7 | Median (Q1, Q3) plot of Anemia Biomarkers by<br>Visit through Week 4 | Biomarker<br>Analysis Set | Subjects with No<br>Transfusion<br>through Week 4 |
| 15.12.6.8 | Median (Q1, Q3) plot of % Change from Baseline of Anemia Biomarkers by Visit through Week 4 | Biomarker<br>Analysis Set | Subjects with No<br>Transfusion<br>through Week 4 |
| 15.12.6.9 | Median (Q1, Q3) plot of Anemia Biomarkers by<br>Visit and TI Response through Week 4 | Biomarker<br>Analysis Set | Subjects with No<br>Transfusion<br>through Week 4 |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 15.12.6.10 | Median (Q1, Q3) plot of % Change from Baseline of Anemia Biomarkers by Visit and TI Response through Week 4 | Biomarker<br>Analysis Set | Subjects with No<br>Transfusion<br>through Week 4 |
| 15.12.6.11 | Forest Plot of Anemia Biomarker Difference at<br>Baseline between TI Responders and Non-<br>responders | Biomarker<br>Analysis Set | |
| 15.12.6.12 | Forest Plot of Anemia Biomarker % Change from Pre-TI Response for TI Responders | Biomarker<br>Analysis Set | TI Responders |
| 15.12.8 | Median (Q1, Q3) plot of % Change from Baseline of C-reactive Protein by Visit | Biomarker<br>Analysis Set | |
| 15.12.9 | Median (Q1, Q3) plot of % Change from Baseline of pSTAT3 by Visit | Biomarker<br>Analysis Set | |
| 15.12.10.1 | Venn Diagram of Spleen Response, TSS Response and TI response at Week 24 | Safety Analysis Set | |
| 15.12.10.2 | Kaplan-Meier Plot for Overall Survival | Safety Analysis Set | |
| 15.12.10.3 | Kaplan-Meier Plot for Leukemia-Free Survival Safety Analysis Se (LFS) | | |
| 15.13.2 | Median (Q1, Q3) Plot Plasma Concentration of MMB and GS-644603 (Linear Scale and Semilogarithmic Scale) | Pharmacokinetic<br>Analysis Set | |
| 16.1.6 | Subjects Who Received Study Drug(s) from Specific Batches | Safety Analysis Set | |
| 16.2.1.1 | Subject Profiles | Safety Analysis Set | |
| 16.2.1.2 | Enrollment | Safety Analysis Set | |
| 16.2.1.3 | Subject Disposition | Safety Analysis Set | |
| 16.2.1.4 | Reasons for Screen Failure | Subjects Screened<br>But Not Enrolled | |
| 16.2.2.1 | Eligibility Criteria Deviations | Safety Analysis Set | |
| 16.2.2.2 | Important Protocol Deviations | Safety Analysis Set | |
| 16.2.3 | Subjects Excluded From Any Analysis Set | Safety Analysis Set | |
| 16.2.4.1 | Demographics | Safety Analysis Set | |
| 16.2.4.2.1 | Baseline Characteristics Part I | Safety Analysis Set | |
| 16.2.4.2.2 | Baseline Characteristics Part II | Safety Analysis Set | |
| 16.2.4.2.3 | Baseline Characteristics Part III | Safety Analysis Set | |
| 16.2.4.3 | Medical History | Safety Analysis Set | |
| 16.2.4.4 | Myelofibrosis Medical History | Safety Analysis Set | |
| 16.2.4.5 | Prior Medications | Safety Analysis Set | |
| 16.2.4.6 | Concomitant Medications | Safety Analysis Set | |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 16.2.4.7 | Prior Myelofibrosis Therapy | Safety Analysis Set | |
| 16.2.5.1 | Study Drug Administration | Safety Analysis Set | |
| 16.2.5.2 | Subjects Who Prematurely Discontinued Study<br>Drug | Safety Analysis Set | |
| 16.2.5.3 | Study Drug Accountability | Safety Analysis Set | |
| 16.2.5.4 | Plasma Pharmacokinetic Sampling Details and Concentrations | Safety Analysis Set | |
| 16.2.7.1.1 | Adverse Events | Safety Analysis Set | |
| 16.2.7.1.2 | Adverse Events for Peripheral Neuropathy SMQ | Safety Analysis Set | |
| 16.2.7.1.3 | Adverse Events for Cataract MST | Safety Analysis Set | |
| 16.2.7.1.4 | Adverse Events for First Dose Effect | Safety Analysis Set | |
| 16.2.7.2.1 | Deaths | All Screened<br>Subjects | |
| 16.2.7.2.2 | Adverse Events Leading to Death | Safety Analysis Set | |
| 16.2.7.3 | Serious Adverse Events | Safety Analysis Set | |
| 16.2.7.4 | Adverse Events with Severity of Grade 3 or Above | Safety Analysis Set | |
| 16.2.7.5.1 | Adverse Events Leading to Premature<br>Discontinuation of Study Drug | Safety Analysis Set | |
| 16.2.7.5.2 | Adverse Events Leading to Dose Reduction or<br>Temporary Interruption of Study Drug | Safety Analysis Set | |
| 16.2.8.1.1.1 | Hematology Results Part 1 | Safety Analysis Set | |
| 16.2.8.1.1.2 | Hematology Results Part 2 | Safety Analysis Set | |
| 16.2.8.1.1.3 | Hematology Results Part 3 | Safety Analysis Set | |
| 16.2.8.1.1.4 | Hematology Results Part 4 | Safety Analysis Set | |
| 16.2.8.1.1.5 | Hematology Results Part 5 | Safety Analysis Set | |
| 16.2.8.1.1.6 | Hematology Results Part 6 | Safety Analysis Set | |
| 16.2.8.1.2.1 | Serum Chemistry Results Part 1 | Safety Analysis Set | |
| 16.2.8.1.2.2 | Serum Chemistry Results Part 2 | Safety Analysis Set | |
| 16.2.8.1.2.3 | Serum Chemistry Results Part 3 | Safety Analysis Set | |
| 16.2.8.1.2.4 | Serum Chemistry Results Part 4 | Safety Analysis Set | |
| 16.2.8.1.2.5 | Serum Chemistry Results Part 5 | Safety Analysis Set | |
| 16.2.8.1.3.1 | Urinalysis Results Part 1 | Safety Analysis Set | |
| 16.2.8.1.3.2 | Urinalysis Results Part 2 | Safety Analysis Set | |
| 16.2.8.1.3.3 | Urinalysis Results Part 3 | Safety Analysis Set | |
| 16.2.8.1.3.4 | Urinalysis Results Part 4 | Safety Analysis Set | |

| TFL Number | Title1 | Title2 | Title3 |
|---|---|---|---|
| 16.2.8.1.4 | Iron Test Results | Safety Analysis Set | |
| 16.2.8.1.5 | Treatment-Emergent Marked Laboratory<br>Abnormalities | Safety Analysis Set | |
| 16.2.8.1.6 | Treatment-Emergent Grade 3 or Above Laboratory Abnormalities | Safety Analysis Set | |
| 16.2.8.2.1 | Vital Signs | Safety Analysis Set | |
| 16.2.8.2.2 | Body Weight and Height | Safety Analysis Set | |
| 16.2.8.3 | Pregnancy Report | Safety Analysis Set | |
| 16.3.1 | Spleen Volume Measurement | Safety Analysis Set | |
| 16.3.2.1 | Response of TSS | Safety Analysis Set | |
| 16.3.2.2 | TSS Measurement | Safety Analysis Set | |
| 16.3.2.3 | Individual Score of MPN-SAF 2.0 by Every 4<br>Weeks | Safety Analysis Set | |
| 16.3.3.1 | RBC Transfusion | Safety Analysis Set | |
| 16.3.3.2 | Transfusion Independent/Dependent by Week 24 | Safety Analysis Set | |
| 16.3.3.3 | Duration of Transfusion Independent for Subjects | Safety Analysis Set | |
| 16.3.4.1 | Hepcidin | Biomarker<br>Analysis Set | |
| 16.3.4.2.1 | Anemia Biomarkers Part 1 | Biomarker<br>Analysis Set | |
| 16.3.4.2.2 | Anemia Biomarkers Part 2 | Biomarker<br>Analysis Set | |
| 16.3.4.2.3 | Anemia Biomarkers for TI Responder Part 1 | Biomarker<br>Analysis Set | |
| 16.3.4.2.4 | Anemia Biomarkers for TI Responder Part 2 | Biomarker<br>Analysis Set | |
| 16.3.4.3 | Liver iron content | Biomarker<br>Analysis Set | |
| 16.3.4.4 | C-reactive Protein | Biomarker<br>Analysis Set | |
| 16.3.4.5 | Phosphorylated STAT3 | Biomarker<br>Analysis Set | |
| 16.3.4.6 | Overall Survival | Safety Analysis Set | |
| 16.3.4.7 | Leukemia-Free Survival | Safety Analysis Set | |
| 16.3.5 | Patient Global Improvement of Change (PGIC) | Safety Analysis Set | |

## **Appendix 2. Study Procedures Table**

| Assessment | Screening<br>(-28 to -21<br>days) | Baseline<br>(-7 +/- 2<br>days) | Enrollment | Week 2 (+/- 3 days) | Week<br>4<br>(+/- 3<br>days) | Week<br>8<br>(+/- 3<br>days) | Week<br>12<br>(+/- 3<br>days) | Week<br>16<br>(+/- 3<br>days) | Week<br>20<br>(+/- 3<br>days) | Week<br>24<br>(+/- 3<br>days) | Early Study<br>Drug<br>Discontinuation | 30 Day<br>Follow-<br>Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | | | | | | | | | | | |
| Medication and medical history | X | | | | | | | | | | | |
| Transfusion recoding | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam and<br>myelofibrosis<br>symptoms assessment | X | X | X | X | X | X | X | X | X | X | X | X |
| DIPSS assessment | X | | | | | | | | | | | |
| Vital signs | X | X | X | | X | X | X | X | X | X | X | X |
| AEs, concomitant medications | | X | X | X | X | X | X | X | X | X | X | X |
| Ophthalmic examination | | X | | | | | | | | X | X | |
| MMB accountability and dispensing <sup>g</sup> | | | X | | X | X | X | X | X | X | X | |
| MMB Dosing at site | | | X | X | X | X | X | X | X | X | | |
| Patient reporting outcom | nes | • | | | | | | | | | • | |
| Modified MPN-SAF<br>TSS | ← | | | | -Daily | | | | | -> | X | |
| PGIC | | | | | | | | | | X | X | |

| Assessment | Screening<br>(-28 to -21<br>days) | Baseline<br>(-7 +/- 2<br>days) | Enrollment | Week 2 (+/- 3 days) | Week<br>4<br>(+/- 3<br>days) | Week<br>8<br>(+/- 3<br>days) | Week<br>12<br>(+/- 3<br>days) | Week<br>16<br>(+/- 3<br>days) | Week<br>20<br>(+/- 3<br>days) | Week<br>24<br>(+/- 3<br>days) | Early Study<br>Drug<br>Discontinuation | 30 Day<br>Follow-<br>Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Assessment | s | | | | | | | | | | | |
| Viral hepatitis B and C | X | | | | | | | | | | | |
| Chemistry | X | | | | | | X | | | X | X | X |
| CBC with differential, reticulocyte count | X | X | | X | X | X | X | X | X | X | X | X |
| Thiamine status | | X | | | | | X | | | X | | |
| Erythropoietin | | X | | | | X | | | X | | | |
| C-reactive protein | X | X | | X | | | X | | | X | X | |
| Urinalysis | X | | | | X | X | X | X | X | X | X | X |
| Serum pregnancy test <sup>a</sup> | X | | | | | | | | | | | |
| Urine pregnancy test | | X | | | X | X | X | X | X | X | X | |
| Biomarker Samples | • | | • | | | | | | | | | |
| Bone marrow biopsy & aspirate | | X | | | | | | | | X | | |
| Buccal swab | | X | | | | | | | | | | |
| Spleen & LIC MRI | | X | | | | | | | | X | X | |
| Iron studies | X | X | | X | X | X | X | X | X | X | | |
| Hepcidin | | X | X | X | X | X | X | X | X | X | | |
| JAK2V617F allele<br>burden and other<br>mutation tests | | X | | | | | | | | X | X | |
| Pharmacodynamics <sup>c,d</sup> | | | $X^d$ | | X | | | | | X | | |
| Pharmacokinetics <sup>e</sup> | | | X | | X | | | | | X | | |

| Assessment | Screening<br>(-28 to -21<br>days) | Baseline<br>(-7 +/- 2<br>days) | Enrollment | Week<br>2<br>(+/- 3<br>days) | Week<br>4<br>(+/- 3<br>days) | Week<br>8<br>(+/- 3<br>days) | Week<br>12<br>(+/- 3<br>days) | Week<br>16<br>(+/- 3<br>days) | Week<br>20<br>(+/- 3<br>days) | Week<br>24<br>(+/- 3<br>days) | Early Study<br>Drug<br>Discontinuation | 30 Day<br>Follow-<br>Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cytokines/chemokines | X | | $X^{f}$ | | X | X | X | X | X | X | | |
| Exploratory signaling (mass cytometry) | | X | | | X | | X | | | X | | |
| CD34 <sup>+</sup> cell count | X | | X | | | | X | | X | | | |
| Gene expression | X | | X | | | | X | | X | | | |
| Immunophenotype (flow cytometry) | X | | X | | | | X | | X | | | |

a For female subject post-menopausal for less than two years, if FSH < 40 mIU/mL a serum pregnancy test will be required

b Hepcidin sample collection will occur at the following times?: baseline visit, between 8am-10am, 6 hours later; enrollment, Weeks 4, 8, 12, 16, 20 and 24 predose (between 8am and 10am) and 6 hours postdose

c Pharmacodynamics biomarker sample collection will occur at the following times: predose, 2,4 and 6 hours postdose at enrollment, then Week 4 and 24.

d Additional exploratory pharmacodynamics sample collection will occur at the following tines: predose, and 2 hours postdose at enrollment only.

PK sample collection at the following times: predose, 6 hours postdose. All other time points: predose only.

f Cytokine sample collection times at enrollment: predose, 6 hours postdose. All other time points: predose only.

g MMB accountability ONLY at Week 24 and ESDD visits.

Appendix 3. Peripheral Neuropathy SMQ AEs

| Name | Code | Level | Scope |
|---|---|---|---|
| Acute painful neuropathy of rapid glycaemic control | 10072909 | PT | Narrow |
| Acute polyneuropathy | 10066699 | PT | Narrow |
| Amyotrophy | 10002027 | PT | Narrow |
| Autoimmune neuropathy | 10070439 | PT | Narrow |
| Axonal neuropathy | 10003882 | PT | Narrow |
| Biopsy peripheral nerve abnormal | 10004846 | PT | Narrow |
| Decreased vibratory sense | 10067502 | PT | Narrow |
| Demyelinating polyneuropathy | 10061811 | PT | Narrow |
| Guillain-Barre syndrome | 10018767 | PT | Narrow |
| Ischaemic neuropathy | 10051307 | PT | Narrow |
| Loss of proprioception | 10057332 | PT | Narrow |
| Miller Fisher syndrome | 10049567 | PT | Narrow |
| Multifocal motor neuropathy | 10065579 | PT | Narrow |
| Myelopathy | 10028570 | PT | Narrow |
| Nerve conduction studies abnormal | 10029175 | PT | Narrow |
| Neuralgia | 10029223 | PT | Narrow |
| Neuritis | 10029240 | PT | Narrow |
| Neuronal neuropathy | 10071579 | PT | Narrow |
| Neuropathic muscular atrophy | 10075469 | PT | Narrow |
| Neuropathy peripheral | 10029331 | PT | Narrow |
| Notalgia paraesthetica | 10072643 | PT | Narrow |
| Peripheral motor neuropathy | 10034580 | PT | Narrow |
| Acute painful neuropathy of rapid glycaemic control | 10072909 | PT | Narrow |
| Acute polyneuropathy | 10066699 | PT | Narrow |
| Amyotrophy | 10002027 | PT | Narrow |
| Angiopathic neuropathy | 10079036 | PT | Narrow |
| Anti-myelin-associated glycoprotein associated polyneuropathy | 10078324 | PT | Narrow |
| Autoimmune neuropathy | 10070439 | PT | Narrow |
| Axonal neuropathy | 10003882 | PT | Narrow |
| Biopsy peripheral nerve abnormal | 10004846 | PT | Narrow |
| Decreased vibratory sense | 10067502 | PT | Narrow |
| Demyelinating polyneuropathy | 10061811 | PT | Narrow |

| Name | Code | Level | Scope |
|--------------------------------------------------|----------|-------|--------|
| Guillain-Barre syndrome | 10018767 | PT | Narrow |
| Ischaemic neuropathy | 10051307 | PT | Narrow |
| Loss of proprioception | 10057332 | PT | Narrow |
| Miller Fisher syndrome | 10049567 | PT | Narrow |
| Multifocal motor neuropathy | 10065579 | PT | Narrow |
| Myelopathy | 10028570 | PT | Narrow |
| Nerve conduction studies abnormal | 10029175 | PT | Narrow |
| Neuralgia | 10029223 | PT | Narrow |
| Neuritis | 10029240 | PT | Narrow |
| Neuronal neuropathy | 10071579 | PT | Narrow |
| Neuropathic muscular atrophy | 10075469 | PT | Narrow |
| Neuropathy peripheral | 10029331 | PT | Narrow |
| Notalgia paraesthetica | 10072643 | PT | Narrow |
| Peripheral motor neuropathy | 10034580 | PT | Narrow |
| Peripheral nervous system function test abnormal | 10034591 | PT | Narrow |
| Peripheral sensorimotor neuropathy | 10056673 | PT | Narrow |
| Peripheral sensory neuropathy | 10034620 | PT | Narrow |
| Polyneuropathy | 10036105 | PT | Narrow |
| Polyneuropathy chronic | 10064135 | PT | Narrow |
| Polyneuropathy idiopathic progressive | 10036111 | PT | Narrow |
| Radiation neuropathy | 10068886 | PT | Narrow |
| Sensorimotor disorder | 10062162 | PT | Narrow |
| Sensory disturbance | 10040026 | PT | Narrow |
| Sensory loss | 10040030 | PT | Narrow |
| Small fibre neuropathy | 10073928 | PT | Narrow |
| Tick paralysis | 10077336 | PT | Narrow |
| Toxic neuropathy | 10067722 | PT | Narrow |

## Appendix 4. Cataract MST AEs

| MEDDRA Term Name | MEDDRA Code | MEDDRA Level |
|----------------------|-------------|--------------|
| Atopic cataract | 10069649 | PT |
| Cataract | 10007739 | PT |
| Cataract congenital | 10007747 | PT |
| Cataract cortical | 10007748 | PT |
| Cataract diabetic | 10007749 | PT |
| Cataract nuclear | 10007759 | PT |
| Cataract operation | 10063797 | PT |
| Cataract subcapsular | 10007764 | PT |
| Cataract traumatic | 10007766 | PT |
| Lens discolouration | 10070549 | PT |
| Lenticular opacities | 10024214 | PT |
| Radiation cataract | 10037756 | PT |
| Toxic cataract | 10044135 | PT |
| Bioptic eye surgery | 10078599 | PT |
| Eye opacity | 10078394 | PT |
| Cornea verticillata | 10077604 | PT |

**Appendix 5.** Leukemic Transformation MST AEs

| MEDDRA Term Name | MEDDRA Code | MEDDRA Level |
|-----------------------------------------------|-------------|--------------|
| Acute megakaryocytic leukaemia | 10000860 | PT |
| Acute megakaryocytic leukaemia (in remission) | 10057194 | PT |
| Acute monocytic leukaemia | 10000871 | PT |
| Acute monocytic leukaemia (in remission) | 10000872 | PT |
| Acute myeloid leukaemia | 10000880 | PT |
| Acute myeloid leukaemia (in remission) | 10000881 | PT |
| Acute myeloid leukaemia recurrent | 10059034 | PT |
| Acute myelomonocytic leukaemia | 10000890 | PT |
| Acute promyelocytic leukaemia | 10001019 | PT |
| Erythraemic myelosis (in remission) | 10015246 | PT |
| Erythroleukaemia | 10015281 | PT |
| Acute biphenotypic leukaemia | 10067399 | PT |
| Acute leukaemia | 10000830 | PT |
| Acute leukaemia in remission | 10060930 | PT |
| Acute undifferentiated leukaemia | 10073479 | PT |
| Blast cell crisis | 10053747 | PT |
| Blast crisis in myelogenous leukaemia | 10050282 | PT |
| Chloroma | 10008583 | PT |
| Chloroma (in remission) | 10008584 | PT |
| Eosinophilic leukaemia | 10014958 | PT |
| Leukaemia basophilic | 10024293 | PT |
| Leukaemia granulocytic | 10024299 | PT |
| Leukaemia monocytic | 10024305 | PT |
| Monocytic leukaemia in remission | 10061295 | PT |
| Myeloid leukaemia | 10028549 | PT |
| Myeloid leukaemia in remission | 10061301 | PT |
| Aleukaemic leukaemia | 10001660 | PT |
| Central nervous system leukaemia | 10066231 | PT |
| Leukaemia | 10024288 | PT |
| Leukaemia cutis | 10053180 | PT |
| Leukaemia in remission | 10061220 | PT |
| Leukaemia recurrent | 10062489 | PT |

| MEDDRA Term Name | MEDDRA Code | MEDDRA Level |
|---------------------------------------|-------------|--------------|
| Leukaemic cardiac infiltration | 10077563 | PT |
| Leukaemic infiltration | 10069360 | PT |
| Leukaemic infiltration extramedullary | 10067117 | PT |
| Leukaemic infiltration gingiva | 10067431 | PT |
| Leukaemic infiltration hepatic | 10058671 | PT |
| Leukaemic infiltration ovary | 10075853 | PT |
| Leukaemic infiltration pulmonary | 10052368 | PT |
| Leukaemic infiltration renal | 10069359 | PT |
| Leukaemic retinopathy | 10059239 | PT |
| Mastocytic leukaemia | 10056450 | PT |
| Neonatal leukaemia | 10028958 | PT |

Appendix 6. Validation document of hepcidin testing from Radboud University



| Method name | Hepcidine in serum/plasma met WCX-TOF-massaspectrometrie methode | | |
|---|---|---|---|
| Work Unit | Iron metabolism | Iron metabolism | |
| Method Sop no. | 036977 In production May 2012 | | |
| Equipment | Microflex LT. | Equipment Sop nr. | 032496 |
| Authors | Name | sign | Date |
| Research technicians | Coby Laarakkers BSc. Erwin Wiegerinck BSc. | Qportal | digital |
| Supervisor | Prof. Dr. Dorine Swinkels,<br>MD/PhD | Qdoc | digital |

| ID | 042010 v 3 |
|---------------------|------------|
| Datum print | |
| Paraaf KAM-adviseur | |

# FH 009815 Validatie/verificatie rapport

KAM-systeem TML

# Radboudumc

| Index | | |
|--------|------------------------------------------------------|----|
| 1. | Generally. | 3 |
| 1.1 | Purpose. | 3 |
| 1.2 | Background. | 3 |
| 1.3 | Responsibilities. | 3 |
| 1.4 | Evaluation period. | 3 |
| 2. | Equipment/ method/ assay. | 3 |
| 3. | Definition and Terminology. | 3 |
| 3.1 | Abbreviations. | 3 |
| 3.2 | Units and decimals. | 4 |
| 4. | Procedure. | 4 |
| 4.1 | Internal standard heavy hepcidin-25 | 4 |
| 4.2 | Calibration hepcidin mass. | 4 |
| 4.3 | Internal Quality Control and Precision. | 5 |
| 4.4 | Linearity curve synthetic Hepcidin-25. | 9 |
| 4.5 | Intra run. | 10 |
| 4.6 | Inter run. | 11 |
| 4.6.1 | Linearity of native hepcidin-25 in serum/plasma (1). | 12 |
| 4.6.2 | Linearity of native hepcidin-25 in serum/plasma (2). | 15 |
| 4.7 | Detection limit | 16 |
| 4.8 | Reference values. | 16 |
| 5. | Clinical validation. | 20 |
| 6 | Archivating | 20 |
| 7. | References. | 21 |
| Bijlag | e meetonnauwkeurigheden. | 23 |

## FH 009815 Validatie/verificatie rapport

KAM-systeem TML



## 1. Generally.

## 1.1 Purpose.

Purpose is to validate the Weak Cation Exchange -Time Of Flight – Mass Spectrometry (WCX-TOF-MS) method for hepcidin-25 in serum/plasma

## 1.2 Background.

Hepcidin is an iron regulating peptide hormone and mainly produced in the liver. There are 3 isoforms hepcidin-20 (20 amino-acids [aa]), hepcidin-22 (22 aa) and hepcidin-24(24 aa) hep24 has recently discovered in samples from kidney patients. Only hepcidin-25(25 aa) has been shown to participate in the regulation of iron metabolism. It is thought to be the major regulator of dietary iron absorption and cellular iron release. It exerts its regulatory function by counteracting the function of ferroportin, the major cellular iron exporter in the membrane of macrophages, hepatocytes and the basolateral site of enterocytes. Hepcidin-25 induces the internalization and degradation of ferroportin, resulting in increased intracellular iron stores, decreased dietary iron absorption and decreased circulating iron concentrations. Several physiologic and pathologic processes regulate the synthesis of hepcidin. Iron deficiency, hypoxia, anemia and HFE-related hemochromatosis lead to a decrease in hepcidin synthesis and subsequent increased iron absorption from the intestine. Infection and inflammation lead to an increase in circulating hepcidin levels and subsequent decrease of iron absorption from the intestine and iron entrapment in the reticulo-endothelial macrophages, which may result in anemia of chronic disease. See for more information: www.hepcidinanalysis.com and (1, 2,8).

Since 2005 we measure hepcidin in our laboratory which resulted in numerous publications in peer reviewed journals.

In the clinic this assay is currently used as a diagnostic or monitoring tool for unexplained i) iron overload or ii) iron deficiency anemia. Moreover, the assay is exploited for clinical studies aiming for a better understanding of the pathophysiology of iron disorders and clinical trials in the monitoring or treatment with newly developed hepcidin modulating agents (11).

## 1.3 Responsibilities.

Performance: Coby Laarakkers, BSc.

Erwin Wiegerinck BSc.

Supervision: Prof. Dr. Dorine Swinkels, MD/ PhD. End responsibility Prof. Dr. Dorine Swinkels, MD/ PhD.

## 1.4 Evaluation period.

Start date: October 2011. Scheduled end date: Mai 2012

## 2. Equipment/ method/ assay.

Equipment: Microflex LT.

Method: WCX-TOF-MS.

Assay: Hepcidin-25 in serum.

## 3. Definition and Terminology.

## 3.1 Abbreviations.

WCX -Weak Cation Exchange.

TOF -Time Of Flight.

MS -Mass Spectrometry.

KAM-systeem TML



#### 3.2 Units and decimals.

| Assay | Unit | Significant figures |
|-------------|------|---------------------|
| Hepcidin-25 | nM | 3 |

#### 4. Procedure.

## 4.1 Internal standard heavy hepcidin-25

#### Procedure.

For this assay we have a custom made heavy hepcidin-25 internal standard (mass 2829.4 Da); DTHF ( $^{13}C_9$ ,  $^{15}N$ )P( $^{13}C_5$ ,  $^{15}N$ )I( $^{13}C_6$ ,  $^{15}N$ )CI( $^{13}C_6$ ,  $^{15}N$ )F( $^{13}C_9$ ,  $^{15}N$ )CCG( $^{15}N$ )CCHRSKCGMCCKT disulfide bridged (Peptide International, AF-179, Lot No221-006221)(9).

10 vials, freeze dried heavy hepcidin-25 are solved in  $H_2O$  in accordance with the manual. Solved heavy hepcidin25+40 of all the 10 vials were put together and mixed. Heavy hepcidin-25 with a concentration of 0.1 mM is aliquoted á 12  $\mu$ L in PCR tubes á 200  $\mu$ L and stored at -80°C in deep freezer "Iron metabolism" room 4.07 M325.04.264.

This internal standard is controlled by 10 x measurement of HiQC and LoQC.

The average of these 10 measurements should not differ more than 0.2 nM of the nominal values of the controls.

Data: H\microflex\2 controle IS hep25+41.

HiQC 2014:  $10.12 \pm 0.2$  nM LoQC 2014:  $2.34 \pm 0.1$  nM

## 4.2 Calibration hepcidin mass.

#### Procedure.

Calibration of the Microflex LT will be performed after ion source cleaning and services.

The calibrator contains hepcidin-20, hepcidin-22, hepcidin-24 (Peptides International, custom made, PCS-37242-PI, synthetic) and hepcidin-25 (Peptides International, PLP-4392-s, synthetic). Hepcidin-20 and 22 are a special gift from Tom Ganz and are isolated from urine (3). The mass values of the hepcidins can be found at UniProtKB (Proteinknowledgebase).

| Peptide | m/z |
|-------------|---------|
| Hepcidin-20 | 2191.77 |
| Hepcidin-22 | 2436.06 |
| Hepcidin-24 | 2673.90 |
| Hepcidin-25 | 2789.40 |


## 4.3 Internal Quality Control and Precision.

#### Procedure.

Precision is calculated by using MedLabQC (version:Philippe Marquis 3.24)

Control charts show the internal quality control. Hepcidin-25 results for the QC controls for the subsequent measurement runs.

#### Material.

HiQC 2014: heparin plasma pool is made by pooling samples from intensive care patients and plasma from an iron depleted HFE-hemochromatosis patient.

LoQC 2014: heparin plasma pool is made by pooling samples from 3 iron depleted hemochromatosis patients and plasma from intensive care patients.

The controls are aliquoted in polypropylene tubes (2 mL) á 250 ul sample. In deep freezer (-80 °C) "Iron metabolism" room 4.07 M325.04.264. number. For both QC's there are about 500 samples in the freezer.

### 4.3.1 Results MedLabQC

### HiQC and LoQC 2014

Hepcidin-25 measurements March 2015





**HiQC 2014** Hepcidin-20 measurements March 2015



**HiQC 2014** Hepcidin-22 measurements March 2015



## **HiQC 2014**



Hepcidin-24 measurements March 2015



| | <b>HiQC 2014</b> | LoQC 2014 |
|---------|------------------|-----------|
| | Hep25 | |
| n | 20 | 20 |
| average | 10.12 nM | 2.34 nM |
| SD | 0.557 nM | 0.157 nM |
| 3x SD | 1.67 nM | 0.47 nM |
| CV | 5.5 % | 6.7 % |

| | | HiQC 2014 | |
|---------|----------|-----------|----------|
| | Hep20 | Hep22 | Hep24 |
| n | 20 | 20 | 20 |
| average | 1.85 nM | 1.12 nM | 1.78 nM |
| SD | 0.224 nM | 0.148 nM | 0.219 nM |
| 3x SD | 0.67 nM | 0.44 nM | 0.66 nM |
| CV | 12.1 % | 13.2 % | 12.3% |



## 4.3.2 Control charts HiQC and LoQC hepcidin-25



Hepcidin-25 measurements March - April 2015.



Hepcidin-25 measurements March - April 2015

Control charts: H\LKN\ijzermetabolisme\Microflex\1-controle kaarten



## 4.4 Linearity curve synthetic Hepcidin-25.

### Procedure.

For this curve we used zero hepcidin serum coming from patient with juvenile haemochromatosis due to a homozygous mutation in the hemojuvelin gene (4). Different concentrations synthetic hepcidine-25 are added to this serum.

**A.** Linearity curve range (0-40 nM): concentrations synthetic hepcidine-25 added: 0, 0.5,1, 2, 3, 5, 7.5, 10, 15, 20 en 40 nM.



Linearity curve (0-40.0 nM) synthetic hepcidin-25 in zero serum with heavy hep25 as internal standard.

### Conclusion.

The curve is linear to at least 40 nM.



## 4.5 Intra run.

## Procedure.

4 patient plasma samples were measured 8 times in one run with WCX-TOF-ms. method with the Microflex LT.

Results (hepcidin-25 in nM).

| n=8 | 1 | 2 | 3 | 4 |
|---------|-------|------|------|------|
| average | 10.34 | 2.59 | 3.52 | 7.40 |
| STD | 0.22 | 0.15 | 0.12 | 0.26 |
| CV (%) | 2.14 | 2.67 | 3.31 | 3.53 |

3 of these 4 samples contained isoforms of hepcidin-25 ( > 1 nM)

Results (hepcidin-20 in nM).

| n=8 | 1 | 3 | 4 |
|---------|------|------|------|
| average | 2.34 | 5.75 | 4.90 |
| STD | 0.18 | 0.35 | 0.21 |
| CV (%) | 7.61 | 6.04 | 4.20 |

Results (hepcidin-22 in nM)

| results (heperum 22 m mvr) | | |
|----------------------------|------|------|
| n=8 | 1 | 4 |
| average | 1.36 | 1.71 |
| STD | 0.12 | 0.13 |
| CV (%) | 8.62 | 7.87 |

# FH 009815 Validatie/verificatie rapport

KAM-systeem TML

Radboudumc

Results (hepcidin-24 in nM)

| n=8 | 1 | 3 | 4 |
|---------|------|------|------|
| average | 2.25 | 1.38 | 2.37 |
| STD | 0.09 | 0.11 | 0.07 |
| CV (%) | 4.01 | 8.22 | 2.89 |

### Conclusie.

Intra run CV for hepcidin-25: < 3.6%.

Intra run CV's for the hepcidin isoforms are higher (between 2.9 and 8.6 %).

## 4.6 Inter run.

### Procedure.

Two plasma samples are measured on 8 different days (in 8 different runs) with the WCX-TOF-ms method for hepcidin-25 on Microflex LT.

## Results (hepcidin-25 in nM).

| n=8 | 5 | 6 |
|---------|-------|------|
| average | 10.47 | 2.58 |
| STD | 0.49 | 0.21 |
| CV (%) | 4.63 | 8.26 |



## Results (hepcidin-20, 22, 24 in nM)

| n=8 | Sample 5<br>Hep20 | Sample 5<br>Hep22 | Sample 5<br>Hep24 |
|---------|-------------------|-------------------|-------------------|
| average | 2.50 | 1.38 | 2.31 |
| STD | 0.34 | 0.16 | 0.39 |
| CV (%) | 13.7 | 11.6 | 16.8 |

#### Conclusie.

Interrun hepcidin-25: CV < 8.3 %

Interrun hepcidin-isoforms: CV: 11.6-16.8 %

# 4.6.1 Linearity of native hepcidin-25 in serum/plasma (1).

#### Material.

4 serum samples of healthy volunteers are selected for this test. Two samples have a hepcidin-25 concentration above 10 nM and 2 samples a concentration below 3 nM.

#### Procedure.

We tested linearity (1) in duplicate and used there for 4 serum samples, 2 with a high hepcidin concentration and 2 with a low hepcidin concentration. 1 High and 1 low sample is measured in duplicate in different mixture ratio on Microflex LT. You can find in table below the used mixture ratios. Based on the known values of the undiluted samples we calculated the rate value of the mixtures. The test should be linear for the evaluated range and the measured values should be equal to the calculated values.

Table: Mixture ratios.

| | Sample | A (low) | Sample B (high) | | Calculated value |
|---|---|---|---|---|---|
| 1 | 1 volume | 50 μL | nvt | 0 μL | = sample A |
| 2 | 3 volumes | 37.5 μL | 1 volume | 12.5 μL | $= (3 \times A + 1 \times B) / 4$ |
| 3 | 2 volumes | 25 μL | 2 volumes | 25 μL | $= (2 \times A + 2 \times B) / 4$ |
| 4 | 1 volume | 12.5 μL | 3 volumes | 37.5 μL | $= (1 \times A + 3 \times B) / 4$ |
| 5 | na | 0 μL | 1 volume | 50 μL | = sample B |



## Results (Hepcidin-25 in nM).

| Samples<br>A1 and B1 | Measured value (avg duplicate) | Calculated value | Difference between measured and calculated value |
|---|---|---|---|
| 1 | 16.1 | 16.1 | 0.0 |
| 2 | 11.6 | 12.8 | 1.2 |
| 3 | 8.2 | 9.5 | 1.3 |
| 4 | 6.0 | 6.1 | 0.1 |
| 5 | 2.8 | 2.8 | 0.0 |

| Samples<br>A2 and B2 | Measured value (avg duplicate) | Calculated value | Difference between measured and calculated value |
|---|---|---|---|
| 1 | 10.1 | 10.1 | 0.0 |
| 2 | 8.1 | 8.2 | 0.1 |
| 3 | 5.9 | 6.3 | 0.4 |
| 4 | 4.5 | 4.5 | 0.0 |
| 5 | 2.6 | 2.6 | 0.0 |







Conclusion: the method is linear to at least 16 nM.



# 4.6.2 Linearity of native hepcidin-25 in serum/plasma (2).

### Procedure.

To test linearity (2) we used 2 samples. These samples were measured in 5 different dilutions see table below and measured in duplicate on Microflex LT.

Table: Dilutions.

| | sample |
|---|-----------|
| 1 | undiluted |
| 2 | 1.25x |
| 3 | 1.66x |
| 4 | 2x |
| 5 | 5x |
| 6 | 10x |

### Material.

We selected 1 serum sample from a healthy volunteer (CH2) with a hepcidin concentration above 10 nM and 1 plasma sample from a kidney patient (KF218) with a high hepcidin value. See for dilutions table above.

## Results (hepcidin-25 in nM).

| | KF218 | CH2 |
|-----------|-------------|------|
| | Hep25 in nM | |
| undiluted | 15.9 | 11.0 |
| 1.25x | 12.0 | 8.1 |
| 1.66x | 9.1 | 6.3 |
| 2.5x | 5.8 | 4.3 |
| 5x | 3.1 | 2.0 |

Measured hepcidin.

| Dil.factor | KF218 | CH2 |
|------------|-------------|-------|
| | Hep25 in nM | |
| 1 | 15.9 | 11.0 |
| 1,25 | 15.0 | 10.2 |
| 1,66 | 15.1 | 10.5 |
| 2,5 | 14.4 | 10.7 |
| 5 | 15.4 | 10.2 |
| avg | 15.15 | 10.51 |
| sd | 0.507 | 0.302 |
| VC | 3.35% | 2.87% |

Calculated hepcidin levels using the measured value and the dilution factor.



Measured hepcidin-25 values: stars = HF218; dots = CH2

#### Conclusion.

Hepcidin measurement in these samples is linear for at least to 15 nM.

### 4.7 Detection limit

The detection limit is determined at 0.5 nM. The signal/noise ratio was >2 for a zero serum added with 0.5 nM synthetic hepcidin-25 (5).

### 4.8 Reference values.

### Procedure.

The reference range of serum hepcidin-25 is <0.5 nM-14.7 nM (median 4.5 nM) for men, <0.5 -12.3 nM (median 2.0 nM) for premenopausal women, and <0.5-15.6 nM (median 4.9 nM) for postmenopausal women. We have also assessed i) references ranges per 5-year age group for men and women; ii) for hepcidin/ferritin ratio and transferrin saturation/hepcidin ratio. These reference levels for the WCX-TOF MS method are derived from those of our ELISA method[6,7], based on the regression line between the ELISA and WCX-TOF MS results obtained for the same samples from patients without hepcidin isoforms[1,7].

We also assessed:

- references ranges for serum hepcidin-25 and hepcidin/ferritin ratio in children (6 months to 3 years old) in the normative population (N=292) as measured by weak cation exchange time-of-flight mass spectrometry (WCX-TOF MS)[9].
- Reference ranges for serum hepcidin-25 during pregnancy [12].

More details on the WCX-TOF MS reference values for hepcidin can be found on our website <a href="https://www.hepcidinanalysis.com">www.hepcidinanalysis.com</a> and in the references.

### 4.9 measurement uncertainty

The measurement uncertainty is 14.1%, calculated by CV  $_{total\ variation\ analyse}$  This is lower than  $\frac{1}{2}$ CV  $_{biological\ variation}$  Calculation see supplement 1



**Results:** 

# MS-method\_hepcidin-25 (nM)

Reference ranges for serum hepcidin (nM) per 5-year age group for adult men and women in the reference population.

| | | | Men (N | =1,066) | | | | Women | (N=882) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% re | ference range | | | | 95% re | ference range |
| Age, years | N | (%) | Median | P2.5 | P97.5 | N | (%) | Median | P2.5 | P97.5 |
| 18-24 | 10 | (1) | 5.3 | 0.8 | 11.0 | 21 | (2) | 1.1 | < 0.5 | 6.3 |
| 25-29 | 16 | (2) | 4.9 | < 0.5 | 15.3 | 28 | (3) | 1.4 | < 0.5 | 6.6 |
| 30-34 | 18 | (2) | 4.2 | < 0.5 | 15.8 | 24 | (3) | 1.9 | < 0.5 | 13.1 |
| 35-39 | 22 | (2) | 3.6 | < 0.5 | 12.1 | 36 | (4) | 1.5 | < 0.5 | 9.9 |
| 40-44 | 19 | (2) | 6.1 | < 0.5 | 11.0 | 65 | (7) | 2.5 | < 0.5 | 15.2 |
| 45-49 | 76 | (7) | 3.4 | < 0.5 | 13.2 | 110 | (12) | 1.6 | < 0.5 | 8.9 |
| 50-54 | 106 | (10) | 4.0 | < 0.5 | 13.8 | 140 | (16) | 2.9 | < 0.5 | 14.3 |
| 55-59 | 173 | (16) | 4.4 | < 0.5 | 15.7 | 129 | (15) | 4.9 | < 0.5 | 13.6 |
| 60-64 | 179 | (17) | 4.5 | < 0.5 | 14.3 | 137 | (16) | 4.7 | < 0.5 | 17.3 |
| 65-69 | 186 | (17) | 5.3 | < 0.5 | 13.9 | 95 | (11) | 4.9 | < 0.5 | 14.2 |
| 70-74 | 133 | (12) | 4.9 | < 0.5 | 17.0 | 62 | (7) | 5.1 | < 0.5 | 24.2 |
| 75-79 | 99 | (9) | 3.8 | < 0.5 | 16.1 | 16 | (2) | 5.4 | 0.8 | 18.4 |
| 80-84 | 22 | (2) | 3.8 | 1.6 | 12.6 | 10 | (1) | 7.2 | < 0.5 | 12.0 |
| ≥85 | 7 | (1) | 6.8 | 1.6 | 12.8 | 9 | (1) | 3.7 | < 0.5 | 15.4 |
| All | 1,066 | (100) | 4.5 | < 0.5 | 14.7 | 882 | (100) | 3.6 | < 0.5 | 14.6 |

Premenopausal women (<55 year): (N=424)

- Median = 2.0 nM
- P2.5 = 0.1 nM (< 0.5 nM)
- P97.5 = 12.3 nM

Postmenopausal women (>=55 year): (N=458)

- Median = 4.9 nM
- P2.5 = 0.2 nM (< 0.5 nM)
- P97.5 = 15.6 nM



Reference ranges for serum hepcidin (nM) in children aged 6 months to 3 years.

| Hepcidin | | 95 | % CI |
|----------|--------|------|-------|
| N | Median | P2.5 | P97.5 |
| 292 | 3.6 | 0.94 | 12.2 |

| Hepcidin | | | | 95% CI | |
|--------------|-----|------|--------|--------|-------|
| Age (months) | N | (%) | Median | P2.5 | P97.5 |
| 3-12 | 111 | (38) | 4.1 | 1.1 | 12.8 |
| 13-18 | 62 | (21) | 3.8 | 0.8 | 12.0 |
| 19-24 | 43 | (15) | 2.5 | 0.9 | 11.8 |
| 25-30 | 38 | (13) | 3.4 | 0.8 | 21.7 |
| 31-36 | 38 | (13) | 3.9 | 0.3 | 14.6 |

| Hepcidin | | | 95% CI | |
|----------|-----|--------|--------|-------|
| Gender | N | Median | P2.5 | P97.5 |
| Male | 207 | 3.6 | 0.9 | 11.9 |
| Female | 85 | 4.0 | 0.8 | 14.0 |

| Hepcidin | | | 959 | % CI |
|---------------------------|-----|--------|------|-------|
| Time of sample collection | N | Median | P2.5 | P97.5 |
| <12.00 pm | 170 | 3.0 | 0.9 | 11.4 |
| 12.00-17.00 pm | 122 | 4.5 | 1.1 | 14.0 |



Reference range for serum hepcidin in specified time periods during pregnancy

| Gestation | | 9 | 95 % refe | rence ra |
|-----------|----|--------|-----------|----------|
| weeks | N | Median | P2.5 | P97.5 |
| 7-15 | 22 | 1.9 | < 0.5 | 8.6 |
| 19-25 | 21 | < 0.5 | < 0.5 | 6.8 |
| 29-35 | 16 | < 0.5 | < 0.5 | 2.4 |

## Hepcidin-25/ferritin (pmol/μg)

Reference ranges for hepcidin/ferritin per 5-year age group for adult men and women in the reference population.

Men: (N=1064)

- Median =  $26.7 \text{ pmol/}\mu\text{g}$
- $P2.5 = 2.9 \text{ pmol/}\mu\text{g}$
- $P97.5 = 87.9 \text{ pmol/}\mu\text{g}$

Premenopausal women (<55 year): (N=424)

- Median =  $35.7 \text{ pmol/}\mu\text{g}$
- P2.5 = 3.0 pmol/µg
- $P97.5 = 167.3 \text{ pmol/}\mu\text{g}$

Postmenopausal women (>=55 year): (N=458)

- Median =  $40.5 \text{ pmol/}\mu\text{g}$
- $P2.5 = 9.1 \text{ pmol/}\mu\text{g}$
- $P97.5 = 143.1 \text{ pmol/}\mu\text{g}$

Reference ranges for hepcidin/ferritin in children aged 6 months to 3 years.



# MS-method\_TSAT/hepcidin-25 (%/nM)

Men: (N=1059)

- Median = 7.3 %/nM
- P2.5 = 1.7 %/nM
- P97.5 = 256.3 %/nM

Premenopausal women (<55 year): (N=422)

- Median = 13.9 %/nM
- P2.5 = 2.0 %/nM
- P97.5 = 330.0 %/nM

Postmenopausal women (>=55 year): (N=457)

- Median = 5.7 %/nM
- P2.5 = 1.5 %/nM
- P97.5 = 73.4 %/nM

## 5. Clinical validation.

Zie www.hepcidinanalysis.com/expertise/(1).

## 6 Archivating

Word-document: H-LKN\ijzermetabolisme\microflex\kwaliteit\validatie rapport hep25

Laboratory notebook: 485

# FH 009815 Validatie/verificatie rapport

KAM-systeem TML



## 7. References.

- 1. <a href="http://www.hepcidinanalysis.com/">http://www.hepcidinanalysis.com/</a>
- 2. Bergmans JP, Kemna EH, Janssen MC, Jacobs EM, Stalenhoef AF, Marx JJ, Swinkels DW. [Hereditary haemochromatosis: novel genes, novel diseases and hepcidin] Ned Tijdschr Geneeskd. 200;151(20):1105-8.
- 3. Park CH, Valore EV, Waring AJ, Ganz T. Hepcidin, a urinary antimicrobial peptide synthesized in the liver. J Biol Chem 2001;276:7806–10.
- 4. van Dijk BA, Kemna EH, Tjalsma H, Klaver SM, Wiegerinck ET, Goossens JP, Slee PH, Breuning MH, Swinkels DW. Effect of the new HJV-L165X mutation on penetrance of HFE. Blood. 2007;109(12):5525-6.
- 5. Kroot JJ, Hendriks JC, Laarakkers CM, Klaver SM, Kemna EH, Tjalsma H, Swinkels DW. (Pre)analytical imprecision, between-subject variability, and daily variations in serum and urine hepcidin: Implications for clinical studies. Anal Biochem 2009;389(2):124-9.
- Kroot JJC. Laarakkers CM. Geurts-Moespot AJ. Grebenchtchikov N. Pickkers P. van Ede AE et al. Immunochemical and Mass-Spectrometry-Based Serum Hepcidin Assays for Iron Metabolism Disorders. Clin Chem 2010;56:1570-9.
- 7. Galesloot TE, Vermeulen SH, Geurts-Moespot AJ, Klaver SM, Kroot JJ, van Tienhoven D, Wetzels JF, Kiemeney LA, Sweep FC, de Heijer M, Swinkels DW. Serum hepcidin: reference ranges and biochemical correlates in the general population. Blood, 2011; 117(25)
- 8. Kroot JJC, Tjalsma H, Fleming R and Swinkels DW . Hepcidin in human iron disorders: diagnostic implications. Clinical Chemistry 2011; 57:12, 1650-1669
- 9. Laarakkers C, Wiegerinck E, Klaver S, Kolodziejcyk M, Gille H, Hohlbaum M, Tjalsma H, Swinkels D. Improved mass spectrometry assay for plasma hepcidin: detection and characterization of a novel hepcidin isoform.. PLoS One, 2013; 8(10).
  - 10. Uijterschout L, Swinkels DW, Domellöf M, Lagerqvist C, Hudig C, Tjalsma H, Vos R, van Goudoever JB, Brus F. Serum hepcidin measured by immunochemical and mass-spectrometric methods and their correlation with iron status indicators in healthy children aged 0.5-3 y. Pediatric Research 2014; 76;409-414
  - 11. van Eijk LT, John AS, Schwoebel F, Summo L, Vauléon S, Zöllner S, Laarakkers CM, Kox M, van der Hoeven JG, Swinkels DW, Riecke K, Pickkers P. Effect of the antihepcidin Spiegelmer lexaptepid on inflammation-induced decrease in serum iron in humans. Blood. 2014;124(17): 2643-6.
  - 12. van Santen S, Kroot JJ, Zijderveld G, Wiegerinck ET, Spaanderman ME, Swinkels DW. The iron regulatory hormone hepcidin is decreased in pregnancy: a prospective longitudinal study. Clin Chem Lab Med 2012; 14: 1-7.

# FH 009815 Validatie/verificatie rapport

KAM-systeem TML



**Invoer referentiewaardes** HELIX / GLIMS\*

Naam invoerder Nvt (geen wijzigingen)

Datum

Handtekening

<sup>\* =</sup> Doorhalen wat niet van toepassing is

Supplement 1

## Bijlage meetonnauwkeurigheden.

Biologische variatie<sub>tussen dag</sub> humaan hepcidin is 48.8% (Murphy et al<sup>1</sup>)

$$CV_{totale\ variatie\ (pre)-analyse} < \frac{1}{2}\ CV_{biologische\ variatie}$$

Berekening:

$$CV_{totale \ variatie \ (pre)-analyse} = \sqrt{\frac{(CV_{analyse})^2 + (CV_{pre-analyse \ 24h})^2}{(10)^2 + (10)^2}}$$

$$CV_{totale \ variatie \ (pre)-analyse} = \sqrt{\frac{(10)^2 + (10)^2}{200}}$$

$$CV_{totale \ variatie \ (pre)-analyse} = \sqrt{\frac{(10)^2 + (10)^2}{200}}$$

$$CV_{totale\ variatie\ (pre)-analyse} = 14.1\%$$

$$CV_{totale\ variatie\ (pre)-analyse} < \frac{1}{2}\ CV_{biologische\ variatie}$$

$$14.1\% < \frac{1}{2} \times 48.8\% \Rightarrow pass$$

Serum en plasma samples mogen een dag bij KT blijven staan. Afspraak is samples dezelfde dag nog in de vriezer.

- 1. Murphy et al, Quantitation of hepcidin from human and mouse serum using liquid chromatography tandem mass spectrometry, Blood, Vol 110, 3.
- 2. The Hitch-hiker's Guide to Measurement Uncertainty (MU) in Clinical LaboratoriesApril 2012
- 3 Graham White, SA Pathology, Flinders Medical Centre, Bedford Park, Adelaide, SA 5042, Australia
- 4 Clin Chem 2011 Sep 57(9): 1334-6. Gross overestimation of total allowable error based on biological variation. Oosterhuis WP

# Appendix 7. Validation document of pSTAT testing from Covance



# **Client Acceptance of Report**

Sponsor: Gilead Sciences

Protocol Title: Detect Phosphorylated STAT3 in IL6 Stimulated Whole Blood (With Additional

Protocol: GS-US-352-1151 (USA)/1153 (EU)/ others

Report Number: LCT13050-QR01-01

LabCorp Clinical Trials Management has reviewed the data in the validation report described above. An audit of the report was finalized by LabCorp Clinical Trials QA on the date below. Please review the report and provide a signature accepting the report and the data within.

Client has 10 business days from date signed by LCT QA below to declare acceptance of report. If no response is received within 10 business days the report is considered final and will be archived internally.

| R. DeMarco Morgan/QA Auditor LabCorp Clinical Trials | 12-Dec-2014 Date |
|---|---|
| Anita Reddy Kevin Kwei Gilead Sciences | 30 - Oct ,2015 |
| Comments: Service Arida Reddy ( Arida Reddy @gileoch.com | 19-10e-9014 BDW |
| Do Cament Jouranded on Ex to anite Reddy on | 14 Bic 2014,<br>RB2<br>14 bic 2014 |
| ms. Reddy auknowledge recipt a 18 Dec 2014. | • |



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

Assay Transfer and Qualification of a Custom Flow Cytometric Assay to Detect Phosphorylated STAT3 in IL6 Stimulated Whole Blood (With Additional Preparation and Storage for Future ELISA Assay)

Flow Cytometry Performed by: LabCorp Clinical Trials 201 Summit View Drive, Suite 200 Brentwood, TN 37027

Conducted for: Gilead Science, Inc. 368 Lakeside Dr. Foster City, CA 94404

Validation Initiation Date: Validation End Date:

Kenneth Pennline, Ph.D.

January 2014 April 2014

Date

Date

LabCorp Clinical Trials Review:

| 04-Dec-2014 |
|------------------|
| ( |
| Date |
| <u>03- Dec</u> 2 |

LabCorp Clinical Trials – Brentwood

(13 Dec 2014)

Supervisor - Advanced Cytometric Applications

Rachael Wilson

# Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

## TABLE OF CONTENTS

| Quality Assurance Statement—Good Clinical Practice | |
|--------------------------------------------------------|------|
| BACKGROUND | - |
| ASSAY DESCRIPTION AND REPORTABLES | |
| Gilead pSTAT3 Stimulation Assay Panel | 4 |
| Gilead pSTAT3 Stimulation Assay Reportables | |
| EXPERIMENTS | .:.6 |
| Phase I: Antibody Titration | 6 |
| Phase II: Assay Linearity | 6 |
| Phase III: Inter-Operator and Intra-Assay Precision | 6 |
| Phase IV: Assay Transfer ELISA testing only | 6 |
| Phase IV: Assay Transfer – Flow Cytometry testing only | 7 |
| MATERIALS AND METHODS | 7 |
| Gilead pSTAT3 Stimulation Assay Method | 7 |
| Reagents | 7 |
| DATA ANALYSIS | 8 |
| ABBREVIATIONS | 8 |
| REFERENCES | 9 |
| ACCEPTANCE CRITERIA | 9 |
| Linearity Acceptance Criteria | 9 |
| nter-Operator Precision Acceptance Criteria | 9 |
| ntra-Assay Precision Acceptance Criteria | 9 |
| Assay Transfer | 9 |
| RESULTS | 10 |
| Phase I: Antibody Titration | 10 |
| Phase II: Assay Linearity | 10 |
| hase III: Inter-Operator and Intra-Assay Precision | 10 |
| hase IV: Assay Transfer ELISA testing only | 10 |
| hase IV: Assay Transfer – Flow Cytometry testing only | 10 |
| Conclusion | 11 |



## Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

## LIST OF APPENDICES

| | 12 |
|---|---|
| Appendix A: Table 1, Linearity - Healthy Donors 1-3 | 12 |
| Appendix B: Table 1, Linearity - Healthy Donors 1-3 - Continued | |
| Appendix C: Table 1, Linearity - Healthy Donors 1-3 - Continued | 14 |
| Appendix D: Table 1, Linearity - Healthy Donors 1-3 - Continued | |
| Appendix E: Table 1, Linearity - Healthy Donors 1-3 - Continued | 16 |
| Appendix F: Table 1, Linearity - Healthy Donors 1-3 - Continued | |
| Appendix G: Table 1, Linearity - Healthy Donors 1-3 - Continued | 18 |
| Appendix H: Table 1, Linearity - Healthy Donors 1-3 - Continued | 19 |
| Appendix I: Table 1, Linearity - Healthy Donors 1-3 - Continued | 20 |
| Appendix J: Table 1, Linearity - Healthy Donors 1-3 - Continued | 21 |
| Appendix K: Table 1, Linearity - Healthy Donors 1-3 - Continued | 22 |
| Appendix L: Table 1, Linearity - Healthy Donors 1-3 - Continued | 23 |
| Appendix M: Table 1, Linearity - Healthy Donors 1-3 - Continued | 24 |
| Appendix N: Table 1, Linearity - Healthy Donors 1-3 - Continued | 25 |
| Appendix O: Table 1, Linearity - Healthy Donors 1-3 - Continued | 26 |
| Appendix P: Table 2, Linearity - Relative Error Calculations - Donor 1 | 27 |
| Appendix O: Table 3, Linearity - Relative Error Calculations - Donor 2 | 28 |
| Appendix R: Table 4, Linearity - Relative Error Calculations - Donor 3 | 29 |
| Appendix S: Table 5 Inter/Intra-Assay Precision | 30 |
| Appendix T: Table 5, Inter/Intra-Assay Precision - Continued | 31 |
| Appendix U: Table 5. Inter/Intra-Assay Precision - Continued | |
| Appendix V: Table 5, Inter/Intra-Assay Precision - Continued | 33 |
| Appendix W: Table 5, Inter/Intra-Assay Precision - Continued | 34 |
| Appendix X: Table 6: Assay Transfer, Flow Assay | 35 |
| Appendix Y: Table 6: Assay Transfer, Flow Assay - Continued | 36 |
| Appendix Z: Table 6: Assay Transfer, Flow Assay - Continued | 37 |
| Appendix AA: Table 6: Assay Transfer. Flow Assay - Continued | 38 |
| Appendix BB: Table 7: Assay Transfer, Flow Assay %Stimulation and Acceptance | 39 |
| Appendix CC: Gating Strategy | 40 |
| LIST OF EQUATIONS | |
| | 7 |
| Equation 1: % stim = (stim - unstim)/unstim x 100 | ammun /<br>Milenike IV |
| Equation 2: %Relative Error (%RE) = [Accepted Value (@2000 cells) - Measured Value (@2000 Cells)*100 | u shiveTh |
| Accepted Value (Im/1000 Cells)* (00 | *************************************** |



# Quality Assurance Statement—Good Clinical Practice

Sponsor:

Gilead Sciences, Inc.

Protocol Number:

GS-US-352-1151 (USA)/1153 (EU)/ others

Protocol Title:

Assay Transfer and Qualification of a Custom Flow Cytometric Assay to Detect Phosphorylated STAT3 in IL6 Stimulated Whole Blood

(With Additional Preparation and Storage for Future ELISA Assay)

The clinical laboratory study was audited according to the Standard Operating Procedures of LabCorp Clinical Trials.

The following attests to the dates that audits were conducted and to the findings reported:

| Date(s) of Audit | Type of Audit | Date Reported to LabCorp Clinical Trials Management |
|---|---|---|
| 21May2014 –<br>12Jun2014 | Qualification Data Audit | 12Jun2014 |
| 05Dec2014 | Assay Transfer Data Audit | 05Dec2014 |
| 12Jun2014 | Report Audit | 12Jun2014 |

| | K. | 16 | 11 | cure | | 11 | 700 |
|----|-----|---------|------|-------|-----|----|-------|
| R. | Del | Marco l | Mor | gan/( | QA. | Au | ditor |
| La | bCo | rp Clin | ical | Tria | ls | | U |

08-Dec- 2012

Date



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

## BACKGROUND

The project involved the assay transfer of an assay that had been developed internally at Gilead Sciences, Inc. Subsequent qualification included reproducibility and linearity experiments, but did not include stability, as that was assessed by client. The work herein qualified the assay for the measurement of pSTAT3 levels in CD3+ and CD3+/CD4+ lymphocytes in healthy donor peripheral whole blood that had been stimulated with Interleukin-6 for use in clinical trials.

## ASSAY DESCRIPTION AND REPORTABLES

The panel and associated reportables for the validation include the following:

## Gilead pSTAT3 Stimulation Assay Panel

| | Panel | | | |
|---------------------|-------------|------|-------------|------|
| Conditions | Tube | FITC | PE | V450 |
| Unstimulated-Tube 1 | FMO-PE | CD3 | blank | CD4 |
| Unstimulated-Tube 2 | Total STAT3 | CD3 | Total STAT3 | CD4 |
| Unstimulated-Tube 3 | pSTAT3 | CD3 | pSTAT3 | CD4 |
| IL-6 Stim Tube 4 | FMO-PE | CD3 | blank | CD4 |
| IL-6 Stim Tube 5 | Total STAT3 | CD3 | Total STAT3 | CD4 |
| IL-6 Stim Tube 6 | pSTAT3 | CD3 | pSTAT3 | CD4 |

## Gilead pSTAT3 Stimulation Assay Reportables

- e %Lymphs
- Region Events CD3+ Lymphs
- %CD3+[Lymphs]
- Region Events CD3+/CD4+ Lymphs
- %CD3+/CD4 [Lymphs]
- MESF FMO-PE unstim (CD3+ Lymphs)
- MESF FMO-PE unstim [CD3+/CD4+ Lymphs]
- %tSTAT3 unstim [CD3+ Lymphs]
- %tSTAT3 unstim [CD3+/CD4+ Lymphs]
- MESF tSTAT3 upstim [CD3+ Lymphs]
- MESF tSTAT3 unstim [CD3+/CD4+ Lymphs]
- %pSTAT3 unstim [CD3+ Lymphs]
- %pSTAT3 unstim [CD3+/CD4+ Lymphs]
- MESF pSTAT3 unstim [CD3+ Lymphs]
- MESF pSTAT3 unstim [CD3+/CD4+ Lymphs]
- MESF FMO-PE STIM [CD3+ Lymphs]
- MESF FMO-PE STIM [CD3+/CD4+ Lymphs]
- %tSTAT3 STIM [CD3+ Lymphs]
- %tSTAT3 STIM [CD3+/CD4+ Lymphs]
- MESF tSTAT3 STIM [CD3+ Lymphs]
- MESF tSTAT3 STIM [CD3+/CD4+ Lymphs]
- %pSTAT3 STIM [CD3+ Lymphs]



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

- %pSTAT3 STIM [CD3+/CD4+ Lymphs]
- MESF pSTAT3 STIM [CD3+ Lymphs]
- MESF pSTAT3 STIM [CD3+/CD4+ Lymphs]
- MFI FMO-PE unstim [CD3+ Lymphs]
- MFI FMO-PE unstim [CD3+/CD4+ Lymphs]
- MFI tSTAT3 unstim [CD3+ Lymphs]
- MFI tSTAT3 unstim [CD3+/CD4+ Lymphs]
- MFI pSTAT3 unstim [CD3+ Lymphs]
- MFI pSTAT3 unstim [CD3+/CD4+ Lymphs]
- MFI FMO-PE STIM [CD3+ Lymphs]
- MFI FMO-PE STIM [CD3+/CD4+ Lymphs]
- MFI tSTAT3 STIM [CD3+ Lymphs]
- MFI tSTAT3 STIM [CD3+/CD4+ Lymphs]
- MFI pSTAT3 STIM [CD3+ Lymphs]
- MFI pSTAT3 STIM [CD3+/CD4+ Lymphs]

## **EXPERIMENTS**

## Phase I: Antibody Titration

This phase was conducted in order to titrate all reagents to saturation within the client method. All single color reagents were titrated within the method on 3 applicable donors (normal whole blood drawn into sodium heparin for surface antibodies, and IL-6 stim/unstim for pSTAT3). Once saturation was determined for each marker, the combined panel was tested on 3 additional donors within the panel. No preparation of ELISA samples was done in this phase.

## Phase II: Assay Linearity

In order to determine the minimum number of lymphocytes required to accurately determine the MESF/MFI and the % positivity of the phosphorylated epitopes of interest, the following was done: 3 normal whole blood samples were drawn into sodium heparin and then assayed within the method starting at between 0.5-1x10^6 cells per tube. The samples were acquired using a stop gate on the lymphocyte population (limiting population) for 2000, 1000, 500, 300, 100, and 50 events. These samples were processed in singlet by one operator. Each sample was acquired in triplicate. The 2000 event sample was used as the basis for determining the relative error of the MESF/MFI and the % positivity.

# Phase III: Inter-Operator and Intra-Assay Precision

2 normal whole blood specimens were drawn into NaHeparin. The samples were shipped back to Brentwood LCT within 1 Day ex-vivo using the Credo GTC4L, 2-8°C shippers from World Courier. The samples were tested immediately within the panel by 2 operators in triplicate. The acquisition stop gate was set to acquire 2000 lymphocytes per client request for this phase.

# Phase IV: Assay Transfer -- ELISA testing only

Reference LA-LCT Assay Qualification Plan GEN82, Cross Laboratory Qualification of Human STAT3 [pY705] ELISA (cell lysate, units/mL)

The Brentwood facility drew 2 NWB donors (6mL NaHeparin tubes, 2 per site) and shipped to each of the processing locations. One 6-mL tube was processed on the same day of receipt and the second 6-mL tube was




Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

processed the next day. Opened sample was discarded after samples have been prepped to ensure that only the sterile, unopened sample is used on Day 2. The 2 vials of blood from each donor were shipped to each LCT Cranford, LCT LA laboratories and to Gilead for further processing. The samples were shipped using World Courier Credo GTC4L, 2-8°C shippers only containing temperature monitors. The specimens were processed in each location on day of receipt by operator 1 (only to lysate point) and again on Day 2 by operator 2 (only to Lysate point). The specimens were processed in quadruplicate (4 stimulated replicates and 4 unstimulated replicates per donor). The Cranford lab prepared double aliquots of each replicate. One set was shipped to LCT-LA for further processing in ELISA; the other set was shipped to Gilead for further processing in ELISA. The LCT-LA lab also processed the samples to the lysate point. One set was retained to complete in the ELISA assay, the other set was shipped back to Gilead for them to complete the ELISA assay. The ELISA runs were performed in triplicate on each lysate replicate by 2 different operators. The Assay Transfer was to be repeated 2 additional times using 2 different normal healthy donor specimens approximately one week after first run. This process was actually repeated on 6 total donors due to variability during runs. Results for the ELISA were compared between Gilead and LCT-LA on these lysates. Additionally, the LCT-LA lab performed the ELISA lysates and performed the entire assay from start to completion on the received whole blood for comparison with Gilead processing from start to completion. Data for all of these comparisons described herein were presented in the corresponding report for Assay Qualification Plan GEN82 and not included, except in conclusion and reference in this report. Acceptance criteria for said ELISA comparison data are also located in Assay Qualification Plan GEN82.

## Phase IV: Assay Transfer - Flow Cytometry testing only

The Brentwood facility drew 3 NWB donors and ship to LCT Cranford flow lab using World Courier Credo GCT4L, 2-8°C shippers. The samples were processed according to CT-BW-SS-SOP-398, Gilead Specific Flow Cytometry Assay to Detect STAT3 in IL6 Stimulated Whole Blood, in triplicate by one operator. Mean, Standard deviation and %CVs were calculated between replicates. Percent stimulation was calculated for each donor as well using the following equation:

Equation 1: % stim =  $(stim - unstim)/unstim \times 100$ 

## **MATERIALS AND METHODS**

## Gilead pSTAT3 Stimulation Assay Method

The assay was performed according to CT-BW-SS-SOP-398, Gilead Specific Flow Cytometry Assay to Detect STAT3 in IL6 Stimulated Whole Blood.

### Reagents

The reagents utilized in the flow cytometric assays are listed below:

- CD3 FITC, clone UCHT1, BD Cat. No. 555916
- CD4 V450, clone RPA-T4, BD Cat No. 560345
- STAT3 PE, clone M59-50, BD Cat No. 560391
- pSTAT3-PE, (Y705), Clone 4/P-STAT3, BD Phosflow Cat No. 612569
- BD Lyse/Fix, BD Cat No. 558049
- BD Perm Buffer III BD PhosFlow Cat No. 558050
- BD Stain Buffer (FBS), BD Cat No. 554656
- Recombinant Human IL-6, R&D Systems Cat No. 206-IL-010
- PBS with 1% BSA Prepared according to CT-BW-REAG-SOP-14, Preparation of 1X Phosphate-Buffered Saline with 2% Bovine Albumin (PBS-BSA with azide), 1X Phosphate-



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

- PBS with 1% BSA Prepared according to CT-BW-REAG-SOP-14, Preparation of 1X
  Phosphate-Buffered Saline with 2% Bovine Albumin (PBS-BSA with azide), 1X PhosphateBuffered Saline with 1% Serum Bovine Albumin (PBS with 1% BSA with azide), and 0.5%
  Serum bovine Albumin (PBS-BSA without azide)
- Ammonium Chloride Based Whole Blood Lysing Reagent Prepared according to CT-BW-REAG-SOP-3, Preparation of Whole Blood Lysing Reagent
- 1% Paraformaldehyde Solution Prepared according to CT-BW-REAG-SOP-4, Preparation of 1%
   Paraformaldehyde Solution

## DATA ANALYSIS

After acquisition, the listmode files were analyzed offline using WinList [Verity Software] 7.0 to generate the reportables described above. Gating scheme is located in Appendix CC.

### **ABBREVIATIONS**

The following abbreviations may appear in the text of this report or in the attached tables.

- tSTA'13 Signal Transducer and Activator of Transcription 3, Total protein
- pSTAT3 Signal Transducer and Activator of Transcription 3, phosphorylated at Tyrosine residue 705
- Y Tyrosine
- %CV -- Coefficient of Variation = 100 x [Standard Deviation/Mean]
- DI Deionized
- ELISA Enzyme-Linked Immunosorbent Assay
- QC Quality Control
- RT Room Temperature (20 to 25°C)
- Universal Precautions -- Treating all patient samples as though they are infectious.
- FMO Fluorescence Minus One
- CD Cluster of Differentiation
- PBS-Phosphate buffered saline
- BSA Bovine Serum Albumin
- WBC White Blood Cell
- RBC Red Blood Cell
- FITC Fluorescein Isothiocyanate
- PE Phycoerythrin
- μL Microliter
- mL Milliliter
- BD Becton Dickinson
- QC Quality Control
- LCT LabCorp Clinical Trials
- RCF Relative Centrifugal Force
- FACSCanto II Fluorescence Activated Cell Sorter Canto II
- SOP Standard Operating Procedure



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

## REFERENCES

- CT-BW-SS-SOP-398, Gilead Specific Flow Cytometry Assay to Detect STAT3 in IL6 Stimulated Whole
- CT-BW-MAINT-SOP-30, Daily Startup, Shutdown, and Maintenance of the Becton Dickinson FACSCanto II Flow Cytometer
- CT-BW-MAINT-SOP-33, Daily Quality Control of the Becton Dickinson FACSCauto II (RUO)
   Flow Cytometer
- CT-BW-REAG-SOP-14, Preparation of 1X Phosphate-Buffered Saline with 2% Bovine Albumin (PBS-BSA with azide), 1X Phosphate-Buffered Saline with 1% Serum Bovine Albumin (PBS with 1% BSA with azide), and 0.5% Serum bovine Albumin (PBS-BSA without azide)
- CT-BW-REAG-SOP-3, Preparation of Whole Blood Lysing Reagent
- CT-BW-REAG-SOP-4, Preparation of 1% Paraformaldehyde Solution
- LA-LCT Assay Qualification Plan GEN82, Cross Laboratory Qualification of Human STAT3 [pY705] ELISA (cell lysate, units/mL)
- White paper: O'Hara et al. 2011. Recommendations for the validation of flow cytometric testing during drug development: Il assays. Journal of Immunological Methods. 363 120-134

## ACCEPTANCE CRITERIA

## Linearity Acceptance Criteria

The linearity was calculated by plotting the expected values at 2000 cells by the measured values a other cell densities. The relative error was then calculated between the values using the equation below:

Equation 2: ABSOLUTE VALUE of the following: %Relative Error (%RE) = [Accepted Value (@2000 cells) - Measured Value (@N-spike])/ Accepted Value (@2000 Cells)\*100.

Acceptance failed when the % Relative Error was greater than 25%. %CVs were also calculated between replicates in this phase. Acceptable %CVs for replicates was less than or equal to 20%

# Inter-Operator Precision Acceptance Criteria

%CVs was calculated between operators. %CV should be ≤25%, with the possible exception of those reportables derived from populations that are present at low frequencies (<5% of the primary population, i.e. lymphocytes). For these discrete populations, the %CV may be higher than 25%, but may not reflect any trend that would indicate that the ability to detect these populations is significantly affected by stability or donor variances between collections.

# Intra-Assay Precision Acceptance Criteria

%CVs was calculated within the replicates for Intra-Assay Precision. %CV should be ≤25% within donor replicates, with the possible exception of those reportables derived from populations that are present at low frequencies (<5% of the primary population, i.e. lymphocytes). For these discrete populations, the %CV may be higher than 25%, but may not reflect any trend that would indicate that the ability to detect these populations is significantly affected by stability or normal donor variances between collections.

## Assay Transfer

%CVs should be the same as Intra-Assay Precision. Additionally, the percentage of stimulation of pSTAT3 should be reflective of what has been seen in normal donors in the course of the validation in Phases I-III. Inter-Donor variability will be determined from data in Phase I-III. The stimulation percentage from Assay Transfer should be within this variability plus/minus 1 standard deviation.




Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

## RESULTS

## Phase I: Antibody Titration

This phase was conducted in order to titrate all reagents to saturation within the client method. Data for this phase is routinely held at LCT Brentwood facility. Titration results only are supplied as part of the validation report, The pSTAT3-PE was used at manufacturer recommended volume of  $20\mu L/\text{test}$ . The tSTAT3-PE was used at manufacturer recommended volume of  $20\mu L/\text{test}$ . The CD3-FITC was used at manufacturer recommended volume of  $20\mu L/\text{test}$ . The CD4-V450 was used at manufacturer recommended volume of  $5\mu L/\text{test}$ .

## Phase II: Assay Linearity

In order to determine the minimum number of lymphocytes required to accurately determine the MESF/MFI, the 2000 event sample was used as the basis for determining the relative error of the MESF/MFI and the % positivity. Data for Linearity experiments are located in Appendices A-R. %CVs that are greater than 20% are flagged in red font throughout the tables. The CVs for pSTAT3 percentages, MFIs and MESFs were consistently acceptable in Donors 2 and 3 for all region counts of greater than 100 events. Donor 1 demonstrated increased variability in the 300 event sample due to an outlier in replicate 2. The calculated %RE reflected these same results, with the acceptance criteria of less than 25% RE being met when greater than 100 events were acquired for Donors 2 and 3, and greater than 300 events for Donor 1. All data outside acceptance criteria are flagged in red within the data tables. For the course of the study, the window of acquisition was set such that greater than 300 events must be acquired (actual stop gate was set to 10,000 lymphocytes).

## Phase III: Inter-Operator and Intra-Assay Precision

A minimum of 2 normal whole blood specimens were drawn into NaHeparin. The samples were shipped to back to the Brentwood LCT within 1 Day ex-vivo using the Credo GTC4L, 2-8°C shippers from World Courier. The samples were tested immediately within the panel by 2 operators in triplicate. The acquisition stop gate was set to acquire 2000 lymphocytes per client request in this phase. Data for this phase are located in Appendices S-W. %CVs outside of the acceptance range occurred for inter-operator only for the %pSTAT3 unstimulated in the CD3+ lymphs and CD3+/CD4+ lymphs, though MESF values for these same populations were acceptable. These values are marked in red. All other values were within acceptance criteria.

# Phase IV: Assay Transfer -- ELISA testing only

Reference LA-LCT Assay Qualification Plan GEN82, Cross Laboratory Qualification of Human STAT3 [pY705] ELISA (cell lysate, units/mL). Data are not included in this report.

# Phase IV: Assay Transfer – Flow Cytometry testing only

The Brentwood facility drew 3 NWB donors and ship to LCT Cranford flow lab using World Courier Credo GCT4L, 2-8°C shippers. The samples were processed according to CT-BW-SS-SOP-398, Gilead Specific Flow Cytometry Assay to Detect STAT3 in IL6 Stimulated Whole Blood, in triplicate by one operator. Mean, Standard deviation and %CVs were calculated between replicates. Data for the replicate statistics and raw data are located in Appendices X-BB. Values outside acceptance criteria are marked in red font. There was one outlier in the percentage of both total and phospho STAT3 in the CD3 and CD3+/CD4+ populations for Donor 2A and Donor 3A samples. The other 2 replicates were within acceptable ranges. The primary parameters of interest are the MFI and the MESF measurements, so the assay transfer is acceptable, as these are within acceptance guidelines. In addition, in Appendix DD, the percentage of stimulation was calculated for each normal donor tested in all validation phases. The mean and standard deviation, then mean + 1 standard deviation and mean -1 standard deviation were calculated. All percentages of stimulations that did



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

not fall within the Mean +/- 1StDev were flagged in pink highlight with red font. All AT samples were within acceptance criteria. Precision Donor 2 and Linearity Donor 1 were outside the 1 standard deviation in the % stimulation based on the MESF in CD3+ (Lymphs). These values were lower in these 2 donors than any other. This is considered normal for these donors.

### Conclusion

These experiments demonstrate that the Gilead pSTAT3 Stimulation Assay is performed with precision. Specimens were received and analyzed up to Day 2 (48-54 hours, per client internal data, not included) when collected in sodium heparin vacutainers and shipped/stored at 2-8°C. The assay transfer experiments to the Cranford Laboratory demonstrated equivalent stimulation and biological variability as seen within the validation studies.

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

# Appendix A: Table 1, Linearity - Healthy Donors 1-3

| Linearity Table 1 | Acquisition Date | %Lymphs | Region Events<br>CD3+ Lymphs | %CD3+ [Lymphs] | Region Events<br>CD3+/CD4+<br>Lymphs | %CD3+/CD4<br>[Lymphs] | MESF FMO-PE<br>unstim [CD3+<br>Lymphs] | MESF FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %tSTAT3 unstim |
|---|---|---|---|---|---|---|---|---|---|
| D1-2000-R1 | 2/5/2014 | 34.1 | 1369 | 77.8 | 608 | 44.4 | 533 | 533 | |
| D1-2000-R2 | 2/5/2014 | 31.4 | 1382 | 78.7 | 581 | 42.0 | 515 | 459 | 41.4 |
| D1-2000-R3 | 2/5/2014 | 33.9 | 1437 | 79.4 | 629 | 43.8 | 540 | 540 | 37.5<br>37.1 |
| Me | | 33.1 | 1396 | 78.6 | 606 | 43.4 | 529 | 511 | |
| Str | | 1.5 | 36.1 | 0.8 | 24.1 | 1.2 | 12.9 | 44.9 | 38.7 |
| %( | | 4.5 | 2.6 | 1.0 | 4.0 | 2.8 | 2.4 | 8.8 | 6.2 |
| D1-1000-R1 | 2/5/2014 | 33.0 | 686 | 76.9 | 261 | 38.1 | 548 | 540 | |
| D1-1000-R2 | 2/5/2014 | 32.6 | 690 | 77.6 | 299 | 43.3 | 533 | 540 | 38.3 |
| D1-1000-R3 | 2/5/2014 | 32.2 | 683 | 78.3 | 297 | 43.5 | 536 | 504 | 31.2 |
| Me | | 32.6 | 686 | 77.6 | 286 | 41.6 | 539 | 528 | 36.6 |
| Str | | 0.4 | 3.5 | 0.7 | 21.4 | 3.1 | 7.9 | | 35.4 |
| %6 | | 1.2 | 0.5 | 0.9 | 7.5 | 7.5 | 1.5 | 20.8 | 3.7 |
| D1-500-R1 | 2/5/2014 | 31.8 | 354 | 79.2 | 173 | 48.9 | 524 | | 10.5 |
| D1-500-R2 | 2/5/2014 | 32,9 | 347 | 77,5 | 127 | 36.6 | 571 | 507 | 31.7 |
| D1-500-R3 | 2/5/2014 | 33.7 | 358 | 78,5 | 151 | 42.2 | 588 | 557 | 30.3 |
| Me | an | 32.8 | 353 | 78.4 | 150 | 42.6 | 561 | 597 | 27.3 |
| Sto | )ev | 1.0 | 5.6 | 0,9 | 23.0 | 6.2 | 33.2 | 554 | 29.8 |
| %( | V | 3.0 | 1.6 | 1,1 | 15.3 | 14.6 | 5.9 | 45.1 | 2.2 |
| D1-300-R1 | 2/5/2014 | 30.8 | 213 | 79.8 | 86 | 40.4 | 540 | 8.1 | 7.4 |
| D1-300-R2 | 2/5/2014 | 35.9 | 199 | 71.8 | 89 | 44.7 | 531 | 589 | 29.0 |
| D1-300-R3 | 2/5/2014 | 32.0 | 221 | 80.7 | 100 | 45.3 | 570 | 586 | 24.6 |
| Me | an | 32.9 | 211 | 77.4 | 92 | 43.5 | 547 | 588 | 21.6 |
| StD | ev | 2.7 | 11.1 | 4.9 | 7.4 | 2.7 | | 588 | 25.1 |
| %( | V | 8.2 | 5.3 | 6.3 | 8.0 | 6.2 | 3.7 | 1.5 | 3.7 |
| D1-100-R1 | 2/5/2014 | 34,6 | 71 | 84.5 | 36 | 50.7 | | 0.3 | 14.7 |
| D1-100-R2 | 2/5/2014 | 32.0 | 71 | 76.3 | 26 | 36.6 | 582 | 537 | 19.4 |
| D1-100-R3 | 2/5/2014 | 32.3 | 65 | 75.6 | 21 | 32.3 | 575 | 647 | 23.7 |
| Me | | 33.0 | 69 | 78.8 | 28 | | 547 | 504 | 13.0 |
| StD | ev | 1.4 | 3,5 | 4.9 | 7.6 | 39.9<br>9.6 | 568 | 563 | 18.7 |
| %0 | V | 4.2 | 5.1 | 6.2 | 27.1 | 24.1 | 18.5 | 74,9 | 5.4 |
| D1-50-R1 | 2/5/2014 | 31.9 | 38 | 86.4 | 15 | 39.5 | 3.3 | 13.3 | 28.9 |
| D1-50-R2 | 2/5/2014 | 24.6 | 37 | 84.1 | 22 | 59.5<br>59.5 | 507 | 413 | 32.4 |
| D1-50-R3 | 2/5/2014 | 32.4 | 30 | 66.7 | 11 | 36.7 | 501 | 771 | 9.1 |
| Me | | 29.6 | 35 | 79.1 | 16 | | 519 | 655 | 14.3 |
| StD | | 4.4 | 4.4 | 10.8 | 5,6 | 45.2 | 509 | 613 | 18.6 |
| %0 | | 14.9 | 12.6 | 13.7 | 35.0 | 12.4<br>27.4 | 9.2 | 182.7 | 12.2 |
| | | | 4440 | 4.245 | 23,0 | 27.4 | 1.8 | 29.8 | 65,6 |





Appendix B: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Linearity Table 1<br>Continued | Acquisition Date | %STAT3 unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>unstim [CD3+<br>Lymphs] | MESF tSTAT3 unstim [CD3+/CD4+ Lymphs] | %pSTAT3 unstim | %pSTAT3 unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>unstim [CD3+<br>Lymphs] | MESF pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF FMO-PE<br>STIM [CD3+<br>Lymphs] | MESF FMO-PE<br>STIM [CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| D1-2000-R1 | 2/5/2014 | 54.4 | 1669 | 1686 | 2.6 | 6.4 | 739 | 777 | 520 | 506 |
| D1-2000-R2 | 2/5/2014 | 48.0 | 1618 | 1607 | 2.8 | 6.3 | 734 | 790 | 520 | 532 |
| D1-2000-R3 | 2/5/2014 | 49.0 | 1611 | 1509 | 1.8 | 4.9 | 733 | 815 | 538 | 533 |
| Me | ean | 50.5 | 1633 | 1634 | 2.4 | 5.9 | 735 | 794 | 526 | 524 |
| St | Dev | 3.4 | 31.7 | 45.0 | 0.5 | 0.8 | 3.2 | 19.3 | 10.4 | 15.3 |
| % | CV | 6.7 | 1.9 | 2.8 | 20.8 | 13.6 | 0.4 | 2.4 | 2.0 | 2.9 |
| D1-1000-R1 | 2/5/2014 | 44.9 | 1607 | 1581 | 3.1 | 6.6 | 746 | 800 | 555 | 569 |
| D1-1000-R2 | 2/5/2014 | 42.7 | 1563 | 1557 | 3.1 | 7.5 | 751 | 837 | 542 | 504 |
| D1-1000-R3 | 2/5/2014 | 44.4 | 1562 | 1543 | 1.9 | 5.7 | 757 | 818 | 538 | 517 |
| M | ean | 44.0 | 1577 | 1560 | 2.7 | 6.6 | 751 | 818 | 545 | 530 |
| St | Dev | 1.2 | 25.7 | 19.2 | 0.7 | 0.9 | 5.5 | 18.5 | 8.9 | 34.4 |
| % | CV | 2.7 | 1,6 | 1.2 | 25,9 | 13.6 | 0.7 | 2.3 | 1.6 | 6.5 |
| D1-500-R1 | 2/5/2014 | 44.7 | 1504 | 1537 | 2.3 | 7.0 | 713 | 805 | 557 | 580 |
| D1-500-R2 | 2/5/2014 | 36.0 | 1479 | 1456 | 3.2 | 6.2 | 756 | 813 | 571 | 570 |
| D1-500-R3 | 2/5/2014 | 37.3 | 1523 | 1429 | 2.0 | 5.8 | 743 | 820 | 565 | 549 |
| M | ean | 39.3 | 1502 | 1474 | 2.5 | 6.3 | 737 | 813 | 564 | 566 |
| St | Dev | 4.7 | 22.1 | 56.2 | 0.6 | 0.6 | 22.1 | 7.5 | 7.0 | 15.8 |
| % | .cv | 12.0 | 1.5 | 3.8 | 24.0 | 9.5 | 3.0 | 0.9 | 1.2 | 2.8 |
| D1-300-R1 | 2/5/2014 | 44.4 | 1463 | 1451 | 0.9 | 2.0 | 754 | 754 | 577 | 582 |
| D1-300-R2 | 2/5/2014 | 37.4 | 1488 | 1547 | 2.4 | 4.8 | 747 | 805 | 580 | 589 |
| D1-300-R3 | 2/5/2014 | 32.4 | 1429 | 1403 | 1.4 | 8.1 | 753 | 815 | 560 | 501 |
| M | ean | 38.1 | 1460 | 1467 | 1,6 | 5.0 | 751 | 791 | 572 | 557 |
| St | Dev | 6.0 | 29.6 | 73.3 | 0.8 | 3.1 | 3.8 | 32.7 | 10.8 | 48.9 |
| 9/ | CV | 15.7 | 2.0 | 5.0 | 50.0 | 62.0 | 0.5 | 4.1 | 1,9 | 8.8 |
| D1-100-R1 | 2/5/2014 | 26.9 | 1398_ | 1343 | 2.9 | 6.1 | 735 | 790 | 557 | 509 |
| D1-100-R2 | 2/5/2014 | 38.5 | 1351 | 1411 | 1.5 | 3.5 | 667 | 761 | 440 | 343 |
| D1-100-R3 | 2/5/2014 | 21.9 | 1414 | 1420 | 0.0 | 5.0 | 724 | 841 | 582 | 495 |
| М | ean | 29.1 | 1388 | 1391 | 1.5 | 4.9 | 709 | 797 | 526 | 449 |
| St | Dev | 8.5 | 32,7 | 42.1 | 1.5 | 1,3 | 36.5 | 40.5 | 75.8 | 92.1 |
| 9 | .cv | 29.2 | 2.4 | 3.0 | 100.0 | 26.5 | 5.1 | 5,1 | 14.4 | 20.5 |
| D1-50-R1 | 2/5/2014 | 37.5 | 1447 | 1484 | 0.0 | 4.8 | 676 | 672 | 808 | 582 |
| D1-50-R2 | 2/5/2014 | 41.2 | 1420 | 1550 | 2.9 | 5,9 | 788 | 771 | 512 | 478 |
| D1-50-R3 | 2/5/2014 | 30.8 | 1178 | 1351 | 3.1 | 5.6 | 825 | 857 | 631 | 582. |
| М | ean | 36.5 | 1348 | 1462 | 2.0 | 5.4 | 763 | 767 | 650 | 547 |
| St | Dev | 5.3 | 148.1 | 101.4 | 1.7 | 0.6 | 77.6 | 92.6 | 148.9 | 60.0 |
| 9 | cv | 14.5 | 11.0 | 6.9 | 85.0 | 11.1 | 10.2 | 12.1 | 22.9 | 11.0 |





# Appendix C: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Linearity Table 1<br>Continued | Acquisition Date | %LSTAT3 STIM<br>[CD3+ Lymphs] | %STAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3 STIM [CD3+ Lymphs] | MESF tSTAT3<br>STIM [CD3+/CD4+<br>Lymphs] | %pSTAT3 STIM<br>[CD3+ Lymphs] | %pSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF pSTAT3<br>STIM [CD3+/CD44<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|
| D1-2000-R1 | 2/5/2014 | 38.4 | 47.4 | 1625 | 1597 | 54.7 | 93.8 | 3063 | |
| D1-2000-R2 | 2/5/2014 | 36,2 | 46.9 | 1610 | 1585 | 53.3 | 92.8 | 2365 | 10779<br>10704 |
| D1-2000-R3 | 2/5/2014 | 35.3 | 45.4 | 1584 | 1566 | 54.7 | 93.6 | 3039 | 10463 |
| Me | | 36.6 | 46.6 | 1606 | 1583 | 54.2 | 93.4 | 2822 | |
| Sti | | 1.6 | 1.0 | 20.7 | 15.6 | 0.8 | 0.5 | 396.2 | 10649<br>165.1 |
| % | | 4.4 | 2.1 | 1.3 | 1.0 | 1.5 | 0.5 | 14.0 | 1.6 |
| D1-1000-R1 | 2/5/2014 | 34.7 | 44.4 | 1551 | 1534 | 53.2 | 95.4 | 2600 | |
| D1-1000-R2 | 2/5/2014 | 28.9 | 39.4 | 1500 | 1487 | 55.4 | 93.7 | 2885 | 10568<br>10367 |
| D1-1000-R3 | 2/5/2014 | 32,4 | 39.8 | 1562 | 1547 | 55.1 | 95.3 | 2882 | |
| Me | ean | 32.0 | 41.2 | 1538 | 1523 | 54.6 | 94.8 | 2789 | 10159 |
| Str | | 2.9 | 2.8 | 33.1 | 31.6 | 1.2 | 1,0 | 163.7 | 10365 |
| % | | 9.1 | 6.8 | 2.2 | 2.1 | 2.2 | 1.1 | 5.9 | 204.5 |
| D1-500-R1 | 2/5/2014 | 28.4 | 35.3 | 1512 | 1461 | 57.6 | 93.6 | 4558 | 2.0 |
| D1-500-R2 | 2/5/2014 | 30.1 | 35.8 | 1525 | 1400 | 47.8 | 92.1 | 1456 | 9971 |
| D1-500-R3 | 2/5/2014 | 22.9 | 25,9 | 1420 | 1381 | 53.9 | 91.4 | 2891 | 10096 |
| Me | an | 27.1 | 32.3 | 1486 | 1414 | 53.1 | 92.4 | 2968 | 9924 |
| StDev | | 3.8 | 5.6 | 57.2 | 41.8 | 4,9 | 1.1 | 1552.4 | 9997 |
| % | | 14.0 | 17.3 | 3.8 | 3.0 | 9.2 | 1.2 | 52,3 | 88.9 |
| D1-300-R1 | 2/5/2014 | 32.4 | 38.0 | 1527 | 1490 | 49.3 | 95.4 | 1670 | 0.9 |
| D1-300-R2 | 2/5/2014 | 21.8 | 30.4 | 1405 | 1405 | 54.8 | 92.1 | 3116 | 10646 |
| D1-300-R3 | 2/5/2014 | 22.8 | 29.6 | 1420 | 1405 | 58.8 | 94.0 | 3665 | 9368 |
| Me | | 25.7 | 32.7 | 1451 | 1433 | 54.3 | 93.8 | 2817 | 9555 |
| StDev | | 5.9 | 4.6 | 66.5 | 49.1 | 4.8 | 1.7 | 1030.6 | 9856 |
| %( | | 23.0 | 14.1 | 4.6 | 3.4 | 8,8 | 1.8 | 36,6 | 690.2<br>7.0 |
| D1-100-R1 | 2/5/2014 | 26.9 | 31.8 | 1507 | 1530 | 54.9 | 97.2 | 5196 | |
| D1-100-R2 | 2/5/2014 | 18.6 | 21.7 | 1272 | 1254 | 46.5 | 88.5 | 1589 | 8829<br>9281 |
| D1-100-R3 | 2/5/2014 | 28.4 | 39.4 | 1377 | 1407 | 43.1 | 90.5 | 1285 | |
| Me | | 24.6 | 31.0 | 1385 | 1397 | 48,2 | 92.1 | 2690 | 8347 |
| StE | | 5.3 | 8.9 | 117.7 | 138.3 | 6.1 | 4.5 | 2175.6 | 8819 |
| %( | | 21.5 | 28.7 | 8.5 | 9.9 | 12.7 | 5.0 | 80.9 | 467.1<br>5.3 |
| D1-50-R1 | 2/5/2014 | 13.8 | 25.0 | 1193 | 1156 | 68.4 | 100.0 | 6627 | |
| D1-50-R2 | 2/5/2014 | 10.5 | 40.0 | 1277 | 1550 | 67.6 | 95.5 | 5005 | 11689 |
| D1-50-R3 | 2/5/2014 | 20.0 | 27.8 | 1407 | 1215 | 43,3 | 90.9 | 1474 | 8720 |
| Me | | 14.8 | 30.9 | 1292 | 1307 | 59.8 | 95.5 | 4369 | 7368 |
| StE | | 4.8 | 8.0 | 107.8 | 212.5 | 14.3 | 4.6 | 2634.8 | 9259 |
| %( | CV | 32.4 | 25.9 | 8.3 | 16.3 | 23.9 | 4.8 | 2634.8<br>50.3 | 2210.4 |



Appendix D: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Linearity Table 1 | Acquisition Date | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[GD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim [CD3+<br>Lymphs] | MFI pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|
| D1-2000-R1 | 2/5/2014 | 218 | 218 | 665 | 671 | 300 | 315 |
| D1-2000-R2 | 2/5/2014 | 211 | 188 | 645 | 641 | 298 | 320 |
| D1-2000-R3 | 2/5/2014 | 221 | 221 | 642 | 641 | 298 | 330 |
| | ean | 217 | 209 | 651 | 651 | 299 | 322 |
| | Dev | 5.1 | 18.2 | 12.5 | 17.3 | 1.2 | 7.6 |
| | CV | 2.4 | 8.7 | 1.9 | 2.7 | 0.4 | 2.4 |
| D1-1000-R1 | 2/5/2014 | 224 | 221 | 641 | 631 | 303 | 324 |
| D1-1000-R2 | 2/5/2014 | 218 | 221 | 623 | 621 | 305 | 339 |
| D1-1000-R3 | 2/5/2014 | 219 | 207 | 623 | 616 | 307 | 331 |
| | ean | 220 | 216 | 629 | 623 | 305 | 331 |
| | Dev | 3.2 | 8.1 | 10.4 | 7.6 | 2.0 | 7.5 |
| | cv | 1.5 | 3.8 | 1.7 | 1.2 | 0.7 | 2.3 |
| D1-500-R1 | 2/5/2014 | 214 | 208 | 601 | 613 | 290 | 326 |
| D1-500-R2 | 2/5/2014 | 233 | 228 | 591 | 582 | 307 | 329 |
| D1-500-R3 | 2/5/2014 | 240 | 243 | 608 | 571 | 302 | 332 |
| Mean | | 229 | 226 | 600 | 589 | 300 | 329 |
| StDev | | 13.5 | 17.6 | 8.5 | 21.8 | 8.7 | 3.0 |
| % | CV CV | 5.9 | 7.8 | 1,4 | 3.7 | 2.9 | 0.9 |
| D1-300-R1 | 2/5/2014 | 221 | 241 | 585 | 580 | 306 | 306 |
| D1-300-R2 | 2/5/2014 | 217 | 239 | 594 | 617 | 303 | 326 |
| D1-300-R3 | 2/5/2014 | 233 | 240 | 571 | 561 | 306 | 330 |
| | ean | 224 | 240 | 583 | 586 | 305 | 321 |
| St | Dev | 8.3 | 1.0 | 11.6 | 28.5 | 1.7 | 12.9 |
| 0/6 | CV CV | 3.7 | 0.4 | 2.0 | 4.9 | 0.6 | 4.0 |
| D1-100-R1 | 2/5/2014 | 238 | 220 | 559 | 538 | 298 | 320 |
| D1-100-R2 | 2/5/2014 | 235 | 264 | 541 | 564 | 271 | 309 |
| D1-100-R3 | 2/5/2014 | 224 | 207 | 566 | 568 | 294 | 340 |
| | ean | 232 | 230 | 555 | 557 | 288 | 323 |
| | Dev | 7.4 | 29.9 | 12.9 | 16.3 | 14.6 | 15.7 |
| 9/ | oCV | 3.2 | 13.0 | 2.3 | 2.9 | 5.1 | 4.9 |
| D1-50-R1 | 2/5/2014 | 208 | 170 | 578 | 593 | 275 | 273 |
| D1-50-R2 | 2/5/2014 | 205 | 313 | 568 | 618 | 319 | 313 |
| D1-50-R3 | 2/5/2014 | 212 | 267 | 473 | 541 | 334 | 347 |
| | ean | 208 | 250 | 540 | 584 | 309 | 311 |
| | Dev | 3.5 | 73.0 | 58.0 | 39.3 | 30.7 | 37.0 |
| | 6CV | 1.7 | 29.2 | 10.7 | 6.7 | 9.9 | 11.9 |



Appendix E: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Linearity Table 1 Continued | Acquisition Date | MFI FMO-PE STIM<br>[CD3+ Lymphs] | MFI FMO-PE STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3 STIM<br>[CD3+ Lymphs] | MFI tSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3 STIM | MFI pSTAT3 STIN<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|
| D1-2000-R1 | 2/5/2014 | 213 | 207 | 648 | 637 | 1203 | 4113 |
| D1-2000-R2 | 2/5/2014 | 213 | 218 | 642 | 632 | 935 | 4085 |
| D1-2000-R3 | 2/5/2014 | 220 | 218 | 632 | 625 | 1194 | 3995 |
| | ean | 215 | 214 | 641 | 631 | 1111 | 4064 |
| | Dev | 4.0 | 6.4 | 8.1 | 6.0 | 152.2 | 61.7 |
| | CV | 1.9 | 3.0 | 1.3 | 1.0 | 13.7 | 1.5 |
| D1-1000-R1 | 2/5/2014 | 227 | 232 | 619 | 612 | 1025 | 4034 |
| D1-1000-R2 | 2/5/2014 | 222 | 207 | 599 | 594 | 1135 | |
| D1-1000-R3 | 2/5/2014 | 220 | 212 | 623 | 617 | 1134 | 3959 |
| Me | ean | 223 | 217 | 614 | 608 | 1098 | 3881 |
| St | Dev | 3.6 | 13.2 | 12.9 | 12.1 | 63.2 | 3958 |
| % | CV | 1.6 | 6.1 | 2,1 | 2.0 | 5.8 | 76.5 |
| D1-500-R1 | 2/5/2014 | 228 | 237 | 604 | 584 | 1774 | 1.9 |
| D1-500-R2 | 2/5/2014 | 233 | 233 | 609 | 560 | 582 | 3811 |
| D1-500-R3 | 2/5/2014 | 231 | 225 | 568 | 553 | 1137 | 3858 |
| Me | ean | 231 | 232 | 594 | 566 | | 3794 |
| Sti | Dev | 2.5 | 6.1 | 22,4 | 16.3 | 1164 | 3821 |
| % | CV | 1.1 | 2.6 | 3.8 | 2,9 | 596.5<br>51.2 | 33.2 |
| D1-300-R1 | 2/5/2014 | 235 | 238 | 610 | 595 | | 0.9 |
| D1-300-R2 | 2/5/2014 | 237 | 241 | 562 | 562 | 665 | 4063 |
| D1-300-R3 | 2/5/2014 | 229 | 205 | 568 | 562 | 1224 | 3586 |
| Me | ean | 234 | 228 | 580 | 573 | 1434 | 3656 |
| Sti | Dev | 4,2 | 20.0 | 26.2 | 19.1 | 1108 | 3768 |
| | CV | 1.8 | 8.8 | 4.5 | 3.3 | 397.5 | 257.6 |
| D1-100-R1 | 2/5/2014 | 228 | 208 | 602 | | 35.9 | 6.8 |
| D1-100-R2 | 2/5/2014 | 181 | 142 | 510 | 611 | 2016 | 3384 |
| D1-100-R3 | 2/5/2014 | 238 | 203 | 551 | 503<br>563 | 634 | 3553 |
| Me | ean | 216 | 184 | 554 | | 515 | 3204 |
| | Dev | 30,4 | 36.7 | 46.1 | 559 | 1055 | 3380 |
| | CV | 14.1 | 19.9 | 8.3 | 54.1 | 834.4 | 174.5 |
| D1-50-R1 | 2/5/2014 | 327 | 238 | 479 | 9.7 | 79.1 | 5.2 |
| D1-50-R2 | 2/5/2014 | 210 | 196 | 512 | 464 | 2557 | 4452 |
| D1-50-R3 | 2/5/2014 | 257 | 238 | 563 | 618 | 1944 | 3343 |
| Me | | 265 | 224 | | 488 | 563 | 488 |
| Stu | | 58.9 | 24.2 | 518 | 523 | 1688 | 2761 |
| % | | 22.2 | 10.8 | 42.3 | 82.9 | 1021.4 | 2045.1 |
| ,,, | | Si this Sa | 10.9 | 8.2 | 15.9 | 60.5 | 74.1 |



## Appendix F: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1: Linearity | Acquisition<br>Date | %Lymphs | Region Events CD3+<br>Lymphs | %CD3+ [Lymphs] | Region Events<br>CD3+/CD4+<br>Lymphs | %CD3+/CD4<br>[Lymphs] | MESF FMO-PE<br>unstim [CD3+<br>'Lymphs] | MESF FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %tSTAT3 unstin |
|---|---|---|---|---|---|---|---|---|---|
| D2-2000-R1 | 2/5/2014 | 13.8 | 1427 | 72.7 | 1055 | 73.9 | 418 | 414 | 88.6 |
| D2-2000-R2 | 2/5/2014 | 18.6 | 1391 | 71.5 | 1027 | 73.8 | 430 | 425 | 84.7 |
| 02-2000-R3 | 2/5/2014 | 19.1 | 1416 | 72.8 | 1031 | 72.8 | 412 | 409 | 85.2 |
| Mean | | 18,8 | 1411 | 72.3 | 1038 | 73.5 | · 420 | 416 | 86.2 |
| StDev | | 0.3 | 18.4 | 0.7 | 15.1 | 0.6 | 9.2 | 8,2 | 2.1 |
| %CV | | 1,6 | 1.3 | 1.0 | 1.5 | 0.8 | 2.2 | 2.0 | 2.4 |
| D2-1000-R1 | 2/5/2014 | 18.2 | 684 | 70.6 | 492 | 71.9 | 385 | 380 | 85.0 |
| D2-1000-R1 | 2/5/2014 | 19.0 | 709 | 72.3 | 515 | 72.6 | 428 | 432 | 81.5 |
| D2-1000-R3 | 2/5/2014 | 18.7 | 715 | 73.5 | 525 | 73.4 | 432 | 413 | 82.9 |
| Mean | 2727201 | 18.6 | 703 | 72.1 | 511 | 72.6 | 415 | 408 | 83.1 |
| StDev | | 0,4 | 16.4 | 1.5 | 16.9 | 0.8 | 26.1 | 26,3 | 1.8 |
| %CV | | 2.2 | 2.3 | 2.1 | 3.3 | 1.1 | 6.3 | 6.4 | 2.2 |
| D2-500-R1 | 2/5/2014 | 18.4 | 336 | 68.7 | 258 | 76.8 | 398 | 393 | 78.8 |
| D2-500-R2 | 2/5/2014 | 17.8 | 323 | 68.0 | 246 | 76.2 | 398 | 383 | 64.4 |
| D2-500-R3 | 2/5/2014 | 18.8 | 350 | 71.4 | 262 | 74.9 | 477 | 457 | 64.1 |
| Mean | Ed Of East 1 | 18.3 | 336 | 69.4 | 255 | 76.0 | 424 | 411 | 69.1 |
| StDev | | 0.5 | 13.5 | 1.8 | 8.3 | 1.0 | 45.6 | 40.1 | 8.4 |
| %CV | | 2.7 | 4.0 | 2.6 | 3.3 | 1.3 | 10.8 | 9.8 | 12.2 |
| D2-300-R1 | 2/5/2014 | 17.8 | 211 | 72.3 | 154 | 73.0 | 468 | 477 | 63.5 |
| D2-300-R1 | 2/5/2014 | 21.5 | 217 | 71.9 | 157 | 72.4 | 474 | 526 | 64.0 |
| D2-300-R3 | 2/5/2014 | 18.0 | 210 | 71.7 | 160 | 76,2 | 469 | 467 | 54.0 |
| Mean | 2; 3/2014 | 19.1 | 213 | 72.0 | 157 | 73.9 | 470 | 490 | 60.5 |
| StDev | | 2.1 | 3.8 | 0.3 | 3.0 | 2.0 | 3.2 | 31.6 | 5.6 |
| %CV | | 11.0 | 1.8 | 0,4 | 1.9 | 2.7 | 0.7 | 6.4 | 9.3 |
| D2-100-R1 | 2/5/2014 | 17.4 | 71 | 70.3 | 59 | 83.1 | 564 | 655 | 53.7 |
| D2-100-R1<br>D2-100-R2 | 2/5/2014 | 22.6 | 67 | 69.8 | 49 | 73.1 | 426 | 403 | 52.4 |
| D2-100-R2<br>D2-100-R3 | 2/5/2014 | 19.1 | 69 | 70.4 | 50 | 72.5 | 481 | 480 | 51.4 |
| Mean | 2/3/2014 | 19.7 | 69 | 70.2 | 53 | 76.2 | 490 | 513 | 52.5 |
| StDev | | 2.7 | 2.0 | 0.3 | 5.5 | 6.0 | 69.5 | 129.1 | 1.2 |
| %CV | | 13.7 | 2,9 | 0.4 | 10.4 | 7.9 | 14.2 | 25.2 | 2.3 |
| D2-50-R1 | 2/5/2014 | 20.3 | 33 | 68,8 | 26 | 78.8 | 627 | 465 | 61.9 |
| D2-50-R1<br>D2-50-R2 | 2/5/2014 | 13.6 | 33 | 67.4 | 25 | 75.8 | 480 | 501 | 42.4 |
| D2-50-R2 | 2/5/2014 | 22.7 | 41 | 83.7 | 28 | 68.3 | 480 | 501 | 45.2 |
| Mean Mean | 2/3/2017 | 20.5 | 36 | 73.3 | 26 | 74.3 | 529 | 489 | 49.8 |
| StDev | | 2.1 | 4.6 | 9.0 | 1.5 | 5.4 | 84.9 | 20.8 | 10.5 |
| %CV | | 10.2 | 12.8 | 12.3 | 5.8 | 7.3 | 16.0 | 4.3 | 21.1 |

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

Appendix G: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1:<br>Linearity -<br>Continued | Acquisition<br>Date | %tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3 unstim [CD3+ Lymphs] | MESF tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3<br>unstim [CD3+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3 unstim [CD3+ Lymphs] | MESF pSTAT3 unstim [CD3+/CD4+ Lymphs] | MESF FMO-PE<br>STIM [CD3+<br>Lymphs] | MESF FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| D2-2000-R1 | 2/5/2014 | 83.3 | 1852 | 1848 | 50.1 | 51.9 | 1238 | 1407 | 434 | 423 |
| D2-2000-R2 | 2/5/2014 | 79.4 | 1761 | 1758 | 50.7 | 51.1 | 1245 | 1386 | 451 | 423 |
| D2-2000-R3 | 2/5/2014 | 79.0 | 1779 | 1764 | 48.5 | 52.0 | 1202 | 1405 | 454 | 435 |
| Me | ean | 80.6 | 1797 | 1790 | 49.8 | 51.7 | 1228 | 1399 | 446 | 437 |
| | Dev | 2,4 | 48.2 | 50.3 | 1.1 | 0.5 | 23.1 | 11.6 | 10.8 | 14.6 |
| % | CV | 3.0 | 2.7 | 2.8 | 2.2 | 1.0 | 1.9 | 0.8 | 2.4 | 3.3 |
| D2-1000-R1 | 2/5/2014 | 79.7 | 1707 | 1702 | 44.3 | 47.4 | 1137 | 1301 | 454 | |
| D2-1000-R2 | 2/5/2014 | 76.2 | 1692 | 1688 | 48.5 | 52.2 | 1204 | 1390 | 450 | 449 |
| D2-1000-R3 | 2/5/2014 | 75.6 | 1642 | 1662 | 49.7 | 50.5 | 1225 | 1368 | 442 | 435 |
| Me | ean | 77.2 | 1680 | 1684 | 47.5 | 50.0 | 1189 | 1353 | | 438 |
| St | Dev | 2.2 | 34.0 | 20.3 | 2.8 | 2,4 | 46.0 | 46:4 | 449 | 441 |
| % | CV | 2.8 | 2.0 | 1.2 | 5.9 | 4,8 | 3.9 | 3.4 | 6.1 | 7.4 |
| D2-500-R1 | 2/5/2014 | 70.8 | 1587 | 1599 | 47.9 | 49.6 | 1194 | | 1.4 | 1.7 |
| D2-500-R2 | 2/5/2014 | 53.7 | 1415 | 1422 | 52.7 | 53.1 | 1296 | 1340 | 383 | 398 |
| D2-500-R3 | 2/5/2014 | 52.0 | 1400 | 1403 | 46.8 | 48.6 | 1178 | 1447 | 440 | 418 |
| Me | an | 58.8 | 1467 | 1475 | 49.1 | 50.4 | 1223 | 1332 | 498 | 481 |
| | Dev | 10.4 | 103.9 | 108.1 | 3.1 | 2.4 | | 1373 | 440 | 432 |
| | CV | 17.7 | 7.1 | 7.3 | 6.3 | 4.8 | 64.0<br>5.2 | 64.2 | 57.5 | 43.3 |
| D2-300-R1 | 2/5/2014 | 52.8 | 1389 | 1408 | 47.0 | 52.4 | 1161 | 4.7 | 13.1 | 10.0 |
| D2-300-R2 | 2/5/2014 | 51.7 | 1418 | 1389 | 49.5 | 52.1 | | 1432 | 511 | 511 |
| D2-300-R3 | 2/5/2014 | 46.0 | 1269 | 1323 | 4 54.0 | 53.5 | 1225 | 1429 | 492 | 480 |
| | an | 50.2 | 1359 | 1373 | 50.2 | 52.7 | 1318 | 1433 | 451 | 437 |
| | Dev | 3.7 | 79.0 | 44.6 | 3.5 | 0.7 | 1235 | 1431 | 485 | 476 |
| | CV | 7.4 | 5.8 | 3.2 | 7.0 | | 78.9 | 2.1 | 30.7 | 37.2 |
| D2-100-R1 | 2/5/2014 | 51.9 | 1301 | 1385 | 41.3 | 1.3 | 6.4 | 0.1 | 6.3 | 7.8 |
| D2-100-R2 | 2/5/2014 | 39.1 | 1254 | 1254 | 53.6 | 44.2<br>53.3 | 1088 | 1163 | 471 | 474 |
| D2-100-R3 | 2/5/2014 | 44.2 | 1277 | 1330 | 40.9 | | 1281 | 1385 | 524 | 527 |
| | an | 45.1 | 1277 | 1323 | | 39.2 | 1066 | 1120 | 409 | 424 |
| | Dev | 6.4 | 23.5 | 65.8 | 45.3<br>7.2 | 45.6 | 1145 | 1223 | 468 | 475 |
| | CV | 14.2 | 1.8 | 5.0 | 15.9 | 7.1 | 118.3 | 142.2 | 57.6 | 51.5 |
| D2-50-R1 | 2/5/2014 | 56.3 | 1301 | | | 15.6 | 10.3 | 11.6 | 12.3 | 10.8 |
| D2-50-R1 | 2/5/2014 | 33.3 | 1193 | 1411 | 36.4 | 43.5 | 1130 | 1139 | <b>5</b> 75 | 575 |
| D2-50-R3 | 2/5/2014 | 33.3 | 1223 | 1230<br>1167 | 45.2 | 40.9 | 1208 | 1215 | 554 | 471 |
| Me | | 41.0 | The second secon | | 36.1 | 45.8 | 995 | 1170 | 517 | 416 |
| | Dev | 13.3 | 1239 | 1269 | 39.2 | 43.4 | 1111 | 1175 | 549 | 487 |
| | CV | 32.4 | 55.7<br>4.5 | 126.7 | 5.2 | 2.5 | 107.8 | 38:2 | 29.4 | 80.7 |
| 70 | ŲT. | 34.4 | 4.5 | 10.0 | 13.3 | 5.8 | 9.7 | 3.3 | 5.4 | 16.6 |



#### Appendix H: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1:<br>Linearity -<br>Continued | Acquisition Date | %STAT3 STIM | %/STAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>STIM [CD3+<br>Lymphs] | MESF tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3 STIM | %pSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|
| D2-2000-R1 | 2/5/2014 | 82.4 | 72.5 | 1679 | 1672 | 91.0 | 99.4 | 13130 | 13881 |
| D2-2000-R2 | 2/5/2014 | 80.4 | 72.8 | 1683 | 1678 | 89.9 | 99.1 | 12904 | 13713 |
| D2-2000-R3 | 2/5/2014 | 81.1 | 72.8 | 1685 | 1672 | 89.5 | 99.1 | 13103 | 13897 |
| | lean | 81.3 | 72.7 | 1682 | 1674 | 90.1 | 99.2 | 13046 | 13830 |
| | tDev | 1.0 | 0.2 | 3.1 | 3.5 | 0.8 | 0.2 | 123.4 | 101.9 |
| | %CV | 1.2 | 0.3 | 0.2 | 0.2 | 0.9 | 0.2 | 0.9 | 0.7 |
| D2-1000-R1 | 2/5/2014 | 77.3 | 66.4 | 1590 | 1547 | 87.7 | 98.6 | 12645 | 13643 |
| D2-1000-R2 | 2/5/2014 | 76.3 | 65.7 | 1574 | 1570 | 89.1 | 98.6 | 12588 | 13330 |
| D2-1000-R3 | 2/5/2014 | 76.2 | 66.5 | 1579 | 1568 | 91.8 | 98.7 | 12568 | 13242 |
| | lean . | 76.6 | 66.2 | 1581 | 1562 | 89.5 | 98.6 | 12600 | 13405 |
| | tDev | 0.6 | 0.4 | 8.2 | 12.7 | 2.1 | 0.1 | 40.0 | 210.8 |
| | %CV | 0.8 | 0.6 | 0.5 | 0.8 | 2.3 | 0.1 | 0.3 | 1.6 |
| D2-500-R1 | 2/5/2014 | 77.8 | 65.5 | 1565 | 1563 | 88.4 | 98.8 | 11960 | 12932 |
| D2-500-R2 | 2/5/2014 | 68.6 | 59.8 | 1472 | 1469 | 91.3 | 99.6 | 12079 | 12916 |
| D2-500-R3 | 2/5/2014 | 65.6 | 58.4 | 1442 | 1464 | 90.9 | 99.2 | 11617 | 12403 |
| | 1ean | 70.7 | 61.2 | 1493 | 1499 | 90.2 | 99.2 | 11885 | 12750 |
| | tDev | 6.4 | 3.8 | 64.1 | 55.8 | 1.6 | 0.4 | 239.9 | 300.9 |
| | %CV | 9.1 | 6.2 | 4.3 | 3.7 | 1.8 | 0.4 | 2.0 | 2,4 |
| D2-300-R1 | 2/5/2014 | 68.7 | 60,6 | 1477 | 1484 | 87.7 | 96.8 | 11419 | 11836 |
| D2-300-R2 | 2/5/2014 | 64.2 | 52.5 | 1363 | 1370 | 90.8 | 96.8 | 10949 | 11836 |
| D2-300-R3 | 2/5/2014 | 61.1 | 51.9 | 1377 | 1372 | 90.0 | 98.8 | 11401 | 12262 |
| | 1ean | 64.7 | 55.0 | 1406 | 1409 | 89.5 | 97.5 | 11256 | 11978 |
| | StDev | 3.8 | 4.9 | 62.2 | 65.2 | 1.6 | 1.2 | 266.3 | 246.0 |
| | %CV | 5.9 | 8.9 | 4.4 | 4.6 | 1.8 | 1.2 | 2.4 | 2.1 |
| D2-100-R1 | 2/5/2014 | 62.8 | 60.4 | 1394 | 1456 | 88.7 | 98.3 | 9847 | 10983 |
| D2-100-R2 | 2/5/2014 | 68.2 | 59.5 | 1370 | 1377 | 92.5 | 100.0 | 11985 | 12085 |
| D2-100-R3 | 2/5/2014 | 58.6 | 41.9 | 1310 | 1269 | 89.9 | 100.0 | 11689 | 12520 |
| | Mean | 63.2 | 53.9 | 1358 | 1367 | 90.4 | 99.4 | 11174 | 11863 |
| | StDev | 4.8 | 10.4 | 43.3 | 93.9 | 1.9 | 1.0 | 1158.4 | 792.3 |
| | %CV | 7.6 | 19.3 | 3.2 | 6.9 | 2.1 | 1.0 | 10.4 | 6.7 |
| D2-50-R1 | 2/5/2014 | 53.1 | 37.5 | 1277 | 1142 | 90.9 | 96.2 | 11641 | 11714 |
| D2-50-R2 | 2/5/2014 | 59.0 | 37.0 | 1334 | 1273 | 84.9 | 100.0 | 11689 | 12442 |
| D2-50-R3 | 2/5/2014 | 40.5 | 34.4 | 1142 | 1079 | 95.1 | 100.0 | 11086 | 10914 |
| to the second second | Mean | 50.9 | 36.3 | 1251 | 1165 | 90.3 | 98.7 | 11472 | 11690 |
| | StDev | 9.5 | 1.7 | 98.6 | 99.0 | 5.1 | 2.2 | 335.1 | 764.3 |
| | %CV | 18.7 | 4.7 | 7.9 | 8.5 | 5.6 | 2.2 | 2.9 | 6.5 |

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

# Appendix I: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1: Linearity<br>Continued | Acquisition Date | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim [CD3+ | MFI pSTAT3<br>unstim<br>[CD3+/CD4+ |
|---|---|---|---|---|---|---|---|
| D2-2000-R1 | 2/5/2014 | 172 | 170 | 736 | | Lymphs] | Lymphs] |
| D2-2000-R2 | 2/5/2014 | 177 | 175 | 701 | 734<br>700 | 497 | 563 |
| D2-2000-R3 | 2/5/2014 | 170 | 168 | 708 | 702 | 499 | 555 |
| | ean | 173 | 171 | 715 | 712 | 483 | 562 |
| | Dev | 3.6 | 3.6 | 18.5 | 19.1 | 493 | 560 |
| | CV | 2.1 | 2,1 | 2.6 | 2.7 | 8.7 | 4.4 |
| D2-1000-R1 | 2/5/2014 | 159 | 157 | 680 | 678 | 1.8 | 0.8 |
| D2-1000-R2 | 2/5/2014 | 176 | 177 | 674 | 672 | 457 | 521 |
| D2-1000-R3 | 2/5/2014 | 178 | 170 | 654 | 662 | 483 | 556 |
| | ean | 171 | 168 | 669 | 671 | 492 | 547 |
| | Dev | 10.4 | 10.1 | 13.6 | | 477 | 541 |
| | CV | 6.1 | 6.0 | 2.0 | 8.1 | 18.2 | 18.2 |
| D2-500-R1 | 2/5/2014 | 164 | 162 | 633 | | 3.8 | 3.4 |
| D2-500-R2 | 2/5/2014 | 164 | 158 | 566 | 638 | 480 | 536 |
| D2-500-R3 | 2/5/2014 | 196 | 188 | 560 | 569 | 519 | 578 |
| Me | an | 175 | 169 | 586 | 561 | 473 | 533 |
| StD | Dev | 18.5 | 16.3 | 40.5 | 589 | 491 | 549 |
| % | CV | 10.6 | 9.6 | 6.9 | 42.3 | 24.8 | 25.2 |
| D2-300-R1 | 2/5/2014 | 192 | 196 | 556 | 7.2 | 5.1 | 4.6 |
| D2-300-R2 | 2/5/2014 | 194 | 215 | 567 | 563 | 467 | 573 |
| D2-300-R3 | 2/5/2014 | 192 | 192 | 509 | 556 | 492 | 571 |
| Me | an | 193 | 201 | 544 | 530 | 528 | 573 |
| StD | Dev | 1.2 | 12.3 | 30.8 | 550 | 496 | 572 |
| <b>%</b> ( | CV | 0.6 | 6.1 | 5.7 | 17.4 | 30.7 | 1.2 |
| D2-100-R1 | 2/5/2014 | 231 | 267 | 521 | 3.2 | 6.2 | 0.2 |
| D2-100-R2 | 2/5/2014 | 175 | 166 | 503 | 554 | 438 | 467 |
| D2-100-R3 | 2/5/2014 | 197 | 197 | 512 | 503 | 514 | 554 |
| Me | an | 201 | 210 | 512 | 533 | 429 | 451 |
| StD | | 28.2 | 51.7 | 9.0 | 530 | 460 | 491 |
| %( | CV | 14.0 | 24.6 | 1.8 | 25.6 | 46.7 | 55.4 |
| D2-50-R1 | 2/5/2014 | 256 | 191 | 521 | 4.8 | 10.2 | 11.3 |
| D2-50-R2 | 2/5/2014 | 197 | 205 | 479 | 564 | 454 | 458 |
| D2-50-R3 | 2/5/2014 | 197 | 205 | 491 | 494 | 485 | 488 |
| Me | | 217 | 200 | | 469 | 401 | 470 |
| StD | ev | 34.1 | 8.1 | 497 | 509 | 447 | 472 |
| %0 | | 15.7 | 4.1 | 21.6 | 49.2 | 42.5 | 15.1 |
| | | | - T+ | 4.3 | 9.7 | 9.5 | 3.2 |





Appendix J: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1: Linearity<br>Continued | Acquisition Date | MFI FMO-PE STIM [CD3+ Lymphs] | MFI FMO-PE STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3 STIM<br>[CD3+ Lymphs] | MFI tSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3 STIM<br>[CD3+ Lymphs] | MFI pSTAT3 STIN<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|
| D2-2000-R1 | 2/5/2014 | 178 | 174 | 669 | 666 | 4987 | 5265 |
| D2-2000-R2 | 2/5/2014 | 185 | 185 | 670 | 668 | 4903 | 5203 |
| D2-2000-R3 | 2/5/2014 | 187 | 179 | 671 | 666 | 4977 | 5271 |
| | an | 183 | 179 | 670 | 667 | 4956 | 5246 |
| | Dev | 4.7 | 5.5 | 1.0 | 1.2 | 45.9 | 37.6 |
| | CV | 2.6 | 3.1 | 0.1 | 0.2 | 0.9 | 0.7 |
| D2-1000-R1 | 2/5/2014 | 186 | 184 | 634 | 617 | 4807 | 5177 |
| D2-1000-R2 | 2/5/2014 | 185 | 179 | 628 | 626 | 4786 | 5061 |
| D2-1000-R3 | 2/5/2014 | 182 | 180 | 630 | 625 | 4778 | 5028 |
| | ean | 184 | 181 | 631 | 623 | 4790 | 5089 |
| | Dev | 2.1 | 2.6 | 3.1 | 4.9 | 15.0 | 78.3 |
| | CV | 1.1 | 1.4 | 0.5 | 0.8 | 0.3 | 1.5 |
| D2-500-R1 | 2/5/2014 | 158 | 164 | 625 | 623 | 4552 | 4913 |
| D2-500-R2 | 2/5/2014 | 181 | 172 | 588 | 587 | 4596 | 4907 |
| D2-500-R3 | 2/5/2014 | 204 | 197 | 577 | 585 | 4425 | 4717 |
| | ean | 181 | 178 | 597 | 598 | 4524 | 4846 |
| | Dev | 23.0 | 17.2 | 25.1 | 21.4 | 88.8 | 111.5 |
| | cv | 12.7 | 9.7 | 4.2 | 3.6 | 2,0 | 2.3 |
| D2-300-R1 | 2/5/2014 | 209 | 209 | 590 | 593 | 4351 | 4506 |
| D2-300-R2 | 2/5/2014 | 202 | 197 | 545 | 548 | 4176 | 4506 |
| D2-300-R3 | 2/5/2014 | 185 | 180 | 551 | 549 | 4344 | 4664 |
| | ean | 199 | 195 | 562 | 563 | 4290 | 4559 |
| | Dev | 12.3 | 14.6 | 24.4 | 25.7 | 99.1 | 91.2 |
| | CV | 6.2 | 7.5 | 4.3 | 4.6 | 2.3 | 2.0 |
| D2-100-R1 | 2/5/2014 | 193 | 194 | 558 | 582 | 3765 | 4189 |
| D2-100-R1 | 2/5/2014 | 214 | 216 | 548 | 551 | 4561 | 4599 |
| D2-100-R3 | 2/5/2014 | 168 | 174 | 525 | 509 | 4452 | 4760 |
| | ean | 192 | 195 | 544 | 547 | 4259 | 4516 |
| | Dev | 23.0 | 21.0 | 16.9 | 36.6 | 431.6 | 294.4 |
| | CV | 12.0 | 10.8 | 3.1 | 6.7 | 10.1 | 6,5 |
| D2-50-R1 | 2/5/2014 | 235 | 235 | 512 | 459 | 4434 | 4461 |
| D2-50-R2 | 2/5/2014 | 226 | 193 | 534 | 510 | 4452 | 4731 |
| D2-50-R3 | 2/5/2014 | 212 | 171 | 459 | 434 | 4227 | 4163 |
| | ean 2/3/2011 | 224 | 200 | 502 | 468 | 4371 | 4452 |
| The second secon | Dev | 11.6 | 32.5 | 38.6 | 38.7 | 125.0 | 284.1 |
| | CV | 5.2 | 16.3 | 7.7 | 8.3 | 2.9 | 6.4 |



Appendix K: Table 1, Linearity - Healthy Donors 1-3 - Continued

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

| Table 1 Continued | Acquisition<br>Date | %Lymphs | Region<br>Events CD3+<br>Lymphs | %CD3+<br>[Lymphs] | Region Events<br>CD3+/CD4+<br>Lymphs | %CD3+/CD4<br>[Lymphs] | MESF FMO-PE<br>unstim [CD3+<br>Lymphs] | MESF FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %tSTAT3<br>unstim [CD3-<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|
| D3-2000-R1 | 2/11/2014 | 26.6 | 1365 | 71.0 | 901 | 66.0 | 396 | 389 | 88.8 |
| D3-2000-R2 | 2/11/2014 | 26.8 | 1371 | 70.6 | 950 | 69.3 | 414 | 413 | 88.7 |
| D3-2000-R3 | 2/11/2014 | 27.5 | 1380 | 71.2 | 949 | 68.8 | 418 | 414 | 88.0 |
| | lean | 27.0 | 1372 | 70.9 | 933 | 68.0 | 409 | 405 | 88.5 |
| | Dev | 0.5 | 7.5 | 0.3 | 28.0 | 1.8 | 11.7 | 14.2 | 0.4 |
| | 6CV | 1.9 | 0.5 | 0.4 | 3.0 | 2.6 | 2.9 | 3.5 | 0.5 |
| D3-1000-R1 | 2/11/2014 | 27.3 | 687 | 70.8 | 482 | 70.2 | 458 | 439 | 87.4 |
| D3-1000-R2 | 2/11/2014 | 28.0 | 689 | 70.7 | 463 | 67.2 | 427 | 432 | 84.9 |
| D3-1000-R3 | 2/11/2014 | 27.4 | 667 | 69.6 | 458 | 68.7 | 435 | 416 | 84.5 |
| M | lean | 27.6 | 681 | 70.4 | 468 | 68.7 | 440 | 429 | |
| | Dev | 0.4 | 12.2 | 0.7 | 12.7 | 1.5 | 16.1 | 11.8 | 85.6 |
| | 6CV | 1.4 | 1.8 | 1.0 | 2,7 | 2,2 | 3.7 | 2.8 | 1.6 |
| D3-500-R1 | 2/11/2014 | 29.8 | 341 | 70.2 | 230 | 67.5 | 433 | 402 | 1.9 |
| D3-500-R2 | 2/11/2014 | 28.7 | 336 | 69.9 | 226 | 67.3 | 428 | 436 | 85.7 |
| D3-500-R3 | 2/11/2014 | 28.5 | 333 | 68.4 | 222 | 66.7 | 452 | 469 | 82.1 |
| M | lean | 29.0 | 337 | 69.5 | 226 | 67.2 | 438 | | 81.0 |
| St | :Dev | 0.7 | 4.0 | 1.0 | 4.0 | 0.4 | 12.7 | 436 | 82.9 |
| 9/ | 6CV | 2.4 | 1.2 | 1.4 | 1.8 | 0.6 | 2.9 | 33.5 | 2.5 |
| D3-300-R1 | 2/11/2014 | 30.4 | 206 | 71.0 | 139 | 67.5 | 395 | 7.7 | 3.0 |
| D3-300-R2 | 2/11/2014 | 30.9 | 204 | 69.6 | 139 | 68.1 | 499 | 378 | 79.6 |
| D3-300-R3 | 2/11/2014 | 31.7 | 195 | 67.5 | 133 | 68.2 | 451 | 487 | 72.9 |
| М | ean | 31.0 | 202 | 69.4 | 137 | 67.9 | | 452 | 74.3 |
| St | Dev | 0.7 | 5.9 | 1.8 | 3.5 | 0.4 | 448<br>52.1 | 439 | 75.6 |
| 9/ | 6CV | 2.3 | 2.9 | 2.6 | 2.6 | 0.6 | | 55,7 | 3.5 |
| D3-100-R1 | 2/11/2014 | 35.7 | 71 | 71.7 | 53 | 74.7 | 11.6 | 12.7 | 4.6 |
| D3-100-R2 | 2/11/2014 | 26.9 | 62 | 63.9 | 39 | 62.9 | 484 | 490 | 76.1 |
| D3-100-R3 | 2/11/2014 | 29.1 | 69 | 72.6 | 47 | 68.1 | 449 | 436 | 73.9 |
| | ean | 30.6 | 67 | 69.4 | 46 | 68.6 | 477 | 481 | 71.8 |
| | Dev | 4.6 | 4.7 | 4.8 | 7.0 | 5.9 | 470 | 469 | 73.9 |
| | 6CV | 15.0 | 7.0 | 6.9 | 15.2 | 8.6 | 18.5 | 28.9 | 2.2 |
| D3-50-R1 | 2/11/2014 | 27.7 | 33 | 70.2 | 22 | | 3.9 | 6.2 | 3.0 |
| D3-50-R2 | 2/11/2014 | 21.0 | 32 | 71.1 | 18 | 66.7 | 508 | 388 | 63.0 |
| D3-50-R3 | 2/11/2014 | 28.4 | 36 | 72.0 | | 56.3 | 518 | 499 | 57.6 |
| | ean | 25.7 | 34 | 72.0 | 19 | 52.8 | 335 | 365 | 42.9 |
| | Dev | 4.1 | 2,1 | | 20 | 58.6 | 454 | 417 | 54.5 |
| | cv | 16.0 | 6.2 | 0.9 | 2.1 | 7.2 | 102.9 | 71.7 | 10.4 |
| | 207 | 10.0 | 0.2 | 1,3 | 10.5 | 12.3 | 22.7 | 17.2 | 19.1 |



Appendix L: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1<br>Continued | Acquisition<br>Date | %tSTAT3 unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>unstim [CD3+<br>Lymphs] | MESF tSTAT3 unstim [CD3+/CD4+ Lymphs] | %pSTAT3<br>unstim [CD3+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3 unstim [CD3+ Lymphs] | MESF pSTAT3 unstim [CD3+/CD4+ Lymphs] | MESF FMO-PE<br>STIM [CD3+<br>Lymphs] | MESF FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| D3-2000-R1 | 2/11/2014 | 93.6 | 2601 | 2660 | 48.8 | 65.8 | 1630 | 2002 | 385 | 391 |
| D3-2000-R2 | 2/11/2014 | 93.0 | 2508 | 2568 | 51.6 | 66.8 | 1720 | 2082 | 410 | 430 |
| D3-2000-R3 | 2/11/2014 | 92.5 | 2503 | 2521 | 50.1 | 65.4 | 1659 | 2023 | 383 | 374 |
| | ean | 93.0 | 2537 | 2583 | 50.2 | 66.0 | 1670 | 2036 | 393 | 398 |
| St | Dev | 0.6 | 55.2 | 70.7 | 1.4 | 0.7 | 45.9 | 41.5 | 15.0 | 28.7 |
| | CV | 0.6 | 2.2 | 2.7 | 2.8 | 1.1 | 2.7 | 2.0 | 3.8 | 7.2 |
| D3-1000-R1 | 2/11/2014 | 91.5 | 2561 | 2576 | 46.7 | 62.0 | 1533 | 1827 | 385 | 388 |
| D3-1000-R2 | 2/11/2014 | 90.5 | 2447 | 2470 | 49.3 | 62.9 | 1615 | 1904 | 420 | 411 |
| D3-1000-R3 | 2/11/2014 | 89.5 | 2384 | 2400 | 49.9 | 64.6 | 1658 | 2016 | 454 | 453 |
| | ean | 90.5 | 2464 | 2482 | 48.6 | 63.2 | 1602 | 1916 | 420 | 417 |
| | Dev | 1.0 | 89.7 | 88.6 | 1.7 | 1.3 | 63.5 | 95.0 | 34.5 | 33.0 |
| 9/ | CV | 1.1 | 3.6 | 3.6 | 3.5 | 2.1 | 4.0 | 5.0 | 8.2 | 7.9 |
| D3-500-R1 | 2/11/2014 | 89.8 | 2347 | 2351 | 46.1 | 63.5 | 1555 | 1937 | 429 | 426 |
| D3-500-R2 | 2/11/2014 | 85.9 | 2397 | 2385 | 50.6 | 64.5 | 1666 | 2010 | 473 | 457 |
| D3-500-R3 | 2/11/2014 | 84.6 | 2255 | 2255 | 46.7 | 59.4 | 1557 | 1887 | 419 | 409 |
| | ean | 86.8 | 2333 | 2330 | 47.8 | 62.5 | 1593 | 1945 | 440 | 431 |
| St | Dev | 2.7 | 72.0 | 67.4 | 2.4 | 2.7 | 63.5 | 61.9 | 28,7 | 24.3 |
| | CV . | 3.1 | 3.1 | 2.9 | 5.0 | 4.3 | 4.0 | 3.2 | 6.5 | 5.6 |
| D3-300-R1 | 2/11/2014 | 84.2 | 2230 | 2144 | 43.0 | 55.7 | 1437 | 1656 | 430 | 430 |
| D3-300-R2 | 2/11/2014 | 79,4 | 2197 | 2229 | 49.5 | 64.5 | 1656 | 1991 | 419 | 402 |
| D3-300-R3 | 2/11/2014 | 81.0 | 2177 | 2197 | 41.7 | 56.7 | 1452 | 1646 | 488 | 518 |
| | ean | 81.5 | 2201 | 2190 | 44.7 | 59.0 | 1515 | 1764 | 446 | 450 |
| | Dev | 2,4 | 26.8 | 42.9 | 4.2 | 4.8 | 122.3 | 196:4 | 37.1 | 60.5 |
| | bCV | 2.9 | 1.2 | 2.0 | 9.4 | 8.1 | 8.1 | 11.1 | 8.3 | 13.4 |
| D3-100-R1 | 2/11/2014 | 77.6 | 2111 | 2118 | 53.1 | 66.7 | 1861 | 1878 | 433 | 433 |
| D3-100-R2 | 2/11/2014 | 76.1 | 2047 | 2053 | 57.1 | 66.0 | 1755 | 1827 | 362 | 395 |
| D3-100-R3 | 2/11/2014 | 83,0 | 2031 | 2049 | 44.6 | 56.5 | 1464 | 1707 | 349 | 347 |
| | ean | 78.9 | 2063 | 2073 | 51.6 | 63.1 | 1693 | 1804 | 381 | 392 |
| | Dev | 3.6 | 42.3 | 38.7 | 6.4 | 5.7 | 205.6 | 87.8 | 45.2 | 43.1 |
| 9/ | 6CV | 4.6 | 2.1 | 1.9 | 12.4 | 9.0 | 12.1 | 4.9 | 11.9 | 11.0 |
| D3-50-R1 | 2/11/2014 | 68.4 | 1844 | 1850 | 41.9 | 65.0 | 1217 | 1907 | 376 | 376 |
| D3-50-R2 | 2/11/2014 | 66.7 | 1739 | 1821 | 43.3 | 73.7 | 1420 | 2066 | 388 | 452 |
| D3-50-R3 | 2/11/2014 | 81.8 | 1635 | 1844 | 44,8 | 61.9 | 1576 | 1697 | 510 | 589 |
| | ean | 72.3 | 1739 | 1838 | 43.3 | 66.9 | 1404 | 1890 | 425 | 472 |
| | Dev | 8.3 | 104.5 | 15.3 | 1.5 | 6.1 | 180.0 | 185;1 | 74.1 | 107.9 |
| 1) | 6CV | 11.5 | 6.0 | 0.8 | 3.5 | 9,1 | 12.8 | 9.8 | 17.4 | 22.9 |



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

Appendix M: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1<br>Continued | Acquisition<br>Date | %tSTAT3 STIM<br>[CD3+ Lymphs] | %tSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>STIM [CD3+<br>Lymphs] | MESF tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3 STIM | %pSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF pSTAT;<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|
| D3-2000-R1 | 2/11/2014 | 88.5 | 92.2 | 2591 | 2604 | 86.6 | 98.5 | 13232 | 15041 |
| D3-2000-R2 | 2/11/2014 | 88.0 | 91.5 | 2612 | 2606 | 88.9 | 98.6 | 13759 | 15182 |
| D3-2000-R3 | 2/11/2014 | 89.3 | 92.3 | 2522 | 2549 | 88.9 | 98.4 | 13719 | 14997 |
| | ean | 88.6 | 92.0 | 2575 | 2586 | 88.1 | 98.5 | 13570 | 15073 |
| | Dev | 0.7 | 0.4 | 47.1 | 32.3 | 1.3 | 0.1 | 293.4 | 96.6 |
| | 6CV | 0.8 | 0.4 | 1.8 | 1.2 | 1.5 | 0.1 | 2.2 | 0.6 |
| D3-1000-R1 | 2/11/2014 | 89.1 | 91,3 | 2527 | 2540 | 89.2 | 98.8 | 13894 | 15253 |
| D3-1000-R2 | 2/11/2014 | 87.9 | 92.9 | 2431 | 2432 | 88.2 | 98.7 | 12866 | 14655 |
| D3-1000-R3 | 2/11/2014 | 85.8 | 90.0 | 2368 | 2361 | 87.7 | 99.3 | 13371 | 14937 |
| | ean | 87.6 | 91.4 | 2442 | 2444 | 88.4 | 98.9 | 13377 | |
| | Dev | 1.7 | 1.5 | 80.1 | 90.1 | 0.8 | 0.3 | 514.0 | 14948<br>299.2 |
| % | CV . | 1.9 | 1.6 | 3.3 | 3.7 | 0.9 | 0.3 | 3.8 | 2.0 |
| D3-500-R1 | 2/11/2014 | 83.0 | 86.2 | 2448 | 2462 | 87.7 | 97.8 | 12512 | |
| D3-500-R2 | 2/11/2014 | 82.4 | 88.4 | 2334 | 2415 | 90.8 | 98.2 | 12682 | 14052 |
| D3-500-R3 | 2/11/2014 | 80.4 | 86.8 | 2240 | 2273 | 86.5 | 98.2 | 12939 | 13322 |
| M | ean | 81.9 | 87.1 | 2341 | 2383 | 88.3 | 98.1 | | 14476 |
| St | Dev | 1.4 | 1.1 | 104.2 | 98.4 | 2.2 | 0.2 | 12711 | 13950 |
| | CV . | 1.7 | 1.3 | 4.5 | 4.1 | 2.5 | 0.2 | 215.0 | 583.7 |
| D3-300-R1 | 2/11/2014 | 81.8 | 86.9 | 2252 | 2269 | 89.8 | 98.6 | 1.7 | 4.2 |
| D3-300-R2 | 2/11/2014 | 81.5 | 87.1 | 2204 | 2308 | 85.3 | 98.6 | 13095 | 14974 |
| D3-300-R3 | 2/11/2014 | 70.6 | 80.3 | 2167 | 2197 | 88.7 | 99.3 | 11780 | 12722 |
| M | ean | 78.0 | 84.8 | 2208 | 2258 | 87.9 | | 11889 | 12636 |
| St | Dev | 6.4 | 3.9 | 42.6 | 56.3 | 2.3 | 98.8 | 12255 | 13444 |
| | CV | 8.2 | 4.6 | 1.9 | 2.5 | 2.6 | 0.4 | 729.8 | 1325.7 |
| D3-100-R1 | 2/11/2014 | 75.0 | 87.0 | 2053 | 1979 | 90.1 | | 6.0 | 9.9 |
| D3-100-R2 | 2/11/2014 | 63,1 | 70.7 | 1991 | 2066 | 91.9 | 100.0 | 12148 | 13038 |
| D3-100-R3 | 2/11/2014 | 71.9 | 77.5 | 2047 | 2053 | 88.4 | 97.4 | 13322 | 13738 |
| | ean | 70.0 | 78.4 | 2030 | 2033 | | 97.9 | 12261 | 13119 |
| | Dev | 6.2 | 8.2 | 34.2 | 46.9 | 90.1 | 98.4 | 12577 | 13298 |
| | CV | 8.9 | 10.5 | 1.7 | 2.3 | 1.8 | 1.4 | 647.7 | 382.9 |
| D3-50-R1 | 2/11/2014 | 66.7 | 79.2 | 1750 | | 2.0 | 1.4 | 5.1 | 2.9 |
| D3-50-R2 | 2/11/2014 | 58.1 | 83.3 | 1805 | 1931 | 84.9 | 95.5 | 11009 | 11077 |
| D3-50-R3 | 2/11/2014 | 73.3 | 68.4 | 1907 | 2105 | 81.3 | 100.0 | 10039 | 12374 |
| | ean | 66.0 | | | 1967 | 83.3 | 100.0 | 6527 | 9886 |
| | Dev | 7.6 | 77.0 | 1821 | 2001 | 83.2 | 98.5 | 9192 | 11112 |
| | CV | 11.5 | 10.0 | 79.7 | 91.8 | 1.8 | 2.6 | 2358.1 | 1244.4 |
| 70 | | 11.3 | 10:0 | 4.4 | 4.6 | 2.2 | 2.6 | 25.7 | 11.2 |

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

Annendix N: Table I. Linearity - Healthy Donors 1-3 - Continued

| Table 1<br>Continued | Acquisition<br>Date | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3 unstim [CD3+ | MFI pSTAT:<br>unstim<br>[CD3+/CD4-<br>Lymphs] |
|---|---|---|---|---|---|---|---|
| D3-2000-R1 | 2/11/2014 | 150 | 147 | 967 | 989 | 609 | 746 |
| D3-2000-R2 | 2/11/2014 | 157 | 156 | 933 | 955 | 642 | <i>7</i> 76 |
| D3-2000-R3 | 2/11/2014 | 158 | 157 | 931 | 938 | 620 | 754 |
| THE RESERVE OF THE PARTY OF THE | ean | 155 | 153 | 944 | 961 | 624 | 759 |
| | Dev | 4.4 | 5.5 | 20.2 | 26.0 | 16.8 | 15.5 |
| | CV | 2.8 | 3.6 | 2.1 | 2.7 | 2.7 | 2.0 |
| D3-1000-R1 | 2/11/2014 | 173 | 166 | 953 | 958 | 573 | 682 |
| D3-1000-R2 | 2/11/2014 | 162 | 163 | 911 | 919 | 604 | 710 |
| D3-1000-R3 | 2/11/2014 | 165 | 158 | 887 | 893 | 619 | 752 |
| | ean | 167 | 162 | 917 | 923 | 599 | 715 |
| | Dev | 5.7 | 4.0 | 33.4 | 32,7 | 23.5 | 35,2 |
| | CV | 3.4 | 2.5 | 3.6 | 3.5 | 3.9 | 4.9 |
| D3-500-R1 | 2/11/2014 | 164 | 152 | 874 | 875 | 581 | 722 |
| D3-500-R2 | 2/11/2014 | 162 | 165 | 892 | 888 | 622 | 749 |
| D3-500-R3 | 2/11/2014 | 171 | 177 | 840 | 840 | 582 | 704 |
| | ean | 166 | 165 | 869 | 868 | 595 | 725 |
| | Dev | 4.7 | 12.5 | 26.4 | 24.8 | 23,4 | 22.6 |
| | CV | 2.8 | 7.6 | 3.0 | 2.9 | 3.9 | 3.1 |
| D3-300-R1 | 2/11/2014 | 150 | 143 | 831 | 799 | 538 | 618 |
| D3-300-R2 | 2/11/2014 | 189 | 184 | 818 | 830 | 618 | 742 |
| D3-300-R3 | 2/11/2014 | 170 | 171 | 811 | 818 | 543 | 615 |
| | ean | 170 | 166 | 820 | 816 | 566 | 658 |
| | Dev | 19.5 | 21.0 | 10.1 | 15.6 | 44.8 | 72.5 |
| | CV | 11.5 | 12.7 | 1.2 | 1.9 | 7.9 | 11.0 |
| D3-100-R1 | 2/11/2014 | 183 | 185 | 787 | 789 | 694 | 701 |
| D3-100-R2 | 2/11/2014 | 170 | 165 | 763 | 765 | 655 | 682 |
| D3-100-R3 | 2/11/2014 | 180 | 182 | 757 | 764 | 547 | 638 |
| | ean | 178 | 177 | 769 | 773 | 632 | 674 |
| St | Dev | 6.8 | 10.8 | 15.9 | 14.2 | 76.2 | 32.3 |
| % | CV | 3.8 | 6.1 | 2.1 | 1.8 | 12.1 | 4.8 |
| D3-50-R1 | 2/11/2014 | 192 | 147 | 688 | 690 | 456 | 711 |
| D3-50-R2 | 2/11/2014 | 196 | 189 | 649 | 680 | 531 | 770 |
| D3-50-R3 | 2/11/2014 | 127 | 138 | 611 | 688 | 589 | 634 |
| | ean | 172 | 158 | 649 | 686 | 525 | 705 |
| St | Dev | 38.7 | 27.2 | 38.5 | 5,3 | 66.7 | 68.2 |
| 0/4 | cV | 22,5 | 17.2 | 5.9 | 0.8 | 12.7 | 9.7 |





Appendix O: Table 1, Linearity - Healthy Donors 1-3 - Continued

| Table 1<br>Continued | Acquisition<br>Date | MFI FMO-PE<br>STIM [CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>STIM [CD3+<br>Lymphs] | MFI tSTAT3 STIM [CD3+/CD4+ Lymphs] | MFI pSTAT3<br>STIM [CD3+<br>Lymphs] | MFI pSTATS<br>STIM<br>[CD3+/CD4+ |
|---|---|---|---|---|---|---|---|
| D3-2000-R1 | 2/11/2014 | 146 | 148 | 964 | 968 | 4845 | Lymphs] |
| D3-2000-R2 | 2/11/2014 | 155 | 163 | 971 | 969 | 5036 | 5500 |
| D3-2000-R3 | 2/11/2014 | 145 | 142 | 938 | 948 | 5021 | 5552<br>5484 |
| | ean | 149 | 151 | 958 | 962 | 4967 | |
| | Dev | 5.5 | 10.8 | 17.4 | 11.8 | 106.2 | 5512 |
| | CV | 3.7 | 7.2 | 1.8 | 1.2 | 2.1 | 35.6 |
| D3-1000-R1 | 2/11/2014 | 146 | 147 | 940 | 945 | 5085 | 0.6 |
| D3-1000-R2 | 2/11/2014 | 159 | 156 | 905 | 905 | 4712 | 5577 |
| D3-1000-R3 | 2/11/2014 | 172 | 171 | 881 | 879 | | 5361 |
| | an | 159 | 158 | 909 | 910 | 4895 | 5463 |
| | Dev | 13.0 | 12.1 | 29.7 | 33.2 | 4897 | 5467 |
| | CV | 8.2 | 7,7 | 3.3 | 3.6 | 186.5 | 108.1 |
| D3-500-R1 | 2/11/2014 | 162 | 161 | 911 | 916 | 3.8 | 2.0 |
| D3-500-R2 | 2/11/2014 | 179 | 173 | 869 | 899 | 4584 | 5142 |
| D3-500-R3 | 2/11/2014 | 159 | 155 | 834 | 846 | 4646 | 4878 |
| Me | an | 167 | 163 | 871 | 887 | 4738 | 5296 |
| StD | Dev | 10.8 | 9.2 | 38,6 | 36.5 | 4656 | 5105 |
| % | CV | 6.5 | 5.6 | 4.4 | 4.1 | 77.5 | 211.4 |
| D3-300-R1 | 2/11/2014 | 163 | 163 | 839 | | 1.7 | 4.1 |
| D3-300-R2 | 2/11/2014 | 158 | 152 | 821 | 845<br>859 | 4795 | 5476 |
| D3-300-R3 | 2/11/2014 | 184 | 196 | 807 | 818 | 4318 | 4660 |
| M∈ | an | 168 | 170 | 822 | 841 | 4358 | 4629 |
| Sto | )ev | 13.8 | 22.9 | 16.0 | | 4490 | 4922 |
| % | CV | 8,2 | 13.5 | 1.9 | 20.8 | 264.6 | 480.3 |
| D3-100-R1 | 2/11/2014 | 164 | 164 | 765 | 2.5 | 5.9 | 9,8 |
| D3-100-R2 | 2/11/2014 | 137 | 150 | 742 | 738<br>770 | 4452 | 4775 |
| D3-100-R3 | 2/11/2014 | 132 | 132 | 763 | THE SECOND PROPERTY OF | 4878 | 5028 |
| Me | an | 144 | 149 | 757 | 765 | 4492 | 4804 |
| StD | ev | 17.2 | 16.0 | 12.7 | 758<br>17.2 | 4607 | 4869 |
| % | CV | 11.9 | 10.7 | 1.7 | | 235.3 | 138.5 |
| D3-50-R1 | 2/11/2014 | 142 | 142 | 653 | 2.3 | 5.1 | 2.8 |
| D3-50-R2 | 2/11/2014 | 147 | 171 | 673 | 720 | 4038 | 4063 |
| D3-50-R3 | 2/11/2014 | 193 | 222 | 711 | 784 | 3686 | 4534 |
| Me | | 161 | 178 | 679 | 733 | 2406 | 3630 |
| StD | | 28.1 | 40.5 | | 746 | 3377 | 4076 |
| | CV | 17.5 | 22.8 | 29.5<br>4.3 | 33.8<br>4.5 | 858.8<br>25.4 | 452.1<br>11.1 |



#### Appendix P: Table 2, Linearity - Relative Error Calculations - Donor 1

| Table 2: Donor 1 Linearity (%RE cutoff is ≥25%) | %tSTAT3<br>unstim [CD3+<br>Lymphs] | %tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>unstirn [CD3+<br>Lymphs] | | %pSTAT3<br>unstim [CD3+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF<br>pSTAT3<br>unstim [CD3+<br>Lymphs] | MESF<br>pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 38.7 | 50.5 | 1633 | 1634 | 2.4 | 5.9 | 735 | 794 |
| %Relative Error- 1000 spike | 8.5 | 12.9 | 3.4 | 4.5 | 12.5 | 11.9 | 2.2 | 3.0 |
| %Relative Error- 500 spike | 23.0 | 22.2 | 8.0 | 9.8 | 4.2 | 6.8 | 0.3 | 2.4 |
| %Relative Error- 300 spike | 35.1 | 24.6 | 10.6 | 10.2 | 33.3 | 15.3 | 2.2 | 0.4 |
| %Relative Error- 100 spike | 51.7 | 42.4 | 15.0 | 14.9 | 37.5 | 16.9 | 3.5 | 0.4 |
| - %Relative Error- 50 spike | 51.9 | 27.7 | 17.5 | 10.5 | 16.7 | 8.5 | 3.8 | 3.4 |

| Table 2: Donor 1 Linearity (%RE cutoff is ≥25%) - Continued | %tSTAT3 STIM [CD3+ Lymphs] | %tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF ISTATS | MESF tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3<br>STIM [CD3+<br>Lymphs] | %pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF<br>pSTAT3 STIM<br>[CD3+<br>Lymphs] | MESF pSTAT3 STIM [CD3+/CD4+ Lymphs] | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 36.6 | 46.6 | 1606 | 1583 | 54.2 | 93.4 | 2822 | 10649 | 217 | 209 |
| %Relative Error- 1000 spike | 12.6 | 11,6 | 4.2 | 3.8 | 0.7 | 1.5 | 1.2 | 2.7 | 1.4 | 3.3 |
| %Relative Error- 500 spike | 26.0 | 30.7 | 7.5 | 10.7 | 2.0 | 1.1 | 5.2 | 6.1 | 5,5 | 8.1 |
| %Relative Error- 300 spike | 29.8 | 29.8 | 9.7 | 9.5 | 0.2 | 0.4 | 0.2 | 7.4 | 3.2 | 14.8 |
| %Relative Error- 100 spike | 32,8 | 33.5 | 13.8 | 11.7 | 11.1 | 1.4 | 4.7 | 17.2 | 6.9 | 10.0 |
| %Relative Error- 50 spike | 59.6 | 33.7 | 19.6 | 17.4 | 10.3 | 2.2 | 54.8 | 13.1 | 4.1 | 19.6 |

| Table 2: Donor 1 Linearity (%RE cutoff is ≥25%) - Continued | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim [CD3+<br>Lymphs] | | MFI FMO-PE<br>STIM [CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI (STAT3 | MFI tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>STIM [CD3+<br>Lymphs] | MFI pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 651 | 651 | 299 | 322 | 215 | 214 | 641 | 631 | 1111 | 4064 |
| %Relative Error- 1000 spike | 3.4 | 4.3 | 2.0 | 2.8 | 3.7 | 1.4 | 4.2 | 3.6 | 1.2 | 2.6 |
| %Relative Error- 500 spike | 7.8 | 9.5 | 0.3 | 2.2 | 7.4 | 8.4 | 7.3 | 10.3 | 4.8 | 6.0 |
| %Relative Error- 300 spike | 10.4 | 10.0 | 2.0 | 0.3 | 8.8 | 6.5 | 9.5 | 9.2 | 0.3 | 7.3 |
| %Relative Error- 100 spike | 14.7 | 14,4 | 3.7 | 0.3 | 0.5 | 14.0 | 13.6 | 11.4 | 5.0 | 16.8 |
| %Relative Error- 50 spike | 17.1 | 10.3 | 3.3 | 3.4 | 23.3 | 4.7 | 19.2 | 17.1 | 51.9 | 32.1 |



## Appendix Q: Table 3, Linearity - Relative Error Calculations - Donor 2

| Table 3: Donor 2 Linearity (%RE cutoff<br>is ≥25%) | %tSTAT3<br>unstim [CD3+<br>Lymphs] | %tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3 unstim [CD3+ Lymphs] | MESF tSTAT3 unstim [CD3+/CD4+ Lymphs] | %pSTAT3 unstim [CD3+ Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3 unstim [CD3+ Lymphs] | MESF pSTAT3 unstim [CD3+/CD4+ Lymphs] |
|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 86.2 | 80.6 | 1797 | 1790 | 49.8 | 51.7 | 1228 | |
| %Relative Error- 1000 spike | 3.6 | 4.2 | 6.5 | 5.9 | 4.6 | | | 1399 |
| %Relative Error- 500 spike | 19.8 | 27.0 | 18,4 | | | 3.3 | 3.2 | 3.3 |
| %Relative Error- 300 spike | | | | 17.6 | 1,4 | 2.5 | 0.4 | 1.9 |
| | 29.8 | 37.7 | 24.4 | 23.3 | 0.8 | 1.9 | 0.6 | 2,3 |
| %Relative Error- 100 spike | 39.1 | 44.0 | 28.9 | 26.1 | 9.0 | 11.8 | | |
| %Relative Error- 50 spike | 42.2 | 49.1 | 31.1 | | | | 6.8 | 12.6 |
| The same of the same | 1 Km 2 Sw | 17.1 | J.i. I | 29.1 | 21.3 | 16.1 | 9.5 | 16.0 |

| Table 3: Donor 2 Linearity (%RE cutoff is ≥25%) - Continued | Lymphs | %tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>STIM [CD3+<br>Lymphs] | MESF tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3<br>STIM [CD3+<br>Lymphs] | %pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF<br>pSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | [CD3+/CD4+ |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 81.3 | 72.7 | 1682 | 1674 | 90.1 | 99.2 | 13046 | | chubusi | Lymphs] |
| %Relative Error- 1000 spike | 5.8 | 8,9 | 6.0 | 5.7 | 0.7 | 0,6 | | 13830 | 173 | 171 |
| %Relative Error- 500 spike | 13.0 | 15.8 | 11.2 | 10.5 | | | 3.4 | 3.1 | 1.2 | 1.8 |
| %Relative Error- 300 spike | | | | | 0.1 | 0.0 | 8.9 | 7.8 | 1.2 | 1.2 |
| | 20.4 | 24.3 | 16,4 | 15.8 | 0.7 | 1.7 | 13.7 | 13.4 | 11.6 | 17.5 |
| %Relative Error- 100 spike | 22.3 | 25.9 | 19.3 | 18.3 | 0.3 | 0.2 | 14.3 | 14.2 | | |
| %Relative Error- 50 spike | 37.4 | 50.1 | 25.6 | 30.4 | 0.2 | 0.5 | | | 16.2 | 22.8 |
| | | - 316 | | 10 Str 1 | 0.2 | 0.5 | 12.1 | 15.5 | 25.4 | 17.0 |

| "able 3: Donor 2 Linearity (%RE cutoff is ≥25%) - Continued | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim [CD3+<br>Lymphs] | MFI pSTAT3 unstim [CD3+/CD4+ Lymphs] | MFI FMO-PE<br>STIM [CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>STIM [CD3+<br>Lymphs] | MFI tSTAT3 STIM [CD3+/CD4+ Lymphs] | MFI pSTAT3<br>STIM [CD3+<br>Lymphs] | MFI pSTAT3<br>STIM<br>(CD3+/CD4+ |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 715 | 712 | 493 | 560 | 183 | 179 | 670 | | | Lymphs] |
| %Relative Error- 1000 spike | 6.4 | 5.8 | 3,2 | 3.4 | 0,5 | | | 667 | 4959 | 5246 |
| %Relative Error- 500 spike | 18.0 | 17.3 | 0,4 | | | 1.1 | 5.8 | 6.6 | 3.3 | 3.0 |
| %Relative Error- 300 spike | | | | 2.0 | 1.1 | 0.6 | 10.9 | 10.3 | 8.7 | 7.6 |
| | 23.9 | 22.8 | 0.6 | 2.1 | 8.7 | 8.9 | 16.1 | 15.6 | 13.4 | 13.1 |
| %Relative Error- 100 spike | 28.4 | 25.6 | 6.7 | 12.3 | 4.9 | 8.9 | 18.8 | | | |
| %Relative Error- 50 spike | 30.5 | 28.5 | 9.3 | 15.7 | 22.4 | | | 18.0 | 14.1 | 13.9 |
| | | | 7.5 | 13.7 | 22.4 | 11.7 | 25.1 | 29.8 | 11.8 | 15.1 |



#### Appendix R: Table 4, Linearity - Relative Error Calculations - Donor 3

| Table 4: Donor 3 Linearity (%RE cutoff is ≥25%) | %tSTAT3<br>unstim<br>[CD3+<br>Lymphs] | %tSTAT3 unstim<br>[CD3+/CD4+<br>Lymphs] | MESF tSTAT3<br>unstim [CD3+<br>Lymphs] | MESF tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %p\$TAT3<br>unstim [CD3+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3<br>unstim [CD3+<br>Lymphs] | MESF pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 88.5 | 93.0 | 2537 | 2583 | 50.2 | 66.0 | 1670 | 2036 |
| %Relative Error- 1000 spike | 3.3 | 2.7 | 2.9 | 3.9 | 3.2 | 4.2 | 4.1 | 5.9 |
| %Relative Error- 500 spike | 6.3 | 6.7 | 8.0 | 9.8 | 4.8 | 5.3 | 4.6 | 4.5 |
| %Relative Error- 300 spike | 14.6 | 12.4 | 13.2 | 15.2 | 11.0 | 10.6 | 9.3 | 13.4 |
| %Relative Error- 100 spike | 16.5 | 15.2 | 18.7 | 19.7 | 2.8 | 4.4 | 1.4 | 11.4 |
| %Relative Error- 50 spike | 38.4 | 22.3 | 31.5 | 28.8 | 13.7 | 1.4 | 15.9 | 7.2 |

| Table 4: Donor 3 Linearity (%RE cutoff is \$25%) - Continued | %tSTAT3<br>STIM [CD3+<br>Lymphs] | | | MESF<br>tSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | | %pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF<br>pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-PE<br>unstim [CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 88.6 | 92.0 | 2575 | 2586 | 88.1 | 98.5 | 13570 | 15073 | 156 | 153 |
| %Relative Error- 1000 spike | 1.1 | 0.7 | 5.2 | 5.5 | 0.3 | 0.4 | 1.4 | 0.8 | 7.7 | 5.9 |
| %Relative Error- 500 spike | 7.6 | 5.3 | 9.1 | 7.8 | 0.2 | 0.4 | 6.3 | 7.5 | 7.1 | 7.8 |
| %Relative Error- 300 spike | 12.0 | 7.8 | 14.3 | 12.7 | 0.2 | 0.3 | 9.7 | 10.8 | 9.7 | 8.5 |
| %Relative Error- 100 spike | 21.0 | 14.8 | 21.2 | 21,4 | 2.3 | 0.1 | 7.3 | 11.8 | 14.8 | 15.7 |
| %Relative Error- 50 spike | 25.5 | 16.3 | 29.3 | 22.6 | 5.6 | 0.0 | 32.3 | 26.3 | 11.0 | 3.3 |

| Fable 4: Donor 3 Linearity (%RE cutoff is<br>>25%) - Continued | MFI tSTAT3<br>unstim [CD3+<br>Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim [CD3+<br>Lymphs] | MFI pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-PE<br>STIM [CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4÷<br>Lymphs] | MFI tSTAT3<br>STIM<br>[CD3+<br>Lymphs] | MFI tSTAT3<br>STIM<br>[CD3+/CD4+<br>[Lymphs] | MFI pSTAT3<br>STIM [CD3+<br>Lymphs] | MFI pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| Accepted Value (AVG @2000 spike) | 944 | 961 | 624 | 759 | 149 | 151 | 958 | 962 | 4967 | 5512 |
| %Relative Error- 1000 spike | 2.9 | 4.0 | 4.0 | 5.8 | 6.7 | 4.6 | 5.1 | 5.4 | 1.4 | 0.8 |
| %Relative Error- 500 spike | 7.9 | 9.7 | 4.6 | 4.5 | 12.1 | 7.9 | 9.1 | 7.8 | 6.3 | 7.4 |
| - %Relative Error- 300 spike | 13.1 | 15.1 | 9.3 | 13.3 | 12.8 | 12.6 | 14.2 | 12.6 | 9.6 | 10.7 |
| %Relative Error- 100 spike | 18.5 | 19.5 | 1.3 | 11.2 | 3.4 | 1.3 | 21.0 | 21.2 | 7.2 | 11.7 |
| %Relative Error- 50 spike | 31.3 | 28,6 | 15.9 | 7.1 | 8.1 | 17.9 | 29.1 | 22.5 | 32.0 | 26.1 |



Appendix S: Table 5, Inter/Intra-Assay Precision

| , Table 5 -<br>inter/Intra-<br>Assay | Acquisition<br>Date | %Lymphs | Region Events<br>CD3+Lymphs | %CD3+<br>[Lymphs] | Region<br>Events<br>CD3+/CD4+<br>Lymphs | %CD3+/CD4<br>[Lymphs] | MESF FMO-<br>PE unstim<br>[CD3+<br>Lymphs] | MESF FMO-<br>PE unstim<br>[CD3+/CD4+<br>Lymphs] | %tSTAT3 unstim [CD3+ Lymphs] | %tSTAT3<br>unstim<br>[CD3+/CD4<br>+ Lymphs] | MESF<br>tSTAT3<br>unstim<br>[CD3+ | MESF<br>tSTAT3<br>unstim<br>[CD3+/CD4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| D1-01-R1 | 2/18/2014 | 21.1 | 1342 | 68.9 | 1002 | 74.7 | 629 | 643 | 73.7 | 78.7 | Lymphs] | Lymphs] |
| D1-01-R2 | 2/18/2014 | 20.9 | 1296 | 66.6 | 903 | 69.7 | 698 | 695 | 70.6 | 77.9 | 3849 | 3870 |
| D1-O1-R3 | 2/18/2014 | 21.0 | 1305 | 67.8 | 926 | 71.0 | 700 | 708 | 69.2 | 78.1 | 3786 | 3785 |
| Mean | -D1-Op1 | 21.0 | 1314 | 67.8 | 944 | 71.8 | 676 | 682 | | | 3711 | 3763 |
| StDev | /-D1-Op1 | 0.1 | 24.4 | 1.2 | 51.8 | 2.6 | 40.4 | 34,4 | 71.2 | 78.2 | 3782 | 3806 |
| %CV | -D1-Op1 | 0.5 | 1.9 | 1.8 | 5.5 | 3.6 | 6.0 | 5.0 | 3.2 | 0.4 | 69.1 | 56.5 |
| D1-02-R1 | 2/18/2014 | 17.7 | 1384 | 71.1 | 1011 | 73.1 | 831 | 820 | | 0.5 | 1.8 | 1.5 |
| D1-O2-R2 | 2/18/2014 | 17.7 | 1410 | 71.6 | 1003 | 71.1 | 850 | 861 | 64.7 | 74.4 | 3513 | 3567 |
| D1-O2-R3 | 2/18/2014 | 18.6 | 1367 | 70.2 | 960 | 70.2 | 858 | 868 | 64.7 | 74.0 | 3561 | 3585 |
| Mean | -D1-Op2 | 18.0 | 1387 | 71.0 | 991 | 71.5 | 846 | | 59.6 | 69.4 | 3410 | 3444 |
| StDev | -D1-Op2 | 0.5 | 21.7 | 0.7 | 27.4 | 1.5 | 13.9 | 850 | 63.0 · | 72.6 | 3495 | 3532 |
| | -D1-Op2 | 2.8 | 1.6 | 1.0 | 2.8 | 2.1 | | 25.9 | 2.9 | 2.8 | 77.2 | 76.7 |
| | A SECTION | West remains | TO SECURITION OF THE PARTY OF T | NOW SHAPE | | Z.I | 1.6 | 3.0 | 4.6 | 3.9 | 2.2 | 2.2 |
| Mean-Inte | r-Op-Donor1 | 19.5 | 1351 | 69.4 | 968 | 71.7 | 761 | 766 | San Line | | | ETF SWOT |
| | er-Op-Donor1 | 2.1 | 51.6 | 2.3 | 33.2 | 0.2 | 120.2 | 766 | 67.1 | 75.4 | 3639 | 3669 |
| %CV-Inte | r-Op-Donor1 | 10.8 | 3.8 | 3.3 | 3.4 | 0.3 | 15.8 | 118.8 | 5.8 | 4.0 | 202.9 | 193.7 |
| D2-O1-R1 | 2/18/2014 | 32.6 | 1494 | 71.9 | 804 | 53.8 | 765 | 15.5 | 8.6 | 5.3 | 5.6 | 5.3 |
| D2-O1-R2 | 2/18/2014 | 34.0 | 1510 | 72.7 | 785 | 52.0 | 760 | 714 | 54.9 | 66.2 | 3221 | 3248 |
| D2-O1-R3 | 2/18/2014 | 32.7 | 1495 | 72.6 | 764 | 51.1 | 738 | 736 | 55.9 | 66.2 | 3228 | 3218 |
| Mean | -D2-Op1 | 33.1 | 1500 | 72.4 | 784 | | | 741 | 51.4 | 61.6 | 3142 | 3187 |
| | -D2-Op1 | 0.8 | 9.0 | 0.4 | 20.0 | 52.3 | 754 | 730 | 54.1 | 64.7 | 3197 | 3218 |
| | -D2-Op1 | 2.4 | 0.6 | 0.6 | 2.6 | 2.7 | 14.4 | 14.4 | 2.4 | 2.7 | 47.8 | 30.5 |
| D2-O2-R1 | 2/18/2014 | 31.9 | 1449 | 70.3 | 767 | | 1.9 | 2.0 | 4.4 | 4.2 | 1.5 | 0.9 |
| D2-O2-R2 | 2/18/2014 | 33.6 | 1475 | 72.1 | 788 | 52.9 | 758 | 723 | 45.1 | 53.1 | 2914 | 2889 |
| D2-O2-R3 | 2/18/2014 | 32.8 | 1482 | 72.1 | 821 | 53.4 | 781 | 751 | 45.9 | 59.5 | 2990 | 3023 |
| Mean | -D2-Op2 | 32.8 | 1469 | 71.5 | | 55.4 | 787 | 767 | 48.5 | 60.2 | 3041 | 3032 |
| | -D2-Op2 | 0.9 | 17.4 | | 792 | 53.9 | 775 | 747 | 46.5 | 57.6 | 2982 | 2981 |
| | D2-Op2 | 2,7 | 1,2 | 1.0 | 27.2 | 1.3 | 15.3 | 22.3 | 1.8 | 3.9 | 63.9 | 80.1 |
| | | Est / | L.C | 1.4 | 3.4 | 2.4 | 2.0 | 3.0 | 3.9 | 6.8 | 2.1 | 2.7 |
| Mean-Inte | r-Op-Donor2 | 33.0 | 1485 | 72.0 | 700 | 50.4 | | NATIONAL PROPERTY. | | | | |
| | er-Op-Donor2 | 0.2 | 21.9 | 0.6 | 788 | 53.1 | 765 | 739 | 50.3 | 61.2 | 3090 | 3100 |
| | r-Op-Donor2 | 0.6 | 1.5 | 0.8 | 5.7 | 1.1 | 14.8 | 12.0 | 5.4 | 5.0 | 152.0 | 167.6 |
| | -P-aniois | 0.0 | 1.3 | 0.8 | 0.7 | 2.1 | 1.9 | 1.6 | 10.7 | 8.2 | 4.9 | 5.4 |



#### Appendix T: Table 5, Inter/Intra-Assay Precision - Continued

| Table 5 -<br>inter/Intra-<br>Assay | Acquisition<br>Date | %pSTAT3 unstim [CD3+ Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4<br>+ Lymphs] | MESF pSTAT3 unstim [CD3+ Lymphs] | MESF pSTAT3 unstim [CD3+/CD4+ Lymphs] | MESF FMO-<br>PESTIM<br>[CD3+<br>Lymphs] | MESF FM O-<br>PESTIM<br>[CD3+/CD4<br>+ Lymphs] |
|---|---|---|---|---|---|---|---|
| D1-O1-R1 | 2/18/2014 | 35.2 | 47.9 | 2253 | 2706 | 687 | 677 |
| D1-O1-R2 | 2/18/2014 | 37.1 | 50.3 | 2361 | 2843 | 711 | 696 |
| D1-01-R3 | 2/18/2014 | 37.0 | 49.7 | 2431 | 2796 | 743 | 701 |
| Mean-l | D1-Op1 | 36.4 | 49.3 | 2348 | 2782 | 714 | 691 |
| | D1-Op1 | 1.1 | 1.2 | 89.7 | 69.6 | 28.1 | 12.7 |
| %CV-I | 01-Op1 | 3.0 | 2.4 | 3.8 | 2.5 | 3.9 | 1.8 |
| D1-02-R1 | 2/18/2014 | 40.9 | 53.4 | 2594 | 3029 | 638 | 642 |
| D1-02-R2 | 2/18/2014 | 39.3 | 52.0 | 2485 | 2938 | 679 | 683 |
| D1-O2-R3 | 2/18/2014 | 40.3 | 52.8 | 2530 | 2975 | 658 | 639 |
| Mean- | D1-Op2 | 40.2 | 52.7 | 2536 | 2981 | 658 | 655 |
| The second secon | D1-Op2 | 0,8 | 0.7 | 54.8 | 45.8 | 20.5 | 24.6 |
| | D1-Op2 | 2.0 | 1.3 | 2.2 | 1.5 | 3.1 | 3.8 |
| DULLA . A | | THE PERSON | THE REPORT OF | A DESCRIPTION | TON STREET | | |
| Mean-Inter | -Op-Donor1 | 38.3 | 51.0 | 2442 | 2882 | 686 | 673 |
| | -Op-Donor1 | 2.7 | 2.4 | 132.9 | 140.7 | 39.6 | 25.5 |
| %CV-Inter | -Op-Donori | 7.0 | 4.7 | 5.4 | 4.9 | 5.8 | 3.8 |
| D2-O1-R1 | 2/18/2014 | 3.2 | 8.0 | 1176 | 1244 | 790 | 740 |
| D2-O1-R2 | 2/18/2014 | 3.0 | 8.1 | 1217 | 1318 | 780 | 775 |
| D2-O1-R3 | 2/18/2014 | 2.8 | 6.2 | 1193 | 1280 | 813 | 825 |
| Mean- | D2-Op1 | 3.0 | 7.4 | 1195 | 1281 | 794 | 780 |
| | D2-Op1 | 0.2 | 1.1 | 20.6 | 37.0 | 16.9 | 42.7 |
| %CV- | D2-Op1 | 6.7 | 14.9 | 1.7 | 2.9 | 2.1 | 5.5 |
| D2-O2-R1 | 2/18/2014 | 6.3 | 14.5 | 1279 | 1405 | 762 | 741 |
| D2-O2-R2 | 2/18/2014 | 6.3 | 12.9 | 1242 | 1411 | 746 | 723 |
| D2-O2-R3 | 2/18/2014 | 6.4 | 15.1 | 1308 | 1508 | 779 | 765 |
| | D2-Op2 | 6.3 | 14.2 | 1276 | 1441 | 762 | 743 |
| | D2-Op2 | 0.1 | 1.1 | 33.1 | 57.8 | 16.5 | 21.1 |
| | D2-Op2 | 1.6 | 7.7 | 2.6 | 4.0 | 2.2 | 2.8 |
| | STRUCK THE | | Endad Hall | | | | |
| Mean-Inter | r-Op-Donor2 | 4.7 | 10.8 | 1236 | 1361 | 778 | 762 |
| | r-Op-Donor2 | 2.3 | 4.8 | 57.3 | 113.1 | 22.6 | 26.2 |
| %CV-Inter | -Op-Donor2 | 48.9 | 44.4 | 4.6 | 8.3 | 2.9 | 3.4 |


Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 



## Appendix U: Table 5, Inter/Intra-Assay Precision - Continued

| | | | | MESF | MESF | | |
|---|---|---|---|---|---|---|---|
| | | %tSTAT3 | %tSTAT3 | tSTAT3 | tSTAT3 | %pSTAT3 | %pSTAT3 |
| Table 5 - | | STIM | STIM | STIM | STIM | STIM | STIM |
| inter/Intr | Acquisition | [CD3+ | [CD3+/CD4 | [CD3+ | [CD3+/CD4 | [CD3+ | [CD3+/CD4+ |
| a-Assay | Date | Lymphs] | + Lymphs] | Lymphs] | +Lymphs] | Lymphs] | Lymphs] |
| D1-01-R1 | 2/18/2014 | 63.3 | 74.8 | 3528 | 3588 | 88.6 | 97.4 |
| D1-01-R2 | 2/18/2014 | 63.6 | 71.6 | 3538 | 3551 | 86.8 | 96.8 |
| D1-O1-R3 | 2/18/2014 | 57.0 | 65.8 | 3340 | 3343 | 87.4 | 96.9 |
| | -D1-Op1 | 61.3 | 70.7 | 3469 | 3494 | 87.6 | 97.0 |
| | -D1-Op1 | 3.7 | 4.6 | 111.5 | 132.1 | 0.9 | 0.3 |
| | -D1-Op1 | 6.0 | 6.5 | 3.2 | 3.8 | 1.0 | 0.3 |
| D1-02-R1 | 2/18/2014 | 46.7 | 58.1 | 3003 | 3003 | 89.5 | 98.1 |
| D1-02-R2 | 2/18/2014 | 46.4 | 57.7 | 3001 | 3005 | 89.0 | 98.0 |
| D1-02-R3 | 2/18/2014 | 46.7 | 57.8 | 2976 | 3073 | 88.8 | 98.1 |
| | -D1-Op2 | 46.6 | 57.9 | 2993 | 3027 | 89.1 | 98.1 |
| | -D1-Op2 | 0.2 | 0.2 | 15.0 | 39.8 | 0.4 | 0.1 |
| %CV- | D1-Op2 | 0.4 | 0.3 | 0.5 | 1.3 | 0.4 | 0.1 |
| STATE OF THE PARTY OF | | A VIETNA | V COUNTY IN | | | A STATE OF | |
| | r-Op-Donor1 | 54.0 | 64.3 | 3231 | 3261 | 88.4 | 97.6 |
| | r-Op-Donor1 | 10.4 | 9.1 | 336.6 | 330.2 | 1.1 | 0.8 |
| | r-Op-Dogor1 | 19.3 | 14.2 | 10.4 | 10.1 | 1.2 | 0.8 |
| D2-01-R1 | 2/18/2014 | 39.6 | 49.6 | 2832 | 2794 | 46.9 | 71.1 |
| D2-O1-R2 | 2/18/2014 | 37.0 | 47.9 | 2769 | 2770 | 44.8 | 68.0 |
| D2-O1-R3 | 2/18/2014 | 41.2 | 51.4 | 2856 | 2842 | 46.0 | 70.0 |
| | -D2-Op1 | 39.3 | 49.6 | 2819 | 2802 | 45.9 | 69.7 |
| | -D2-Op1 | 2.1 | 1.8 | 44.9 | 36.7 | 1.1 | 1.6 |
| | D2-Op1 | 5.3 | 3.6 | 1.6 | 1.3 | 2.4 | 2.3 |
| D2-O2-R1 | 2/18/2014 | 35.1 | 43.8 | 2678 | 2654 | 47.3 | 72.1 |
| D2-O2-R2 | 2/18/2014 | 37.4 | 45.6 | 2713 | 2717 | 48.1 | 68.8 |
| D2-O2-R3 | 2/18/2014 | 33.8 | 44.3 | 2666 | 2667 | 47.3 | 69.1 |
| | D2-Op2 | 35.4 | 44.6 | 2686 | 2679 | 47.6 | 70.0 |
| | -D2-Op2 | 1.8 | 0.9 | 24.4 | 33,3 | 0.5 | 1.8 |
| %CV- | D2-Op2 | 5.1 | 2.0 | 0.9 | 1.2 | 1.1 | 2.6 |
| | | | | | BUILDING STATE | | |
| | r-Op-Donor2 | 37.4 | 47.1 | 2753 | 2741 | 46.8 | 69.9 |
| | r-Op-Donor2 | 2.8 | 3.5 | 94.0 | 87.0 | 1.2 | 0.2 |
| %CV-Inter | -Op-Donor2 | 7.5 | 7.4 | 3.4 | 3.2 | 2.6 | 0.3 |


Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 





# Appendix V: Table 5, Inter/Intra-Assay Precision - Continued

| Table 5 -<br>inter/Intra-<br>Assay | Acquisition<br>Date | MESF<br>pSTAT3<br>STIM [CD3+<br>Lymphs] | MESF<br>pSTAT3 STIM<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFItSTAT3<br>unstim [GD3+<br>Lymphs] | MFI tSTAT3 unstim [CD3+/CD4+ Lymphs] |
|---|---|---|---|---|---|---|---|
| D1-O1-R1 | 2/18/2014 | 19904 | 21127 | 161 | 164 | 868 | 872 |
| D1-O1-R2 | 2/18/2014 | 19804 | 21139 | 177 | 176 | 855 | 855 |
| D1-O1-R3 | 2/18/2014 | 18073 | 19237 | 177 | 179 | 839 | 850 |
| Mean- | D1-Op1 | 19260 | 20501 | 172 | 173 | 854 | 859 |
| StDev | -D1-Op1 | 1029.5 | 1094.7 | 9.2 | 7.9 | 14.5 | 11.5 |
| | D1-Op1 | 5.3 | 5.3 | 5.3 | 4.6 | 1.7 | 1.3 |
| D1-O2-R1 | 2/18/2014 | 22534 | 24484 | 208 | 206 | 797 | 809 |
| D1-O2-R2 | 2/18/2014 | 22165 | 23891 | 213 | 215 | 807 | 812 |
| D1-02-R3 | 2/18/2014 | 21179 | 22802 | 214 | 217 | 775 | 783 |
| Mean- | D1-Op2 | 21959 | 23726 | 212 | 213 | 793 | 801 |
| THE PERSON NAMED IN COLUMN TWO IS NOT THE OWNER. | -D1-Op2 | 700.5 | 853.1 | 3.2 | 5.9 | 16.4 | 15.9 |
| | D1-Op2 | 3.2 | 3.6 | 1.5 | 2.8 | 2.1 | 2.0 |
| | | | The state of the state of | | P. Co. Sec | The second second | and the same of th |
| Mean-Inte | r-Op-Donor1 | 20610 | 22114 | 192 | 193 | 824 | 830 |
| StDev-Inte | r-Op-Donor1 | 1908.5 | 2280.4 | 28.3 | 28.3 | 43.1 | 41.0 |
| %CV-Inte | r-Op-Donor1 | 9.3 | 10.3 | 1.4.7 | 14.7 | 5.2 | 4.9 |
| D2-O1-R1 | 2/18/2014 | 2511 | 12197 | 193 | 181 | 735 | 741 |
| D2-O1-R2 | 2/18/2014 | 2291 | 12229 | 192 | 186 | 737 | 735 |
| D2-O1-R3 | 2/18/2014 | 2344 | 12277 | 186 | 187 | 718 | 728 |
| Mean | -D2-Op1 | 2382 | 12234 | 190 | 185 | 730 | 735 |
| | -D2-Op1 | 114.8 | 40.3 | 3.8 | 3.2 | 10.4 | 6.5 |
| | 02-Op1 | 4.8 | 0.3 | 2.0 | 1.7 | 1,4 | 0.9 |
| D2-O2-R1 | 2/18/2014 | 2.583 | 13065 | 191 | 183 | 670 | 664 |
| D2-O2-R2 | 2/18/2014 | 2663 | 11766 | 196 | 189 | 686 | 693 |
| D2-O2-R3 | 2/18/2014 | 2489 | 11976 | 198 | 193 | 697 | 695 |
| Mean | -D2-Op2 | 2578 | 12276 | 195 | 188 | 684 | 684 |
| THE RESERVE THE PROPERTY OF THE PERSON NAMED IN | -D2-Op2 | 87.1 | 708.7 | 3.6 | 5.0 | 13.6 | 17.3 |
| | D2-Op2 | 3.4 | 5.8 | 1.8 | 2.7 | 2.0 | 2.5 |
| * S. L. L. L. | SELVENIA | | | | | | |
| Mean-Inte | r-Op-Donor2 | 2480 | 12255 | 193 | 187 | 707 | 710 |
| | r-Op-Donor2 | 138.6 | 29.7 | 3,5 | 2,1 | 32.5 | 36.1 |
| %CV-Inte | r-Op-Donor2 | 5,6 | 0.2 | 1.8 | 1.1 | 4.6 | 5.1 |



## Appendix W: Table 5, Inter/Intra-Assay Precision - Continued

| Table 5 -<br>inter/Intra-<br>Assay | Acquisitio<br>n Date | MFI pSTAT3 unstim [CD3+ Lymphs] | MFI pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-<br>PESTIM<br>[CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3 STIM [CD3+ Lymphs] | MFI tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3 STIM [CD3+ Lymphs] | MFI pSTAT3 STIM [CD3+/CD4+ |
|---|---|---|---|---|---|---|---|---|---|
| D1-01-R1 | 2/18/2014 | 527 | 625 | 174 | 172 | 800 | 813 | 4011 | 4240 |
| D1-O1-R2 | 2/18/2014 | 551 | 655 | 180 | 176 | 803 | 805 | 3992 | 4242 |
| D1-01-R3 | 2/18/2014 | 566 | 645 | 188 | 178 | 760 | 761 | 3666 | 3885 |
| Mean-D | 1-Op1 | 548 | 642 | 181 | 175 | 788 | 793 | 3890 | 4122 |
| StDev-D | | 19.7 | 15.3 | 7.0 | 3.1 | 24.0 | 28.0 | 193.9 | 7 74 544 |
| %CV-D: | 1-Op1 | 3.6 | 2.4 | 3.9 | 1.8 | 3.0 | 3.5 | 5.0 | 205.5 |
| D1-02-R1 | 2/18/2014 | 601 | 694 | 163 | 164 | 689 | 689 | 4502 | |
| D1-02-R2 | 2/18/2014 | 577 | 675 | 173 | 173 | 688 | 689 | 4434 | 4864 |
| D1-O2-R3 | 2/18/2014 | 587 | 683 | 167 | 163 | 683 | 704 | 4250 | |
| Mean-D1-Op2 | | 588 | 684 | 168 | 167 | 687 | 694 | | 4552 |
| StDev-D1-Op2 | | 12.1 | 9.5 | 5.0 | 5.5 | 3.2 | 8.7 | 4395 | 4723 |
| %CV-D1-Op2 | | 2.1 | 1.4 | 3.0 | 3,3 | 0.5 | 1.3 | 130.4 | 158.2 |
| STATE OF STREET | a. Or a street | | A STATE OF THE STA | LIFY THE | S. J. | | 1.5 | 3.0 | 3.3 |
| Mean-Inter-Op-Donor1 | | 568 | 663 | 175 | 171 | 738 | 744 | 44.42 | SAME SAME |
| StDev-Inter- | Op-Donor1 | 28.3 | 29.7 | 9.2 | 5.7 | 71.4 | 70.0 | 4143 | 4423 |
| %CV-Inter-C | | 5.0 | 4.5 | 5.3 | 3.3 | 9.7 | 9.4 | 357.1 | 425.0 |
| D2-O1-R1 | 2/18/2014 | 288 | 303 | 198 | 187 | 652 | 644 | 8.6 | 9.6 |
| D2-O1-R2 | 2/18/2014 | 297 | 320 | 196 | 195 | 639 | 639 | 583 | 2542 |
| D2-O1-R3 | 2/18/2014 | 291 | 311 | 204 | 207 | 657 | | 535 | 2548 |
| Mean-D | 2-Op1 | 292 | 311 | 199 | 196 | | 654 | 547 | 2557 |
| StDev-D | | 4.6 | 8,5 | 4.2 | 10.1 | 649 | 646 | 555 | 2549 |
| %CV-D2 | | 1.6 | 2.7 | 2.1 | 5.2 | 9.3 | 7.6 | 25.0 | 7.5 |
| D2-O2-R1 | 2/18/2014 | 311 | 339 | 192 | 187 | 1.4 | 1.2 | 4.5 | 0.3 |
| D2-O2-R2 | 2/18/2014 | 303 | 341 | 188 | 183 | 619 | 614 | 599 | 2714 |
| D2-02-R3 | 2/18/2014 | 318 | 363 | 196 | 193 | 627 | 628 | 616 | 2458 |
| Mean-D2 | | 311 | 348 | | | 617 | 617 | 578 | 2499 |
| | | 7.5 | 13.3 | 192 | 188 | 621 | 620 | 598 | 2557 |
| StDev-D2-Op2<br>%CV-D2-Op2 | | 2.4 | 3.8 | 4.0<br>2.1 | 5.0 | 5.3 | 7.4 | 19.0 | 137.5 |
| 70.2 | | 2.7 | 3.0 | Z. 1 | 2.7 | 0.9 | 1.2 | 3.2 | 5.4 |
| Mean-Inter-C | In-Donor? | 302 | 330 | 100 | 400 | CONTRACT OF | | | |
| StDev-Inter-C | | 13.4 | 26.2 | 196<br>4.9 | 192 | 635 | 633 | 577 | 2553 |
| %CV-Inter-C | | 4.4 | 7.9 | 2.5 | 5.7 | 19.8 | 18.4 | 30.4 | 5.7 |
| -10-1 MINGS C | h portors | ा≽ क | 7.3 | 4.0 | 3.0 | 3.1 | 2.9 | 5.3 | 0.2 |





Appendix X: Table 6: Assay Transfer, Flow Assay

| Table 6: Assay<br>Transfer | Acquisition<br>Date | %Lymphs | Region Events<br>CD3+ Lymphs | %CD3+<br>[Lymphs] | Region<br>Events<br>CD3+/CD4+<br>Lymphs | %CD3+/CD4<br>[Lymphs] | PEunstim | MESF FM O-<br>PE unstim<br>[CD3+/CD4+<br>Lymphs] | %tSTAT3<br>unstim<br>[CD3+<br>Lymphs] | %tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|
| DONOR1A | 4/22/2014 | 20.7 | 4214 | 81.1 | 2643 | 62.7 | 1080 | 1075 | 46.2 | 44.8 |
| DONOR1B | 4/22/2014 | 34.5 | 6213 | 79.0 | 4010 | 64.5 | 874 | 876 | 44.7 | 46.9 |
| DONOR1C | 4/22/2014 | 33,9 | 6033 | 79.4 | 3956 | 65.6 | 874 | 884 | 39.9 | 42.9 |
| Mea | n | 29.7 | 5487 | 79.8 | 3536 | 64.3 | 943 | 945 | 43.6 | 44.9 |
| StDev | | 7,8 | 1105.8 | 1.1 | 774.1 | 1.5 | 118.9 | 112.7 | 3.3 | 2.0 |
| %CV | | 26.3 | 20.2 | 1.4 | 21.9 | 2.3 | 12.6 | 11.9 | 7.6 | 4.5 |
| DONOR2A | 4/22/2014 | 27.9 | 4647 | 66.8 | 3447 | 74.2 | 739 | 743 | 19.0 | 19.0 |
| DONOR2B | 4/22/2014 | 27.8 | 4551 | 66.0 | 3369 | 74.0 | 776 | 768 | 42.7 | 42.2 |
| DONOR2C | 4/22/2014 | 26.6 | 5354 | 67.0 | 3967 | 74.1 | 824 | 811 | 43.6 | 41.5 |
| Mea | n | 27.4 | 4851 | 66.6 | 3594 | 74.1 | 780 | 774 | 35.1 | 34.2 |
| StDe | ev | 0.7 | 438.5 | 0.5 | 325.1 | 0.1 | 42.6 | 34.4 | 14.0 | 13.2 |
| %C | V | 2.6 | 9.0 | 0.8 | 9.0 | 0.1 | 5.5 | 4.4 | 39.9 | 38.6 |
| DONOR3A | 4/22/2014 | 16.5 | 4000 | 53.4 | 2614 | 65.4 | 756 | 751 | 56.1 | 54.6 |
| DONOR3B | 4/22/2014 | 15.9 | 4104 | 55.0 | 2656 | 64.7 | 616 | 624 | 22.0 | 22.1 |
| DONOR3C | 4/22/2014 | 15.9 | 4300 | 56.8 | 2788 | 64.8 | 642 | 640 | 21.6 | 22.6 |
| Mean | | 16.1 | 4135 | 55.1 | 2686 | 65.0 | 671 | 672 | 33.2 | 33.1 |
| StD | | 0.3 | 152.3 | 1.7 | 90.8 | 0.4 | 74.5 | 69.2 | 19.8 | 18.6 |
| %C | | 1.9 | 3.7 | 3.1 | . 3.4 | 0.6 | 11.1 | 10.3 | 59.5 | 56.2 |





Appendix Y: Table 6: Assay Transfer, Flow Assay - Continued

| Table 6: Assay Transfer | Acquisition<br>Date | MESF<br>tSTAT3<br>unstim<br>[CD3+<br>Lymphs] | MESF<br>tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+<br>Lymphs] | %pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3 unstim [CD3+ Lymphs] | MESF pSTAT3 unstim [CD3+/CD4+ Lymphs] | MESF FMO-<br>PESTIM<br>[CD3+<br>Lymphs] | MESF FMO<br>PESTIM<br>[CD3+/CD4-<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|
| DONOR1A | 4/22/2014 | 2014 | 1982 | 10.4 | 11.0 | 1270 | 1261 | 726 | 729 |
| DONOR1B | 4/22/2014 | 1998 | 1987 | 8.8 | 8.8 | 1235 | 1264 | 692 | 679 |
| DONOR1C | 4/22/2014 | 1903 | 1949 | 9.5 | 10.4 | 1287 | 1395 | 742 | 733 |
| Mean | | 1972 | 1973 | 9.6 | 10.1 | 1264 | 1307 | 720 | 714 |
| StDev | | 60.0 | 20.6 | 0.8 | 1.1 | 26.5 | 76.5 | 25.5 | 30.1 |
| %CV | | 3.0 | 1.0 | 8.3 | 10.9 | 2.1 | 5,9 | 3.5 | 4.2 |
| DONORZA | 4/22/2014 | 1538 | 1517 | 10.5 | 13.6 | 1150 | 1221 | 916 | 909 |
| DONOR2B | 4/22/2014 | 1960 | 1930 | 15.5 | 19.3 | 1320 | 1414 | 777 | 772 |
| DONOR2C | 4/22/2014 | 1969 | 1929 | 17.6 | 22.1 | 1365 | 1488 | 842 | 831 |
| Mean | | 1822 | 1792 | 14.5 | 18.3 | 1278 | 1374 | 845 | 837 |
| StDev | | 246.3 | 238.2 | 3.6 | 4.3 | 113.4 | 137.8 | 69.5 | 68.7 |
| %CV | | 13.5 | 13.3 | 24.8 | 23.5 | 8.9 | 10,0 | 8.2 | 8.2 |
| DONOR3A DONOR3A | 4/22/2014 | 2188 | 2151 | 19.0 | 23.9 | 1379 | 1494 | 655 | 647 |
| DONOR3B | 4/22/2014 | 1593 | 1592 | 10.4 | 13.2 | 1104 | 1174 | 643 | 639 |
| DONOR3C | 4/22/2014 | 1604 | 1606 | 10.8 | 13.5 | 1133 | 1203 | 704 | 688 |
| Mean | | 1795 | 1783 | 13.4 | 16.9 | 1205 | 1290 | 667 | 658 |
| StDev | | 340.4 | 318.8 | 4.9 | 6.1 | 151.1 | 177.0 | 32.3 | 26.3 |
| %CV | | 19.0 | 17.9 | 36.6 | 36.1 | 12.5 | 13.7 | 4.8 | 4.0 |





Appendix Z: Table 6: Assay Transfer, Flow Assay - Continued

| Table 6:<br>Assay<br>Transfer | Acquisition<br>Date | %tSTAT3<br>STIM<br>[CD3+<br>Lymphs] | %tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF<br>tSTAT3<br>STIM<br>[CD3+<br>Lymphs] | MESF<br>tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | %pSTAT3<br>STIM<br>[CD3+<br>Lymphs] | %pSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MESF pSTAT3 STIM [CD3+ Lymphs] | MESF pSTAT3 STIM [CD3+/CD4+ Lymphs] | MFI FMO-<br>PE unstim<br>[CD3+<br>Lymphs] | MFI FMO-PE<br>unstim<br>[CD3+/CD4+<br>Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| DONOR1A | 4/22/2014 | 36.3 | 34.3 | 1851 | 1803 | 86.5 | 93.2 | 12627 | 13083 | 368 | 366 |
| DONOR1B | 4/22/2014 | 31.0 | 28.2 | 1766 | 1708 | 89.1 | 95.3 | 12540 | 12901 | 298 | 299 |
| DONOR1C | 4/22/2014 | 32.5 | 29.9 | 1796 | 1734 | 88.2 | 94.3 | 12038 | 12309 | 298 | 301 |
| | ean | 33.3 | 30.8 | 1804 | 1748 | 87.9 | 94.3 | 12402 | 12764 | 321 | 322 |
| | Dev | 2.7 | 3.1 | 43.1 | 49.1 | 1.3 | 1.1 | 317.9 | 404.7 | 40.4 | 38.1 |
| | CV | 8.1 | 10.1 | 2.4 | 2.8 | 1.5 | 1.2 | 2.6 | 3.2 | 12.6 | 11.8 |
| DONOR2A | 4/22/2014 | 50.6 | 50.4 | 2093 | 2080 | 83.9 | 97.3 | 13484 | 14897 | 252 | 253 |
| DONOR23 | 4/22/2014 | 45.2 | 44.3 | 1991 | 1968 | 83.0 | 97.5 | 14121 | 15651 | 265 | 262 |
| DONORZC | 4/22/2014 | 30,7 | 30.1 | 1771 | 1744 | 82.6 | 97.0 | 13284 | 14856 | 281 | 277 |
| | ean | 42.2 | 41.6 | 1952 | 1931 | 83.2 | 97.3 | 13630 | 15135 | 266 | 264 |
| | Dev | 10.3 | 10.4 | 164.6 | 171.1 | 0.7 | 0.3 | 437.1 | 447.6 | 14.5 | 12.1 |
| | CV | 24.4 | 25.0 | 8.4 | 8.9 | 0.8 | 0.3 | 3.2 | 3.0 | 5.5 | 4.6 |
| DONORSA | 4/22/2014 | 26.8 | 26.6 | 1692 | 1682 | 85.4 | 94.0 | 10881 | 11883 | 258 | 256 |
| DONOR3B | 4/22/2014 | 23.0 | 23.7 | 1613 | 1619 | 85.6 | 95.1 | 11717 | 12874 | 210 ; | 213 |
| DONOR3C | 4/22/2014 | 27.7 | 28.1 | 1699 | 1693 | 86.2 | 95.0 | 11071 | 12140 | 219 | 218 |
| | ean | 25.8 | 26.1 | 1668 | 1665 | 85.7 | 94.7 | 11223 | 12299 | 229 | 229 |
| | Dev | 2.5 | 2.2 | 47.8 | 39.9 | 0.4 | 0.6 | 438.2 | 514.3 | 25.5 | 23.5 |
| | CV | 9.7 | 8.4 | 2,9 | 2.4 | 0.5 | 0.6 | 3.9 | 4.2 | 11.1 | 10.3 |



Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

#### Appendix AA: Table 6: Assay Transfer, Flow Assay - Continued

| Table 6:<br>Assay<br>Transfer | Acquisition<br>Date | Lymphs] | MFI tSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3<br>unstim<br>[CD3+<br>Lymphs] | MFI pSTAT3<br>unstim<br>[CD3+/CD4+<br>Lymphs] | MFI FMO-PE<br>STIM [CD3+<br>Lymphs] | MFI FMO-PE<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI tSTAT3<br>STIM [CD3+<br>Lymphs] | MFI tSTAT3<br>STIM<br>[CD3+/CD4+<br>Lymphs] | MFI pSTAT3 STIM [CD3+ Lymphs] | MFI pSTAT3 STIM [CD3+/CD4- Lymphs] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| DONOR1A | 4/22/2014 | 685 | 674 | 432 | 429 | 248 | 249 | 629 | 613 | 4262 | 4415 |
| DONOR1B | 4/22/2014 | 679 | 676 | 421 | 430 | 236 | 232 | 601 | 581 | 4233 | 4354 |
| DONOR1C | 4/22/2014 | 647 | 663 | 438 | 475 | 253 | 250 | 611 | 590 | 4064 | 4155 |
| Me | ean | 670 | 671 | 430 | 445 | 246 | 244 | 614 | 595 | 4186 | 4308 |
| Sti | Dev | 20.4 | 7.0 | 8.6 | 26.3 | 8.7 | 10.1 | 14.2 | 16.5 | 106.9 | 136.0 |
| % | CV | 3.0 | 1.0 | 2.0 | 5.9 | 3.5 | 4,1 | 2.3 | 2.8 | 2.6 | 3.2 |
| DONOR2A | 4/22/2014 | 523 | 516 | 392 | 416 | 312 | 310 | 711 | 707 | 4550 | 5025 |
| DONOR2B | 4/22/2014 | 666 | 656 | 449 | 481 | 265 | 263 | 677 | 669 | 4764 | 5278 |
| DONOR2C | 4/22/2014 | 669 | 656 | 465 | 506 | 287 | 284 | 602 | 593 | 4483 | 5011 |
| Me | ean | 619 | 609 | 435 | 468 | 288 | 286 | 663 | 656 | 4599 | 5105 |
| Sti | Dev | 83.4 | 80.8 | 38.4 | 46.5 | 23.5 | 23.5 | 55.8 | 58.0 | 146.8 | 150.3 |
| % | CA | 13.5 | 13.3 | 8.8 | 9.9 | 8.2 | 8.2 | 8.4 | 8.8 | 3.2 | 2.9 |
| DONOR3A | 4/22/2014 | 743 | 731 | 469 | 509 | 224 | 221 | 576 | 572 | 3675 | 4012 |
| DONOR3B | 4/22/2014 | 543 | 538 | 376 | 400 | 220 | 218 | 549 | 551. | 3956 | 4345 |
| DONOR3C | 4/22/2014 | 546 | 546 | 386 | 410 | 240 | 235 | 578 | 576 | 3739 | 4098 |
| Me | an | 611 | 605 | 410 | 440 | 228 | 225 | 568 | 566 | 3790 | 4152 |
| Sti | Dev | 114.6 | 109.2 | 51,1 | 60.3 | 10.6 | 9.1 | 16.2 | 13.4 | 147.3 | 172.9 |
| % | CA | 18.8 | 18.0 | 12.5 | 13.7 | 4.6 | 4.0 | 2.9 | 2.4 | 3.9 | 4.2 |

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

Appendix BB: Table 7: Assay Transfer, Flow Assay %Stimulation and Acceptance

| Table 7: %Stimulation and Assay Transfer Accepance | in CD3+ (Lymphs) Based on %pSTAT | in CD3+/CD4+ (Lymphs) Based on %pSTAT | in CD3+ (Lymphs) Based on MESF pSTAT | in CD3+/CD4+ (Lymphs) Based on MESF pSTAT |
|---|---|---|---|---|
| AT-Donor 1 (AVG R1-R3) | 815.6 | 833.7 | 881.0 | 876.6 |
| AT-Donor 2 (AVG R1-R3) | 473.8 | 431.7 | 967.0 | 1001,5 |
| AT-Donor 3 (AVG R1-R3) | 539.6 | 460.4 | 831.0 | 853.4 |
| Precision-Donor 1 (AVG R1-R3) | 140.7 | 96.8 | 720.3 | 636.9 |
| Precision-Donor 2 (AVG R1-R3) | 1430.0 | 841.9 | 99.3 | 855.0 |
| LinDonor 1 @2000 Cells (AVG R1-R3) | 2158.3 | 1483.1 | 283.9 | 1241.2 |
| LinDonor 2 @2000 Cells (AVG R1-R3) | 80.8 | 92.1 | 962,0 | 888.9 |
| LinDonor 3 @2000 Cells (AVG R1-R3) | 74.7 | 49.2 | 713.0 | 635.0 |
| Mean Biological Variability | 714.2 | 536.1 | 682,2 | 873.6 |
| StDEV Biological Variability | 740.2 | 496.1 | 321.1 | 194.7 |
| Mean + 1StDEV | 1454.4 | 1032.2 | 1003.3 | 1068.3 |
| Mean - 1StDEV | -26.0 | 40.0 | 361.1 | 678.9 |



Appendix CC: Gating Strategy

Validation Report LCT13050-QR01-01 Gilead pSTAT3 Stim Cytometry Assay 26-Apr-2014 

